### Janssen Research & Development \*

### Statistical Analysis Plan Amendment 3

A Phase 3 Randomized, Double-blind, Placebo-controlled, Multi-center Study to Evaluate the Efficacy and Safety of Pimodivir in Combination With the Standard-of-care Treatment in Adolescent, Adult, and Elderly Non-hospitalized Subjects With Influenza A Infection who Are at Risk of Developing Complications

Protocol 63623872FLZ3002; Phase 3

**JNJ-63623872-ZCD** (Pimodivir)

Status: Approved Date: 1 July 2020

**Prepared by:** Janssen Research & Development, a division of Janssen Pharmaceutica NV

**Document No.:** EDMS-ERI-151898626, 5.0

**Compliance:** The study described in this report was performed according to the principles of Good Clinical Practice (GCP).

# **Confidentiality Statement**

The information provided herein contains Company trade secrets, commercial or financial information that the Company customarily holds close and treats as confidential. The information is being provided under the assurance that the recipient will maintain the confidentiality of the information under applicable statutes, regulations, rules, protective orders or otherwise.

# **TABLE OF CONTENTS**

| TABLE | OF CONTENTS | <mark>2</mark> |
|---|---|---|
| AMEN | DMENT HISTORY | 5 |
| ABBRI | EVIATIONS | 12 |
| 1. II | NTRODUCTION | 13 |
| 1.1. | Trial Objectives | |
| 1.2. | Trial Design | |
| 1.3. | Statistical Hypotheses for Trial Objectives | |
| 1.4. | Sample Size Justification | |
| 1.5. | Randomization and Blinding | |
| 2. G | SENERAL ANALYSIS DEFINITIONS | 18 |
| 2.1. | Visit Windows, Phase Definitions and Baseline | 18 |
| 2.1.1. | Phase Definitions | 18 |
| 2.1.2. | Analysis visits | 19 |
| 2.1.3. | Analysis timepoints | 19 |
| 2.1.4. | Use of records per analysis visit and timepoint | 19 |
| 2.1.5. | Unscheduled Assessments | 20 |
| 2.2. | Analysis Sets | 21 |
| 2.2.1. | All Randomized Analysis Sets | 21 |
| 2.2.1.1 | . All Randomized Analysis Set (RAND) | 21 |
| 2.2.1.2 | . Randomized and/or Treated Analysis Set (RT) | 21 |
| 2.2.2. | Efficacy Analysis Sets | |
| 2.2.2.1 | \ | |
| 2.2.2.2 | | |
| 2.2.2.3 | \ | |
| 2.2.3. | Safety Analysis Set | 23 |
| 2.2.3.1 | | |
| 2.2.4. | Pharmacokinetics (PK) Analysis Set | |
| 2.2.5. | Pharmacodynamics (PD) Analysis Set | |
| 2.3. | Definition of Subgroups | |
| 2.4. | Study Day and Relative Day | |
| 2.5. | Baseline and Endpoint | |
| 2.6. | Other Definitions | 27 |
| | NTERIM ANALYSIS AND DATA MONITORING COMMITTEE REVIEW | |
| 3.1. | Interim Analysis | |
| 3.2. | Independent Data Monitoring Committee | 28 |
| | SUBJECT INFORMATION | |
| 4.1. | Demographics and Baseline Characteristics | |
| 4.2. | Disposition Information. | |
| 4.3. | Treatment Compliance | |
| 4.4. | Extent of Exposure | |
| 4.5. | Protocol Deviations | |
| 4.6. | Prior and Concomitant Medications | |
| 4.7. | Medical history | 32 |
| | FFICACY | |
| 5.1. | Analysis Specifications | |
| 5.1.1. | Level of Significance | |
| 5.1.2. | Data Handling Rules | 34 |

| 5.1.3. | Stratification Factors | |
|---|---|---|
| 5.2. | Primary Efficacy Endpoint(s) | |
| 5.2.1. | Definition | 35 |
| 5.2.2. | Estimand | |
| 5.2.3. | Analysis Methods | |
| 5.3. | Major Secondary Endpoints | |
| 5.3.1. | Definition | |
| 5.3.1. | | |
| 5.3.1.2 | · | |
| 5.3.1.3 | | |
| 5.3.1.4 | | |
| 5.3.2. | Analysis Methods | |
| 5.3.2. | | |
| 5.3.2.2 | · · | |
| 5.3.2.3 | | |
| 5.3.2.4 | | |
| 5.4. | Exploratory Endpoints | |
| 5.4.1. | | 55 |
| 5.4.1. | 1 | |
| 5.4.2. | Analysis Methods | 56 |
| 5.4.2. | 1. Impact of Influenza (Flu-iiQ™ Modules 2, 3, 4) | 50 |
| 6. | TASTE AND SWALLOWABILITY | 57 |
| 6.1. | Definition | - |
| 6.2. | Analysis Methods | |
| | SAFETY | |
| 7.1. | Adverse Events | |
| 7.1.1. | Definitions | |
| 7.1.2. | Analysis Methods | |
| 7.2. | Clinical Laboratory Tests | |
| 7.2.1. | Definitions | |
| 7.2.2. | Analysis Methods | |
| 7.3. | Vital Signs | |
| 7.3.1. | Definitions | |
| 7.3.2. | Analysis Methods | |
| 7.4. | Physical examinations | |
| 7.5. | Electrocardiogram | |
| 7.5.1.<br>7.5.2. | Definitions | |
| 1.5.2. | Arialysis Methods | 00 |
| 8. I | RESISTANCE | 67 |
| 8.1. | Viral Phenotype | |
| 8.2. | Viral Genotype | 67 |
| | DUADMA COMBITACO/DUADMA CODYNAMICO | - |
| | PHARMACOKINETICS/PHARMACODYNAMICS | |
| 9.1.<br>9.2. | PharmacokineticsPharmacodynamic Relationships | |
| 9.2. | Pharmacokinetic/Pharmacodynamic Relationships | 00 |
| 10. I | HEALTH ECONOMICS | 70 |
| 10.1. | Definitions | 70 |
| 10.2. | Analysis Methods | |
| ATTA | CHMENTS | 72 |
| ATTA | CHMENT 1. : ANTICIPATED EVENTS AND ANTICIPATED EVENT GROUPS | 72 |
| | ATTACHMENT 2. : WHO TOXICITY GRADING SCALE FOR DETERMINING THE SEVERITY OF ADVERSE EVENTS (FEB 2003)75 | |

| ATTACHMENT 3. | : WHO GRADING SCALE VITAL SIGNS | . 80 |
|---------------|---------------------------------|------|
| ATTACHMENT 4. | : ECG ABNORMALITIES | . 81 |
| ATTACHMENT 5. | : EQ-5D VALUATION INDEX | . 82 |

#### AMENDMENT HISTORY

Amendments are listed beginning with the most recent amendment.

## Amendment 3 (1 July 2020)

The overall reason for the amendment: The overall reason for the amendment is to describe additional data presentations required to assess the impact of the COVID-19 pandemic. In addition, censoring due to hospitalization for the primary endpoint is clarified. The derivation of the endpoint time to resolution of fever was clarified and more detail regarding the definition of a treatment emergent adverse event was added. Also, to make general updates to the text including minor grammatical, formatting, or spelling changes throughout the SAP for clarification purposes.

### The table below gives an overview of the changes in all applicable sections

**Summary of changes:** End date time of the last phase is clarified.

2.1.1 Phase Definitions

**Summary of changes:** It was clarified that the safety follow-up visit and Day 28 final study visit are to be included as analysis visits.

2.1.2 Analysis Visits

**Summary of changes:** Exclusion criterion 13 was added to the list for determining inclusion in the per protocol analysis set. The use of concomitant medications that may have affected the efficacy was removed from the list.

2.2.2.2 Per Protocol Set (PP)

**Summary of changes:** Clarification that analyses including the subgroup 'study period' will be performed separately for each category of the subgroup and not by including the subgroup as an interaction term in the statistical model was added. The subgroup COVID-19 impacted was added.

2.3 Definition of Subgroups

**Summary of changes:** The definition of the last study visit for vital signs, ECG, and central laboratory data was added.

2.5 Baseline and Endpoint

**Summary of changes:** Added the number (%) of subjects within the analysis sets impacted by COVID-19 to the disposition information.

4.2 Disposition Information

**Summary of changes:** Added listings for protocol deviations related to COVID-19.

4.5 Protocol Deviations

**Summary of changes:** Added a tabulation of concomitant medications administered to treat COVID-19 infection.

4.6 Prior and Concomitant Medications

**Summary of changes:** The value to be imputed when the  $log_{10}$  TCID<sub>50</sub> viral titer is recorded as '<0.75' was changed from '0.75' to '0.74' to avoid confusion with actual values recorded as '0.75'.

5.1.2 Data Handling Rules

**Summary of changes:** Added Baloxavir Marboxil to the list of influenza antivirals.

5.1.3 Stratification Factors

**Summary of changes:** The determination of whether a symptom was pre-existing, or not, was added. Also censoring due to hospitalization was clarified.

5.2 Primary Efficacy Endpoint(s)

**Summary of changes:** The derivation of the secondary endpoint time to resolution of fever was clarified.

5.3.1.3 Clinical outcomes

**Summary of changes:** Documented that implausible values recorded by the subject for body temperature on the ePRO device will not be included in any analysis.

5.3.2.3 Clinical outcomes

**Summary of changes:** The derivation of the duration of an adverse event was added. The definition of a treatment-emergent adverse event was clarified.

7.1 Adverse Events

**Summary of changes:** Tabulations and listings of COVID-19 related AEs were added.

7.1.2 Analysis Methods

### Amendment 2 (07 November 2019)

The overall reason for the amendment: The overall reason for the amendment is to address the FDA 8 May 2019 comments regarding amendment 1 of the statistical analysis plan for this study. Also, to make general updates to the text including minor grammatical, formatting, or spelling changes throughout the SAP for clarification purposes. The estimand was updated to state that the Kaplan-Meier estimate of median time to resolution of the 7 primary influenza-related symptoms would be the primary method for treatment effect estimation. Sensitivity analyses to account for missing assessments in the time to resolution primary endpoint were included. Also, two new subgroups were added namely influenza season and study period (pre interim, post interim). All changes are outlined below.

## The table below gives an overview of the changes in all applicable sections

**Summary of changes:** The criterion: "Subjects did not switch to another influenza antiviral as a part of the SOC during the treatment period" was added to the definition of the per protocol analysis set.

2.2.2 Efficacy Analysis Sets

**Summary of changes:** Two new subgroups were added namely influenza season and study period (pre interim, post interim).

2.3 Definition of Subgroups

Summary of changes: Detailing the definition of baseline ECG measurement was added.

2.5 Baseline and Endpoint

**Summary of changes:** Section 2.6 was changed from Oseltamivir Subset to Other Definitions to include text detailing potential analyses for other regions or countries.

2.6 Other Definitions

**Summary of changes:** The primary method for treatment effect estimation was changed to the Kaplan-Meier estimate of median time to resolution of the 7 primary influenza-related symptoms as per Agency's request.

5.2.2 Estimand

**Summary of changes:** Sensitivity analyses for the primary endpoint were included as per Agency's request.

5.2.3 Analysis Methods

**Summary of changes:** Adverse events leading to study discontinuation was added to the list for the adverse event summary table. A table of influenza-related complications as assessed by the investigator was added. Additional tables to characterize adverse events of diarrhea were added including: number of days from first dose of study drug to onset of event; total duration of diarrhea episodes; number of days from last dose to resolution of the event; severity grade of the event; and any concomitant medication given to treat the event.

7.1.2 Analysis Methods

**Summary of changes:** Details regarding how to use ECG measurements taken while the subject was not in a supine position were added.

7.5.1 Definitions

**Summary of changes:** A table showing descriptive statistics for the pimodivir plasma concentration over time was added.

9 Pharmacokinetics/Pharmacodynamics

**Summary of changes:** Tables for the PK parameter  $C_{trough}$  by safety endpoints were removed. Adverse events at least possibly related to study drug was added as a safety endpoint for assessing the relationship between the PK parameter  $AUC_{12h}$  and safety.

9.2 Pharmacokinetic/Pharmacodynamic Relationships

# Amendment 1 (28 March 2019)

**The overall reason for the amendment:** The overall reason for the amendment is to update the analysis sets and endpoints due to changes made to the protocol (Clinical Protocol Amendment 1, 08-Feb-2018). Also, to make general updates to the text including minor grammatical, formatting, or spelling changes throughout the SAP for clarification purposes. Three new sections are added: one to describe the derivation of the actual values of the stratification factors, one to describe the oseltamivir subset of subjects in detail, and one to include analysis of pharmacokinetic parameters and pharmacodynamic analyses. A new efficacy analysis set, the intent-to-treat non-infected set, is included. Two new secondary endpoints based on a clinically relevant change from baseline in EQ-5D VAS are included. A new secondary clinical endpoint of incidence of adjudicated treatment-emergent influenza complications including hospital admission and an analysis of confirmed diarrhea adverse events are included. One additional definition of resolution of influenza symptoms and related time-to-event endpoint is added, based on an improvement from baseline. Secondary endpoints of time to resolution for each of the 10 individual influenza-related symptoms questions included in Module 1 of the Flu-iiQ<sup>TM</sup> PRO were added to replace the time to resolution endpoint based on all 10 influenza-related symptoms. The composite symptom score endpoint based on all 10 influenza-related symptoms was replaced by 2 new secondary endpoints: composite symptom score for systemic symptoms and composite symptom score for respiratory symptoms. The assigned analysis timepoints for the PRO assessments of Flu-iiQ<sup>TM</sup> and temperature were updated to be more aligned with the ePRO entry time windows.

# The table below gives an overview of the changes in all applicable sections

**Summary of changes:** The assigned analysis timepoints for the PRO assessments of Flu-iiQ<sup>TM</sup> and temperature were updated to be more aligned with the ePRO entry time windows.

#### 2.1.3 Analysis Timepoints

**Summary of changes:** The definition of confirmed influenza A was modified to remove confirmation based on local lab testing, affecting the ITT-i analysis set. An additional analysis set was defined for the analysis of the primary endpoint and the two key secondary endpoints. Additional analysis sets were defined for the pharmacodynamic analyses and the analysis of pharmacokinetics parameters.

## 2.2.2 Efficacy Analysis Sets

**Summary of changes:** Baseline resistance categories were defined based on influenza polymerase basic protein 2 genotype and phenotype. Baseline fever was added as a new subgroup for the analysis of time to resolution of fever. General re-formatting to assist readability of the section.

## 2.3 Definition of Subgroups

**Summary of changes:** A new section (2.6) was added to describe the subset of subjects who have oseltamivir use as part of their SOC treatment to support marketing authorization approval in EMA.

2.6 Oseltamivir Subset

**Summary of changes:** A new section (5.1.3) was added to describe how the actual values of the stratification factors are derived.

5.1.3 Stratification Factors

**Summary of changes:** The text describing the estimand is updated to bring it into line with the ICH E9 addendum guidance.

5.2.2 Estimand

**Summary of changes:** The specification of the statistical models for the analysis of the primary endpoint was clarified, including how missing data for the baseline covariate will be handled. Descriptive statistics to assess the amount of missing data for the primary endpoint was added.

5.2.3 Analysis Methods

**Summary of changes:** An extra definition of the time to resolution of the 7 primary influenzarelated symptoms was added as a sensitivity analysis.

The time to resolution of all influenza-related symptoms was replaced by time to resolution of each of the 10 individual influenza-related symptoms questions. The composite symptom score based on all 10 influenza-related symptoms was replaced by 2 new secondary endpoints: composite symptom score for systemic symptoms and composite symptom score for respiratory symptoms.

- 5.3.1.1 Symptoms of Influenza
- 5.3.2.1 Symptoms of Influenza (Flu-iiQ<sup>TM</sup> Module 1)

**Summary of changes:** The change from baseline in EQ-5D VAS is categorized in two ways providing two additional endpoints.

5.3.1.2 Other Patient Reported Outcome

**Summary of changes:** A new clinical endpoint of incidence of adjudicated treatment-emergent influenza complications including hospital admission is included.

- 5.3.2.3 Clinical outcomes
- 5.3.3.3 Clinical outcomes

**Summary of changes:** A bootstrapping method for calculating the median time to event with 95% confidence interval from the accelerated failure time model was added.

# 5.3.2 Analysis Methods

**Summary of changes:** Additional details regarding number of loose stools per day and stool consistency will be collected for subjects who report diarrhea adverse events. A confirmed diarrhea event is defined and the analysis of these events is described. Additional tabulations of AEs are described for inclusion in the plain language summary document.

#### 7.1.1 Definitions

#### 7.1.2 Analysis Methods

**Summary of changes:** A new section was added to describe the analysis of the pharmacokinetic parameters and their relationships with efficacy and safety.

- 9 Pharmacokinetics/Pharmacodynamics
- 9.1 Pharmacokinetics
- 9.2 Pharmacokinetic/Pharmacodynamic Relationships

#### **ABBREVIATIONS**

AE adverse event

AFT accelerated failure time

ATC Anatomical Therapeutic Chemical

AUC area under the curve

 $AUC_{12h}$  area under the plasma concentration-time curve from time 0 to 12 hours

bid bis in die; twice daily
BMI body mass index
CI confidence interval

C<sub>max</sub> maximum plasma concentration COPD Chronic Obstructive Pulmonary Disease

CTP clinical trial protocol

C<sub>trough</sub> Plasma concentration just prior to the beginning or at the end of a dosing interval

CV coefficient of variation
DBP diastolic blood pressure
DMC Data Monitoring Committee
DPS Data Presentation Specifications
EC<sub>50</sub> 50% effective concentration

ECG Electrocardiogram

eCRF electronic case report form EMA European Medicines Agency

ePRO electronic Patient-reported Outcome (device used for recording of patient-reported outcomes)

EQ-5D European Quality of Life 5 Dimensions

FDA Food and Drug Administration

GMR geometric mean ratio

IC<sub>50</sub> 50% inhibitory concentration ICF informed consent form

ICH International Conference on Harmonization
IDMC Independent Data Monitoring Committee

ITT Intent-To-Treat

ITT-i Intent-To-Treat infected
ITT-ni Intent-To-Treat non-infected
IWRS Interactive web response system

LOD limit of detection LOQ limit of quantification

MedDRA Medical Dictionary for Regulatory Activities

MT mid-turbinate

NAI neuraminidase inhibitor

OST oseltamivir

PB2 polymerase basic protein 2 PCR polymerase chain reaction PD pharmacodynamic(s)

PGIC Patient Global Impression of Change PGIS Patient Global Impression of Severity

PK pharmacokinetic(s)
PP Per Protocol
PT preferred term

qRT-PCR quantitative real time polymerase chain reaction

SAE serious adverse event
SAP statistical analysis plan
SBP systolic blood pressure
SDTM Study Data Tabulation Model

SI international system SOC standard-of-care

TEAE Treatment-emergent adverse event

 $T_{max}$  Time to reach  $C_{max}$  VAS visual analogue scale

#### 1. INTRODUCTION

This statistical analysis plan (SAP) contains definitions of analysis sets, derived variables and statistical methods for the analysis of efficacy and safety of the investigational compound pimodivir (JNJ-63623872). Separate documents for mock shells and table of contents for TFLs (DPS) are also produced. The SAP is to be interpreted in conjunction with the protocol.

Pimodivir (formerly known as VX-787 and JNJ-63623872) is a non-nucleotide inhibitor of the polymerase basic protein 2 (PB2) subunit of the influenza A virus polymerase complex and is currently in Phase 3 development as a treatment for influenza A infection.

# 1.1. Trial Objectives

#### **Primary Objective**

The primary objective is to evaluate superiority of pimodivir in combination with standard-of-care (SOC) treatment compared to placebo in combination with SOC treatment, with respect to the time to resolution of influenza-related symptoms.

### **Secondary Objectives**

The secondary objectives are:

- To investigate the safety and tolerability of pimodivir in combination with SOC treatment compared to placebo in combination with SOC treatment.
- To evaluate superiority with respect to the hospital admission rate 28 days after initiation of treatment in the pimodivir in combination with SOC treatment arm, compared to the placebo in combination with SOC treatment arm.
- To evaluate superiority with respect to the incidence of complications associated with influenza after the start of study treatment in the pimodivir in combination with SOC treatment arm, compared to the placebo in combination with SOC treatment arm.
- To investigate time to resolution of each of the 10 individual influenza-related symptoms as assessed by the PRO measure Flu-iiQ<sup>TM</sup>.
- To investigate the time to return to daily activities as assessed by the subject in the pimodivir in combination with SOC treatment arm, compared to the placebo in combination with SOC treatment arm.
- To investigate the time to resolution of fever in the pimodivir in combination with SOC treatment arm, compared to the placebo in combination with SOC treatment arm.
- To investigate all-cause mortality in the pimodivir in combination with SOC treatment arm, compared to the placebo in combination with SOC treatment arm.
- To assess the pharmacokinetics (PK) of pimodivir and to explore the PK/pharmacodynamic (PD) relationships of pimodivir for efficacy and safety.
- To investigate the acceptability (taste and swallowability) of the pimodivir formulation in adolescents.

- To investigate the emergence of viral resistance against pimodivir detected by genotyping and/or phenotyping.
- To evaluate superiority with respect to time to viral negativity in the pimodivir treatment arm compared to the control arm by quantitative real time polymerase chain reaction (qRT-PCR) and viral culture.

### 1.2. Trial Design

This is a Phase 3, randomized, double-blind, placebo-controlled, multicenter study to evaluate the efficacy and safety of pimodivir in combination with SOC treatment versus placebo in combination with SOC treatment in adolescent (13 to 17 years), adult (18 to 65 years), and elderly (>65 to ≤85 years) non-hospitalized subjects with influenza A infection who are at risk of developing complications. A target of 720 subjects will be randomly assigned in this study with 360 subjects planned per treatment arm. The aim is to enroll a minimum of 72 adolescent subjects in this study in selected countries and study sites consistent with local regulations. The target population of the study are influenza-infected, non-hospitalized subjects who, due to their age (65 to 85 years) or underlying comorbidities (regardless of age), are at increased risk of developing influenza-related complications. The randomization will be stratified by type of baseline SOC (including or not including antiviral treatment) and time since onset of symptoms (first administration of study drug ≤48 hours or >48 hours since onset of influenza symptoms). The study population should consist of at least 60% of subjects with first administration of study drug ≤48 hours since onset of influenza symptoms.

Subjects who meet all eligibility criteria will be randomized in a 1:1 ratio to receive 1 of the following 2 treatments:

- Treatment Arm 1: pimodivir 600 mg bid for 5 days + SOC treatment\*
- Treatment Arm 2: pimodivir placebo bid for 5 days + SOC treatment\*

\* SOC treatment will be determined by the investigator based on local practice, and may include influenza antivirals and/or supportive care only. The choice to use influenza antivirals as part of the SOC should be made before randomization. The influenza antiviral should be started no later than Day 2 morning (up to noon). An influenza antiviral as part of the SOC cannot be changed (eg, switching one influenza antiviral for another) during the treatment period, with the exception that an influenza antiviral may be discontinued in the case of a suspected adverse event (AE).

# 1.3. Statistical Hypotheses for Trial Objectives

The time to resolution of the 7 primary influenza-related symptoms, as assessed by a PRO measure (Flu-iiQ<sup>TM</sup>), with pimodivir in combination with SOC treatment is statistically superior to treatment with placebo in combination with SOC treatment in subjects with influenza A infection who are at risk of developing complications.

### 1.4. Sample Size Justification

The study will aim to enroll 720 subjects, with 360 subjects per treatment arm.

The sample size is based on the primary endpoint of time to resolution of influenza-related symptoms. Time to resolution of influenza-related symptoms, ie, the proposed primary endpoint, will be based on the subjects' ratings on 7 items from the symptoms domain of the Flu-iiQ<sup>TM</sup> (cough, sore throat, headache, nasal congestion, feeling feverish, body aches and pains, and fatigue).

For the sample size, it is assumed that the recovery time is distributed similar to the time of symptom recovery in uncomplicated influenza, albeit with a somewhat longer average time to recovery due to the increased risk for complications and the increased time to recover for this population.

An underlying log-logistic distribution of the recovery time is assumed with a scale parameter of 0.55 and an intercept of 5.0 (in hours). Using the Gehan-Wilcoxon test to analyze the data and based on the assumption that the time to recovery is improved with 25%, a sample size of 600 subjects (randomized 1:1) will have an estimated power of 90% as based on 10,000 simulations. It is expected that approximately 15% of the total enrolled subjects may not be centrally-confirmed influenza A positive, resulting in a total of 720 subjects to be enrolled.

The effect of different distributional assumptions has been assessed, using estimates of the intercept and scale parameter from the accelerated failure time (AFT) model of time to resolution of influenza symptoms for both the log-logistic and log-normal distributions, based on data from the pimodivir Phase 2 Study 63623872FLZ2001. These estimates are provided in Table 1. The scale parameter is a measure for variability of the recovery times. The intercept is a constant that cancels out in effect size estimation/simulations.

Table 1: Estimates of Intercept and Scale Parameter From Study 63623872FLZ2001

| Model | Parameter | Estimate | 95% CI |
|--------------|-----------|----------|------------------|
| Log-logistic | Intercept | 3.8546 | (3.2000, 4.5092) |
| | Scale | 0.5213 | (0.4633, 0.5867) |
| Log-normal | Intercept | 3.6277 | (2.8897 4.3656) |
| | Scale | 0.9880 | (0.8919 1.0945) |

For a trial with a sample size of 600 patients, recovery times were simulated based on the log-logistic model and separately also based on the log-normal distribution, assuming that the time to recovery is reduced by 25% in the pimodivir with SOC treatment arm compared to the placebo with SOC treatment arm, and that the subjects are randomized in a 1:1 ratio between the 2 treatment groups. To consider the variability in the intercept and scale parameters, the simulated recovery times were derived using the estimate of each parameter and using the upper limit of the 95% confidence interval (CI) for each parameter. A trial was simulated 10,000 times.

The Gehan-Wilcoxon test, log-logistic AFT model, and log-normal AFT model were used to analyze each of the 10,000 simulated datasets, for each recovery time distribution (log-logistic, log-normal) and for each parameter estimate (estimate, upper limit of the 95% CI). The power, for each statistical test, was estimated as the number of datasets where the 1-sided p-value from the test was <0.025 out of the 10,000 simulated datasets.

Table 2 provides the estimates of power for each statistical test and simulated time to resolution of influenza symptoms distributions.

**Table 2:** Estimated Power From 3 Statistical Tests

| | | Estimated Power (%) | |
|---|---|---|---|
| Simulated Distribution of Recovery Time | Gehan-Wilcoxon | AFT Log-logistic Model | AFT Log-normal Model |
| Log-logistic (estimate) | 97.3 | 97.3 | 96.2 |
| Log-logistic (upper CL) | 93.3 | 93.4 | 91.3 |
| Log-normal (estimate) | 93.7 | 94.2 | 94.8 |
| Log-normal (upper CL) | 88.3 | 89.1 | 89.6 |

For the simulated recovery times based on the log-logistic model, the estimated power was greater than 90% when using both the estimate and the upper limit of the 95% CI for the intercept and scale parameter from the Phase 2 study.

For the simulated recovery times based on the log-normal model, the estimated power was greater than 90% and greater than 85% when using the estimate and the upper limit of the 95% CI, respectively, for the intercept and scale parameters from the Phase 2 study.

The sample size considerations are not based on accrual time and estimates of median survival times because all patients will have the same follow-up time by study design (28 days) and censoring is independent from time point of enrollment in the study, making accrual time not a concern. Also, the treatment effect is expressed as a 25% improvement (reduction) in time to resolution of influenza symptoms, and therefore does not require median times for sample size and power calculations.

#### 1.5. Randomization and Blinding

#### **Treatment Allocation: Procedures for Randomization**

Central randomization will be implemented in this study. Subjects will be randomly assigned to 1 of 2 treatment arms in a 1:1 ratio based on a computer-generated randomization schedule prepared before the study by or under the supervision of the sponsor. The randomization will be balanced by using randomly permuted blocks and will be stratified by type of baseline SOC (including or not including influenza antiviral treatment) and time since onset of symptoms (first administration of study drug  $\leq$ 48 hours or >48 hours since onset of influenza symptoms). The interactive web response system (IWRS) will assign a unique treatment code, which will dictate the treatment assignment and matching study drug kit for the subject. The requestor must use his or her own user identification and personal identification number when contacting the IWRS, and will then give the relevant subject details to uniquely identify the subject.

#### **Blinding**

The investigator will not be provided with randomization codes. The codes will be maintained within the IWRS, which has the functionality to allow the investigator to break the blind for an individual subject.

Data that may potentially unblind the treatment assignment (ie, study drug plasma concentrations) will be handled with special care to ensure that the integrity of the blind is maintained and the potential for bias is minimized. This can include making special provisions, such as segregating the data in question from view by the investigators, clinical team, or others as appropriate until the time of database lock and unblinding.

Under normal circumstances, the blind should not be broken until all subjects have completed the study and the database is finalized. Otherwise, the blind should be broken only if specific emergency treatment/course of action would be dictated by knowing the treatment status of the subject. In such cases, the investigator may in an emergency determine the identity of the treatment by contacting the IWRS. It is recommended that the investigator contact the sponsor or its designee if possible to discuss the particular situation, before breaking the blind. Telephone contact with the sponsor or its designee will be available 24 hours per day, 7 days per week. In the event the blind is broken, the sponsor must be informed as soon as possible. The date, time, and reason for the unblinding must be documented in the IWRS, in the appropriate section of the electronic case report form (eCRF) and in the source documents. The documentation received from the IWRS indicating the code break must be retained with the subject's source documents in a secure manner.

#### 2. GENERAL ANALYSIS DEFINITIONS

All analysis dataset preparations and statistical analyses will be performed using SAS® version 9.2 or higher.

### 2.1. Visit Windows, Phase Definitions and Baseline

The study is set up as shown in Figure 1. The phases will be constructed as shown in Table 3.

Figure 1: Study time line.

| Day | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 14 | 28 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm 1 | Scr. | | Pimod<br>+ So | | 00 mg<br>eatmei | | Follow-up | | | | | | |
| Arm 2 | Scr. | | | ebo bio<br>treatm | d + SO<br>nent | )C | | | | F | ollow-up | | |

Note: Depending on the time of screening/enrollment, subjects will receive 1 dose (evening) or 2 doses (morning and evening) of study drug on Day 1. For subjects who receive only 1 dose of pimodivir or placebo on Day 1 (evening), dosing should continue until the morning of Day 6 so that all subjects receive 10 doses in total.

#### 2.1.1. Phase Definitions

**Table 3: Construction of phases** 

| Trial phase | Start date | End date |
|---|---|---|
| Screening (phase 1) | The date of signing the informed consent with 00:00 as a time part | 1 minute before the first study drug intake |
| Treatment (phase 2) *1 | Datetime of first study drug intake*2 | Datetime of last investigational medication intake*2 + 24 hours |
| Follow-up (phase 3) | End of the treatment phase +1 minute | Trial termination date (or date of last contact if later) |

<sup>\*1:</sup> A treatment period will be constructed in the derived datasets with the same start and end date as the treatment phase.

Additionally the treatment phase and follow-up phase will be combined in the analysis.

In case the time part of first medication intake is missing the randomization time will be used, if available. If the randomization time is also missing then the time part of first medication intake will be imputed with 8:00 if the first medication was taken in the morning or with 20:00 if the first medication was taken in the evening. In case the time of the last medication intake is missing, the time part will be imputed with 8:00 if the last medication was taken in the morning or with 20:00 if the last medication was taken in the evening.

The last phase, whichever it is for a subject, always ends on 23:59 of the day of trial termination (or date of last contact if later).

Assessments will be assigned to phases based on their start datetime, but seconds will not be taken into account. If only one assessment is expected per day and the day part of the start date of the assessment is present but the time part is missing, the assessment will be treated as if it happened

<sup>\*2:</sup> In case the time part of the medication intake is missing the imputed time part will be used as described below.

at 00:00 of the day of the assessment (except for Adverse Events see details in Section 7.1). No imputations on missing times/time parts will be made in the analysis datasets.

In case more than one assessment per day is expected and the time part is missing:

- 1. Allocate according to the timepoint: Morning=00:00, Evening=20:00
- 2. If 1 timepoint is missing on day x: Check the non-missing timepoint of the other record on this day x. Allocate this record to the timepoint of day x that is not already covered. Then apply 1.
- 3. If both timepoints are missing on day x: Allocate using the values of XXSPID, ie, lowest number is morning, highest number is evening. Then apply 1.

# 2.1.2. Analysis visits

In general, AVISIT will be derived as the day of a scheduled visit, assessment or self-assessment as recorded in the respective SDTM, including the safety follow-up visit and the Day 28 final study visit (eg, 'Day 4'). AVISITN will be the numeric counterpart (eg, for 'Day 4' AVISITN will be 4). The AVISIT for scheduled measurements before first intake will be set to 'Screening' with AVISITN = -1. For specifications on the baseline record and endpoint record see Section 2.5.

For post-baseline assessments of the Flu-iiQ<sup>TM</sup>, Temperature (as recorded by the subject on the ePRO device), Daily Activities Resumption (Return to daily activity), Patient Global Impression of Severity (PGIS), Patient Global Impression of Change (PGIC) and the European Quality of Life 5 Dimensions (EQ-5D) questionnaires, AVISIT and AVISITN will be derived from the number of days in the study relative to the start of study treatment (reldy, see Section 2.4). Post-baseline assessments taken from 00:00 until 02:00 will be assigned to the day before (eg, a recording on Day 4 at 01:00 will be assigned AVISIT= Day 3).

## 2.1.3. Analysis timepoints

In general, for parameters that were assessed more than once daily, the analysis time point (ATPT) will be the time point as reported in the database.

For the PRO assessments of the FLU-iiQ<sup>TM</sup> and temperature all post-baseline records from day 1, 02:01 onwards will be assigned to an analysis time point (ATPT) using the following windows: morning = from 02:01 until 14:00 and evening = from 14:01 until 02:00. The measurements taken from 00:00 until 02:00 will be assigned to the evening of the day before (eg, a recording on Day 4 at 01:00 will be assigned AVISIT= Day 3, ATPT=Evening).

## 2.1.4. Use of records per analysis visit and timepoint

To ensure only one record is used per analysis visit and timepoint for the PRO assessments of the FLU-iiQ<sup>TM</sup> only one questionnaire (collection of questions answered on the same datetime) per analysis visit and timepoint should be selected for analysis. The selected questionnaire will be used for all analyses of all modules of the FLU-iiQ<sup>TM</sup> questionnaire. The following rules should be followed to select the questionnaire. Only questionnaires for which 50% of the items are available to construct a Composite symptom score are considered.

1. Determine the maximum score of the individual 7 primary influenza-related symptoms per questionnaire and select the questionnaire with the highest maximum score on an individual question.

- 2. If more than one questionnaire is still selected, the questionnaire which yields the highest composite symptom score based on 7 primary influenza-related symptoms within an analysis visit and timepoint is used.
- 3. If more than one questionnaire is still selected, the questionnaire latest in time is used.
- 4. If more than one questionnaire is still selected, the questionnaire with the highest sequence number is used.

To ensure only one record is used per analysis visit for the Return to daily activity and PGIS questionnaires only one questionnaire should be selected for analysis. Following rules should be followed to select the questionnaire.

- 1. The questionnaire latest in time is used.
- 2. If more than one questionnaire is still selected, the questionnaire with the highest sequence number is used.

To ensure only one record is used per analysis visit for the PGIC and EQ-5D questionnaires the following rules should be followed to select the questionnaire.

Listed below (Table 4) are the visit windows and the target days for each visit where PGIC and EQ-5D are recorded. The reference day is Study Day 1, the date of first intake of study drug.

- 1. If a subject has 2 or more actual visits in one visit window, the visit closest to the target day will be used as the protocol visit for that visit window.
- 2. If 2 actual visits are equidistant from the target day within a visit window, the later visit is used.

Table 4: Visit Windows for PGIC and EQ-5D

| Scheduled Visit<br>Number | Time Interval (label on output) | Time Interval (Day)* | Target Time Point (Day) |
|---|---|---|---|
| 6 | Day 6 | [2 to 10] | 6 |
| 14 | Day 14 | [11 to 20] | 14 |
| 28 | Day 28 | [21 to 38] | 28 |

<sup>\*</sup>Relative to Study Day 1

To ensure only one record is used per analysis visit and analysis timepoint for the temperature, the following rules should be followed to select the temperature measurement.

- 1. The measurement with the highest temperature is used.
- 2. If more than one measurement is still selected, the measurement latest in time is used.
- 3. If more than one measurement is still selected, the measurement with the highest sequence number is used.

#### 2.1.5. Unscheduled Assessments

In general, all scheduled assessments after first administration of study drug will be used. Unscheduled assessments will not be used in descriptive statistics or any per-time point analysis, but will be shown in listings as applicable. Pre-dose unscheduled assessments will be taken into

account for baseline determination and post first dose unscheduled assessments will be taken into account for worst-case determination.

For PRO assessments, both scheduled and unscheduled assessments will be taken into account to determine which assessment will be used per analysis visit/timepoint as described in Section 2.1.4.

For the time to response endpoints, recordings taken at unscheduled visits will be taken into account.

### 2.2. Analysis Sets

### 2.2.1. All Randomized Analysis Sets

### 2.2.1.1. All Randomized Analysis Set (RAND)

All randomized subjects with a randomization date time at or before the date time of first intake of study drug, or with a randomization date time and no study drug intake.

# 2.2.1.2. Randomized and/or Treated Analysis Set (RT)

All randomized subjects and/or all subjects who received at least 1 dose of study drug. The Randomized and/or Treated Analysis Set (RT) will be used in all listings unless specified otherwise for a specific display.

## 2.2.2. Efficacy Analysis Sets

Efficacy will be analyzed on the intent-to-treat infected (ITT-i) set and by randomized treatment. The primary efficacy endpoint will also be analyzed on the Per Protocol set. The primary efficacy endpoint and the two most important secondary endpoints (ie, 'Incidence of treatment-emergent adjudicated influenza complications' and 'Incidence of hospital admission 28 days after treatment initiation') will also be analyzed on the intent-to-treat non-infected (ITT-ni) set and by randomized treatment.

### 2.2.2.1. Intent-To-Treat infected (ITT-i) set

All subjects from the RAND analysis set who receive at least 1 dose of study drug and who have a confirmed infection with influenza A. Confirmation of influenza A infection will be obtained from virology data. If there are no virology data available at final analysis, then a subject will be excluded from the ITT-i set.

A subject is considered to have a confirmed infection with influenza A if he/she has:

• at least one positive PCR result from central lab testing at baseline or pre-baseline;

else

• at least two positive PCR results from central lab testing post-baseline.

Note: viral load (PCR) results from central lab testing recorded as 'TARGET NOT DETECTED' will be considered as negative, all other non-missing results as positive.

Note: if no viral load measurement is available prior to first dose of study drug, then the first result from the central lab testing obtained up to and including 30 minutes after first dose of study drug will be considered as the baseline assessment.

Note: viral load results from central lab testing obtained from leftover samples from the local virology test will be considered in determining confirmed infection with influenza A.

# 2.2.2.2. Per Protocol Set (PP)

All subjects in the ITT-i set without major protocol deviations that may have an impact on the efficacy analysis.

Decisions regarding which subjects are included in the per protocol set will be made before database lock on the following criteria. Subjects will be included in the PP set in case:

- Subjects missed at most 3 doses in total or at most 2 consecutive doses. On the day of randomization or the next day at least one dose needs to be taken.
- The actual treatment must be the same as the planned treatment
- No unblinding may have taken place
- Subjects may not violate inclusion criteria 2, 3, 5, and 12 and exclusion criteria 1, 6, 9, 12, and 13. For details of these in/exclusion criteria refer to Table 5.
- Screening PRO assessments (Pre-existing Symptom Questionnaire and Flu-iiQ<sup>TM</sup> Module 1) performed on the ePRO device before randomization.
- Completed the pre-existing symptoms questionnaire and have at least 3 post-baseline FluiiQ<sup>TM</sup> measurements.
- Influenza antiviral as part of the SOC was started no later than Day 2 morning.
- Subjects did not switch to another influenza antiviral as a part of the SOC during the treatment period.

Table 5: Details of inclusion and exclusion criteria to be fulfilled for inclusion in the per protocol analysis set

| Inclusion/ | Criterion | Description |
|---|---|---|
| Exclusion | number | |
| Inclusion | 2 | Present to the clinic with symptoms suggestive of a diagnosis of acute influenza and have at least 1 respiratory symptom and at least 1 systemic symptom, both scored as at least 'moderate' if the symptom did not pre-exist before influenza onset, or scored worse than usual if the symptom pre-existed as determined by subject's ratings on Module 1 of the Flu-iiQ <sup>TM</sup> and the Pre-existing Symptom Questionnaire in the ePRO device. Symptoms must include the following by category: 1. Respiratory symptoms: cough, sore throat, nasal congestion, 2. Systemic symptoms: headache, body aches or pain, feverishness, fatigue. |
| Inclusion | 3 | Tested positive for influenza A infection after the onset of symptoms, using a rapid influenza diagnostic test (RIDT) or, if available, a PCR-based or other rapid molecular diagnostic assay. |
| Inclusion | 5 | Enrollment and initiation of study drug treatment ≤72hours after onset of influenza symptoms. |
| Inclusion | 12 | Subjects 13 to 65 years of age, inclusive must also have at least one of the following: a. Cardiovascular or cerebrovascular disease (including congenital heart disease, chronic heart failure, coronary artery disease, or stroke: excluding isolated hypertension) b. Chronic lung disease (eg, asthma, chronic obstructive lung disease [COPD] or cystic fibrosis) |

 $CONFIDENTIAL-FOIA\ Exemptions\ Apply\ in\ U.S.$ 

| Inclusion/ | Criterion | Description |
|---|---|---|
| Exclusion | number | |
| | | c. Weakened immune system due to disease or medication (eg, subjects with human |
| | | immunodeficiency virus [HIV], cancer, or chronic liver or kidney disease |
| | | [presence of kidney damage for > 3 months, defined by structural or functional |
| | | abnormalities of the kidney, with or without decreased GFR manifested by: |
| | | pathological abnormalities; OR markers of kidney damage, including |
| | | abnormalities in the composition of the blood or urine or abnormalities in |
| | | imaging tests], or subjects taking chronic systemic steroids). |
| Exclusion | 1 | Received more than 1 dose of influenza antiviral medication (eg, OST or zanamivir), or |
| | | any dose of ribavirin within 2 weeks, prior to first study drug intake, or received IV |
| | | peramivir more than 1 day prior to screening. |
| Exclusion | 6 | Severely immunocompromised in the opinion of the investigator (eg, known cluster of |
| | | differentiation 4 <sup>+</sup> [CD4 <sup>+</sup> ] count <200 cells/mm <sup>3</sup> , absolute neutrophil count <750/mm <sup>3</sup> , |
| | | first course of chemotherapy completed within 2 weeks prior to screening, history of |
| | | stem cell transplant within 1 year prior to screening, history of a lung transplant). |
| Exclusion | 9 | Taken any disallowed therapies before the planned first dose of study drug. |
| Exclusion | 12 | Subject has any condition that could prevent, limit, or confound the protocol-specified |
| | | assessments (eg, subject is unable to swallow tablets, unable to complete PROs, or is |
| | | illiterate), or in the opinion of the investigator, participation would not be in the best |
| | | interest of the subject (eg, compromise the well-being). |
| Exclusion | 13 | |
| | | abnormalities, ECG findings, or physical examination findings that, in the opinion of the |
| | | investigator, would place the subject at an unreasonably increased risk through |
| | | participation in this study. The investigator should consider the laboratory parameter |
| | | criteria for study drug discontinuation when screening a subject for enrollment. |

# 2.2.2.3. Intent-To-Treat non-infected (ITT-ni) Set

All subjects from the RAND analysis set who receive at least 1 dose of study drug and who do not have a confirmed infection with influenza A.

# 2.2.3. Safety Analysis Set

# 2.2.3.1. Safety Set or All Subjects Treated (AST)

All safety endpoints will be evaluated on the Safety population, consisting of all subjects who received at least one dose of study drug and will be analyzed by treatment arm as treated.

# 2.2.4. Pharmacokinetics (PK) Analysis Set

The PK analysis set is defined as subjects who have received at least 1 dose of pimodivir and have at least 1 valid blood sample drawn for PK analysis.

# 2.2.5. Pharmacodynamics (PD) Analysis Set

The PD analysis set is defined as all subjects in the PK analysis set for whom at least one PK parameter could be derived.

# 2.3. Definition of Subgroups

See Table 6 for the definitions of all the subgroups. The third column in the table indicates for which endpoints the subgroup is applied.

Descriptive statistics will be produced for the different subgroups.

In demographics and baseline disease characteristics, the following subgroups will be used:

- Region
- Influenza A subtype category
- Age group
- Time since onset of influenza symptoms (actual)
- Type of SOC at baseline (actual)
- Influenza season
- Study period
- Baseline resistance
- Any baseline polymorphism
- COVID-19 impacted

Stratification factors (actual) will be used as subgroups for concomitant medication.

For the primary and two most important secondary endpoints (ie, 'Incidence of treatment-emergent adjudicated influenza complications' and 'Incidence of hospital admission 28 days after treatment initiation') the subgroup with subgroup\*treatment interaction term will be added in the statistical analysis models, except for the study period subgroup, where the analysis will be performed separately for each individual category of the subgroup. For further details see Section 5.2.3 and Section 5.3.2. For other endpoints, the statistical analysis will be performed separately for each individual category of the subgroup.

Table 6: Subgroups with their definition

| Subgroup | Definition | Endpoints |
|---|---|---|
| Region | Based on country according to UN classification of Geographic regions <sup>[5]</sup> : • Europe/Africa • Northern-America • Latin America and the Caribbean • Asia and Oceania | - Efficacy (primary and secondary<br>endpoints, excluding viral kinetics<br>endpoints) |
| Age group (years) Type of SOC at baseline (actual) | <ul> <li>13-17 years</li> <li>18-65 years</li> <li>66-85 years</li> <li>SOC including influenza antiviral treatment</li> <li>SOC not including influenza antiviral treatment</li> </ul> | - Efficacy (primary and secondary endpoints, excluding viral kinetics endpoints) - All safety - All efficacy - Viral phenotype - Viral genotype - Safety (AE summary, AEs and SAEs by MedDRA system organ class and preferred term, influenzarelated complications, laboratory toxicity) |
| Time (hours)<br>from onset<br>influenza<br>symptoms to | <ul><li>≤48 hours</li><li>&gt;48 hours</li></ul> | - All efficacy<br>- Viral phenotype<br>- Viral genotype |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| Subgroup | Definition | Endpoints |
|---|---|---|
| first study drug | | • |
| intake (actual) | | |
| Influenza A | • A/H1N1 | - Efficacy (primary and two most |
| subtype | • A/H3N2 | important secondary endpoints |
| category | Other | only) |
| | | - All viral kinetics |
| | | - Viral phenotype |
| Baseline | Polymorphism on one or any of these amino-acid | - Viral genotype - Efficacy (primary endpoint only) |
| polymorphism | positions of interest: | - All viral kinetics |
| (based on | • Q306 | - Viral phenotype |
| influenza PB2 | • F323 | - Viral genotype |
| genotype) | • S324 | |
| | • F325 | |
| | • S337 | |
| | • H357 | |
| | • F363 | |
| | • K376 | |
| | • T378 | |
| | • F404 | |
| | • Q406 | |
| | • M431 | |
| - · | • N510 | 707 |
| Baseline | Based on fold change (FC) in EC <sub>50</sub> for pimodivir: | - Efficacy (primary endpoint only) |
| resistance | • FC ≤4 | - All viral kinetics |
| (based on influenza PB2 | • FC >4 | - Viral phenotype<br>- Viral genotype |
| phenotype) | | - virai genotype |
| Baseline Fever | Baseline (temperature ≥37.0°C) as recorded as part of the vital signs assessment | - Resolution of fever only |
| Influenza season | Northern Hemisphere 2017/2018 | - Efficacy (primary and two most |
| | Southern Hemisphere 2018 | important secondary endpoints |
| | Northern Hemisphere 2018/2019 | only) |
| | Southern Hemisphere 2019 | - All viral kinetics |
| | Northern Hemisphere 2019/2020 | - Viral phenotype |
| | Southern Hemisphere 2020 | - Viral genotype |
| | and so on, to capture all enrolled subjects | |
| Study period | • Pre interim (subjects enrolled for the interim analysis, ie randomized before or on February 28, 2020) | - Efficacy (primary and two most important secondary endpoints only) |
| | • Post interim (subjects enrolled after the interim | - Safety (AE summary, AEs and |
| | analysis, ie randomized after February 28, | SAEs by MedDRA system organ |
| | 2020) | class and preferred term, influenza- |
| | | related complications, laboratory |
| COVID-19 | • Yes | toxicity) - Efficacy (primary and two most |
| impacted | • Yes • No | important secondary endpoints |
| impacied | • INO | only) |
| | | - Safety (AE summary, AEs and |
| | | SAEs by MedDRA system organ |
| | | class and preferred term, influenza- |
| | | related complications, laboratory |
| | | toxicity) |

25

Influenza season is defined as follow:

Subjects enrolled from 1<sup>st</sup> October 2017 to 31<sup>st</sup> March 2018 are considered to be in the Northern Hemisphere 2017/2018 category and subjects enrolled from 1<sup>st</sup> April 2018 to 30<sup>th</sup> September 2018 are considered to be in the Southern Hemisphere 2018 category. Subjects enrolled from 1<sup>st</sup> October 2018 to 31<sup>st</sup> March 2019 are considered to be in the Northern Hemisphere 2018/2019 category and subjects enrolled from 1<sup>st</sup> April 2019 to 30<sup>th</sup> September 2019 are considered to be in the Southern Hemisphere 2019 category, and so on.

A subject is considered to be impacted by the COVID-19 pandemic if they experienced at least one of the following:

- discontinued from the study (or study drug) due to COVID-19
- had a COVID-19 related AE
- had a COVID-19 related protocol deviation (major or minor)

Additional subgroup analysis may be specified in a separate analysis plan and reported separately from the clinical study report.

# 2.4. Study Day and Relative Day

Reference date refers to the start date of the first study drug administration. All efficacy and safety assessments at all visits will be assigned a day relative to this date.

The relative day (reldy) will be defined as:

 $reldy = visit \ date - reference \ date + 1$  for visits on or after the reference date,

 $reldy = visit \ date - reference \ date$  for visits before the reference date.

Consequently there is no 'day 0' defined.

# 2.5. Baseline and Endpoint

The baseline analysis visit is defined as the last assessment before the first intake of the study drug, with the possible exception for height, weight, and virology results from central lab testing. Height and weight are only recorded once, at the screening/baseline visit, and the values recorded at this visit will be allocated to the baseline analysis visit irrespective of start of study drug. For the virology parameters, if no measurement is available prior to first dose of study drug, then the first result from central lab testing obtained up to and including 30 minutes after first dose of study drug will be considered as the baseline assessment and will be flagged in the analysis dataset.

As specified in the protocol, an ECG recording within 1 calendar day before signing of the informed consent form (ICF/assent form) can be used as baseline ECG requirement, if no ECG measurement was performed between signing ICF and first study drug intake.

For programming purposes, the baseline record will be doubled in the ADAM datasets, the doubled record will be renamed with AVISIT = 'Baseline', AVISITN = 0 and will be assigned to the treatment phase.

For viral phenotyping, the last visit (Endpoint) is defined as the last study visit/timepoint for which an EC<sub>50</sub> and/or IC<sub>50</sub> result is available (including unscheduled visit results).

For vital signs, ECG and central laboratory data the last study visit (Endpoint) is defined as the last scheduled study visit/timepoint and will be either the final study visit (at Day 28) or the safety follow-up visit.

#### 2.6. Other Definitions

For FDA marketing authorization approval in the US all subjects will be included in the analysis.

The oseltamivir subset (OST subset) contains only those subjects whose SOC treatment contains oseltamivir (OST). The first dose of OST may be given before the subject was randomized but should be started no later than Day 2 morning (up to noon). The complete analysis will be repeated restricted to the OST subset to support marketing authorization approval in EMA.

Analyses to support authorization approval in other regions or countries will include all subjects unless the Health Authority of the region or country requests otherwise and may be specified in a separate analysis plan and may also be reported separately.

#### 3. INTERIM ANALYSIS AND DATA MONITORING COMMITTEE REVIEW

# 3.1. Interim Analysis

An interim analysis will be implemented to re-estimate the study sample size and to perform an assessment of futility. The maximum total number of subjects that may be enrolled in the study will be approximately 1,080. This interim analysis will be implemented through an IDMC, providing recommendations to a Sponsor Committee. Only the IDMC and the independent Statistical Support Group will be unblinded to the data. Details will be specified in the IDMC charter.

Details on the statistical decision rules will be provided in the IDMC SAP. The interim analysis will be conducted at the end of the first influenza season when between 360 and 540 subjects have been enrolled or during the season when 540 subjects have been enrolled. Further details will be specified in the IDMC charter.

# 3.2. Independent Data Monitoring Committee

An IDMC will be established to monitor data on a regular basis. The committee will meet periodically to review interim data. After the review, the IDMC will make recommendations regarding the continuation of the study. The details will be provided in a separate IDMC charter.

The IDMC will consist of at least 3 members, including one medical expert in the relevant therapeutic area and at least one statistician knowledgeable about statistical methods for clinical studies and sequential analysis of study data. One of these individuals will chair the Committee. The IDMC responsibilities, authorities, and procedures will be documented in its charter.

#### 4. SUBJECT INFORMATION

All general analyses will be done on the ITT-i Set and the Safety Set unless specified otherwise for a specific display.

### 4.1. Demographics and Baseline Characteristics

Demographics and baseline disease characteristics will also be done on the PP and ITT-ni sets. Descriptive statistics or frequency tabulation will be provided for the following parameters.

- Demographic parameters:
  - Sex (Male, Female)
  - Race (White, Black or African American, Asian, American Indian or Alaska Native, Native Hawaiian or Other Pacific Islander, Multiple). The specification of the category 'Multiple' will only be listed. The 'Not reported' category will not be added for the denominator.
  - Ethnicity (Hispanic or Latino, Not Hispanic or Latino)
  - Country
  - Geographic region (Based on country according to UN classification of Geographic regions<sup>[5]</sup>: Europe/Africa, Northern-America, Latin America and the Caribbean, Asia and Oceania)
  - Age (years and categories: 13-17 years [ $\geq$ 13 <18], 18-65 years [ $\geq$ 18  $\leq$ 65], 66-85 years [>65  $\leq$ 85])
  - Age (years and categories: Adolescents (12-17 years) [≥12 ≤17], Adults (18-64 years) [≥18 ≤64], From 65 to 84 years [≥65 ≤84], 85 years and over [≥85])
  - Weight at baseline (kg)
  - Height at baseline (cm)
  - BMI at baseline = Weight at baseline (kg) / (Height at baseline (m))<sup>2</sup> (rounded to 1 decimal. Although available in the raw data, BMI will be recalculated from last weight and height measurement before start of treatment)
  - Current Tobacco use: tobacco, cigarettes, cigars, patches/gum, pipes, E-cigarettes or equivalent, smokeless tobacco (Yes, No, Missing) Note that 'No' also includes exsmokers
  - Childbearing potential (only listed)
- Baseline disease characteristics:
  - Influenza A subtype category (A/H1N1, A/H3N2, other)
  - Baseline influenza A viral load (log10 vp/mL), assessed by qRT-PCR
  - Baseline influenza A viral titer (log10 TCID50/mL) assessed by viral culture
  - Broad respiratory panel (show the reported pathogen)
  - Baseline composite symptom score of 10 influenza-related symptoms
  - Return to daily activities questionnaire baseline category

- Patient Global Impression of Severity of Influenza symptoms at baseline
- EQ-5D VAS at baseline
- EQ-5D Valuation index at baseline
- Respiration rate at baseline (breaths/min)
- Heart rate (beats/min)
- Temperature (°C) at baseline
- qRT-PCR negativity at baseline
- Viral culture negativity at baseline
- Time since onset of influenza symptoms, as randomized ( $\leq 48$  hours, > 48 hours)
- Time since onset of influenza symptoms, actual time (hours) [the actual time will be calculated from start date and time of acute respiratory symptoms until datetime of first study drug intake, if the time is missing, the midpoint of the time interval as recorded per CRF will be used]
- Time since onset of influenza symptoms, actual time ( $\leq 48$  hours, > 48 hours)
- Type of SOC at baseline, as randomized (including or not including antiviral treatment),
- Type of SOC at baseline, actual (including or not including antiviral treatment), for the SOC including antiviral treatment the influenza antiviral will also be shown.
- SOC including oseltamivir (yes, no)
- Type of influenza A diagnostic assay (Rapid antigen-based diagnostic test, Rapid molecular diagnostic test)
- Baseline resistance
- Any baseline polymorphism

# 4.2. Disposition Information

Summaries will be provided for the following disposition information:

- Number of subjects screened, screening failures, randomized, randomized and not treated, randomized and/or treated, randomized and treated, randomized and no confirmed influenza A, ITT-i set, ITT-ni set, per protocol set, and safety set. The planned treatment arm will be shown, except for the randomized and/or treated and safety sets where the actual treatment will be shown. For the ITT-i, ITT-ni, per protocol and safety analysis sets the number (%) of subjects within that set impacted by the COVID-19 pandemic will also be presented.
- Number of subjects who completed/discontinued treatment and/or the trial, with the reasons of discontinuation.
- Kaplan-Meier curves of the time to completion or discontinuation (in days) of the treatment/trial per treatment group. Note at the final analysis all subjects will have completed or discontinued the treatment/trial and no subjects will be censored.
- Number of subjects with a visit at each scheduled analysis time point by phase.
- Number of subjects enrolled per month, quarter, season, and year of enrolment

# 4.3. Treatment Compliance

Treatment compliance for pimodivir/placebo is calculated as the actual number of doses taken, as a percentage of the planned number of doses. The actual number of doses taken will be derived from the drug accountability information (DA domain) as the difference between the amount of drug dispensed and the drug returned (in case both amounts are known), otherwise treatment compliance will be missing.

For placebo or pimodivir this number needs to be divided by 2 as the study uses 300 mg tablets. The planned number of medication is 20 tablets of placebo or pimodivir hence the planned number of doses per medication equals 10 doses. Note that the planned number of doses is irrespective of whether the subject discontinued during the treatment phase.

Dosing compliance will be summarized descriptively in the treatment phase and by discontinuing the trial during the treatment period (Yes, No).

### 4.4. Extent of Exposure

The extent of exposure (hours) is defined as datetime of last study drug intake – datetime of first study drug intake + 12 hours. Note: treatment interruptions will not be taken into account.

Extent of exposure will be summarized descriptively in the treatment phase.

#### 4.5. Protocol Deviations

The number and percentage of subjects with major protocol deviations will be tabulated overall and per coded major protocol deviation.

A listing will be made of all major protocol deviations and separately for major protocol deviations related to COVID-19 for the subjects in the safety set.

A listing will be made of minor protocol deviations related to COVID-19 for the subjects in the safety set.

Additionally, for subjects in the ITT-i set, the number and percentage of subjects with a reason for exclusion from the per protocol set will be tabulated overall and for each reason for exclusion (see Section 2.2.2.2)

A listing will also be made of all reasons for exclusion from the per protocol set for subjects in the ITT-i set.

#### 4.6. Prior and Concomitant Medications

Medications reported from 7 days before first dose of study drug and up to last contact date will be summarized by preferred term using the World Health Organization-Drug Dictionary for the ITT-i Set and the Safety Set as frequency tables in 2 parts:

1. Prior medication: medication that started before the first dose of study drug, regardless of when dosing of the medication ended

2. Concomitant medication: medication received at or after the first dose of study drug, medication that was received before initial dosing and continued after initial dosing of study drug, or medication with missing stop date.

(Medication that started before the first dose of study drug and continued after the first dose of study drug will be summarized as prior medication and separately as concomitant medication.)

A frequency tabulation of concomitant medication will be shown by Anatomical Therapeutic Chemical (ATC) class level up to level 3. Frequency tabulations will be made for concomitant antibiotics, type of SOC, corticosteroids, and medication administered to treat COVID-19 infection by ATC class. Additionally, tabulations will be made of concomitant corticosteroids and antibiotics administered because of adverse events reported as influenza complications.

The ATC level 2 code J01 will be used to identify concomitant antibiotics.

The ATC level 2 code H02 and the ATC level 4 codes M01BA, R03BA, and R03AK will be used for identifying corticosteroids.

Separate frequency tabulations will be made for antipyretic medication. The ATC level 3 codes N02BA and N02BE and the generic medication names paracetamol, ibuprofen, and acetylsalicylic acid will be used to identify antipyretic medications.

If a prior/concomitant therapy record misses components of its start and/or stop dates (time and/or day and/or month and/or year), the following actions will be taken:

- 1. In case of partial start or stop date/times, the concomitant therapy records will be allocated to prior and/or concomitant using the available partial information, without imputations.
- 2. In case of a completely missing start date, the prior and/or concomitant therapy will be considered as having started before the trial.
- 3. In case of a completely missing end date, the prior and/or concomitant therapy will be considered as ongoing at the end of the trial.

# 4.7. Medical history

The influenza vaccination status will be tabulated by:

- Vaccinated in previous season, not in current season
- Vaccinated in current season, not in previous season
- Vaccinated in previous and current season.
- Not vaccinated in previous and current season

The use of antiviral influenza medication prior to the study drug initiation will be tabulated separately.

Influenza history will be listed, including information on first acute respiratory symptoms, influenza vaccination status and previous antiviral influenza therapy.

Other medical history will be tabulated by subcategory and/or will be listed.

#### 5. EFFICACY

Descriptive statistics will be used for all efficacy endpoints and will be tabulated by treatment arm and stratification factors (baseline SOC and time since onset of symptoms). For the analyses restricted to subjects who received OST as part of their SOC, type of baseline SOC will not be included as a stratification factor or model parameter.

# 5.1. Analysis Specifications

## 5.1.1. Level of Significance

As a confirmatory strategy, to account for multiplicity in the statistical evaluation of the most important efficacy endpoints, hierarchical testing will be applied to control for overall Type I error. The following endpoints are included in the confirmatory strategy:

#### **Primary Endpoint**

• Time to resolution of the 7 primary influenza-related symptoms (cough, sore throat, headache, nasal congestion, feeling feverish, body aches and pains, fatigue)

#### Secondary Endpoints

- Incidence of complications associated with influenza after the start of study treatment
- Hospital admission rates 28 days after treatment initiation

First, the primary endpoint will be tested for superiority of pimodivir in combination with SOC over placebo in combination with SOC at the 2-sided 5% significance level. If superiority is shown on the primary endpoint, the first secondary endpoint in the sequence as indicated above will be tested for superiority at the same significance level. If superiority is shown for this secondary endpoint, the second (and last) secondary endpoint in sequence will be tested. In case superiority is not shown for an endpoint, no further endpoints in the sequence will be tested for superiority.

This testing procedure will be applied on the ITT-i set.

The final analysis on the ITT-i set (to support FDA marketing authorization approval) and the final analysis on the OST subset (to support marketing authorization approval in EMA) will be performed independently, using a 5% two-sided significance level for each.

# Statistical Methodology for Evaluation at the Final Analysis

The p-values for the final analysis of the primary endpoint and the two most important secondary endpoints will be based on an inverse-normal combination test. For the primary endpoint, the p-values are obtained from the Gehan-Wilcoxon test. For incidence of complications associated with influenza after the start of study treatment and Hospital admission rates 28 days after treatment initiation the p-values will be obtained from a logistic regression model (see Sections 5.3.2 and 5.3.2.2).

All p-values below are one-sided p-values, to evaluate rejection of the null hypothesis that pimodivir is not better than placebo.

#### Let:

- p = p-value from the analysis of the 'pre interim' category of the 'study period' subgroup
- q = p-value from the analysis of the 'post interim' category of the 'study period' subgroup
- $N_1$  = actual sample size at interim, ie the number of subjects in the 'All randomized analysis set (RAND)' included in the interim analysis.
- N = per-protocol sample size (=720)
- $w_1 = \operatorname{sqrt}(N_1/N)$
- $w_2 = sqrt(1-(N_1/N))$
- $\varphi^{-1}(x)$  the inverse of the standard normal cumulative distribution function in x

The p-values resulting from the following combination test should be below the pre-specified alpha to claim superiority:

1- 
$$\varphi(C(p,q))$$
, where  $C(p,q) = w_1 * \varphi^{-1}(1-p) + w_2 * \varphi^{-1}(1-q)$ 

# 5.1.2. Data Handling Rules

For analysis purposes the log<sub>10</sub> qRT-PCR viral load will be imputed with 2.12 when the result is 'TARGET DETECTED' (ie, below limit of quantification: <2.18) and with 2.05 if result is 'TARGET NOT DETECTED' (ie, below limit of detection: <2.05). The log<sub>10</sub> TCID<sub>50</sub> viral titer will be imputed with 0.74 when the result is '<0.75' (below limit of detection and quantification).

#### 5.1.3. Stratification Factors

The actual values of the stratification factors will be used for all analyses.

The concomitant medications indicated as standard-of-care treatment on the concomitant medication form will be used for determining the actual strata for type of baseline SOC. If no influenza antiviral is recorded it will be assumed that the subject received SOC not including influenza antiviral. The following ATC level 4 code and generic medication names indicate an influenza antiviral:

- J05AH (including neuraminidase inhibitors)
- Laninamivir
- Umifenovir
- Amantadine
- Rimantadine
- Ribavirin
- Baloxavir Marboxil

The datetime when first acute respiratory symptoms appeared and the datetime of first dose of study drug will be used for determining the actual strata for time since symptom onset relative to

treatment initiation. There will be no missing stratification factor values for randomized subjects receiving study drug.

# 5.2. Primary Efficacy Endpoint(s)

#### 5.2.1. Definition

The primary efficacy analysis will be based on the ITT-i analysis set and consists of the analysis of the time to resolution of the 7 primary influenza-related symptoms.

Time to resolution of the 7 primary influenza-related symptoms (cough, sore throat, headache, nasal congestion, feeling feverish, body aches and pains, fatigue) is defined as the time in hours from initiation of study treatment to when all symptoms are considered resolved for at least 24 hours. A symptom is considered resolved, depending on pre-existence of the symptom:

- The symptom is pre-existing:
  - The symptom is considered resolved if post-baseline severity is equal or lower than the pre-existing severity
- The symptom is not pre-existing:
  - The symptom is considered resolved if its severity is scored at most mild postbaseline

A symptom is considered not pre-existing if the response to the question in the pre-existing symptoms questionnaire is 'None'. Any other non-missing response indicates that the symptom is pre-existing.

The time of resolution is the first of a successive series of 3 recordings in which all symptoms for each of the 3 assessments are considered resolved (as defined above) for all 7 primary influenza symptoms. The 3 successive recordings may have been done over 4 scheduled successive analysis timepoints, in case of 1 missing in between timepoint.

In case influenza symptoms are not resolved, data will be censored.

Censoring will be done as follows:

- 1) Last non-missing record(s) indicate resolution of influenza symptoms (but insufficient recordings to meet the time to resolution)
  - Censoring will be done at the first record of resolution from the last series of recordings of resolution of influenza symptoms
- 2) Last non-missing record does not indicate resolution of influenza symptoms
  - Censoring will be done after the last observation, which is 08:00 on the same day if the last observation was a diary entry from 00:01 until 02:00, 20:00 on the same day if the last observation was a diary entry from 02:01 until 14:00, and 08:00 the next day if the last entry was a diary entry from 14:01 until 00:00.
- 3) Additionally, in the following cases the subject will be censored using a time-to equal to the maximum time across all subjects:

- o death,
- o if a subject had not resolved the influenza symptoms at time of hospitalization and/or during hospitalization, and no further data on symptom resolution is available

Subjects not completing the pre-existing symptom questionnaire, or completing it after study day 1, will have values for each individual question imputed with the median response category of all subjects in the ITT-i set.

#### 5.2.2. Estimand

The population of interest is adolescent, adult, and elderly non-hospitalized subjects with a confirmed influenza A infection who are at risk of developing complications.

The primary variable of interest is the time to resolution (in hours) of the 7 primary influenzarelated symptoms (cough, sore throat, headache, nasal congestion, feeling feverish, body aches and pains, fatigue). Resolution is achieved if all 7 symptoms are scored as none or mild, or, are equal to or lower than the pre-influenza severity for 24 hours expressed in 3 successive recordings or 4 successive recordings where 1 in between missing recording is allowed.

The intercurrent event of use of SOC is handled in a treatment policy strategy as the primary endpoint is derived in the same way irrespective of the components of SOC, that could include influenza antivirals. For missing recordings, the composite strategy is applied. Missing recordings due to death or hospitalization are covered by using the maximum time over all subjects as the censored resolution time. Additionally, 1 missing datapoint, not due to death or hospitalization is allowed in the definition of resolution. When multiple missing recordings, not due to death or hospitalization, prevent the subject from resolving with 3 successive recordings over the full 28-day study period, censoring will be applied, but the timepoint of censoring will depend on whether the last available recording indicates resolution or not. If the last recording indicates resolution, then censoring is at the first record of resolution from the last series of recordings of resolution of influenza symptoms. If the last recording does not indicate resolution, then censoring is done at the first scheduled timepoint after the last observation.

The size of the treatment effect will be estimated by the Kaplan-Meier estimate of median time to resolution of the 7 primary influenza-related symptoms in each treatment group. A Gehan-Wilcoxon test controlling for the stratification factors will be conducted to formally compare the time to resolution of the 7 primary influenza-related symptoms between pimodivir and placebo.

### 5.2.3. Analysis Methods

The time to resolution of the 7 primary influenza-related symptoms will be estimated from a Kaplan-Meier analysis. The difference in time to resolution of the 7 primary influenza-related symptoms between treatment groups will be tested using a Gehan-Wilcoxon test controlling for the stratification factors, ie, type of baseline SOC and time since onset of symptoms.

Kaplan-Meier curves, overall and by stratum, and a stratified log-rank test will also be provided. Additionally, the data will be analyzed using an accelerated failure time model and a Cox
proportional hazards model. Both models will be adjusted for stratification factors and baseline symptom domain score.

These models are described in Section 5.3.2.

If the baseline symptom domain score is missing, then the baseline score will be imputed as the median score from all subjects in the ITT-i set.

Sensitivity analyses to account for missing assessments in the derivation of the primary endpoint will be performed to assess the robustness of the results of the primary analysis.

Three different imputation methods based on imputation of the resolution of the 7 primary influenza-related symptoms due to missing questionnaires on single timepoints will be implemented:

- 1. Impute all timepoints with missing questionnaires as resolution of the 7 primary influenzarelated symptoms, but only after the first timepoint indicating resolution after the last timepoint indicating non-resolution (no later timepoints indicate non-resolution) – and subsequently derive the primary endpoint for the patient.
- 2. Impute all timepoints with missing questionnaires as non-resolution of the 7 primary influenza-related symptoms and subsequently derive the primary endpoint for the patient.
- 3. Impute all timepoints in a consecutive series of the timepoints with a missing questionnaire as resolution of the 7 primary influenza-related symptoms, but only if this series of consecutive missing timepoints are in between 2 timepoints that indicate resolution and subsequently derive the primary endpoint for the patient.

The statistical analysis for the primary endpoint derived after applying each of the three different imputation methods will be performed.

If no Flu-iiQ<sup>TM</sup> questionnaire is completed on a calendar day this will result in having 2 missing timepoints. To assess the amount of missing data for the primary endpoint the following tables will be provided by treatment group and overall:

1. The number and percentage of subjects completing the Flu-iiQ<sup>TM</sup> questionnaires for each analysis visit up to Day 28 visit. Subjects are expected to complete the Flu-iiQ<sup>TM</sup> questionnaire twice daily. If the subject only completes the questionnaire once for a particular analysis visit, then they will be considered as completing 50% of the questionnaires for that visit. Note that the baseline visit may occur on the same day as first administration of study drug. Subsequently, if the first dose of study drug was prior to 5pm then 2 questionnaires would be expected to be completed, and if the first dose of study drug was at or after 5pm then only 1 questionnaire would be expected to be completed on analysis visit Day 1. If the baseline questionnaire was completed the day before first dose, then one baseline questionnaire and either 1 or 2 questionnaires on the

day of first dose would be expected to be completed depending on the timing of the first dose of study drug.

2. For each subject the percentage of missing Flu-iiQ<sup>TM</sup> questionnaires will be calculated as (1 - (the number of completed questionnaires until the Day 28 visit inclusive/planned number of questionnaires))\*100. The planned number of questionnaires for a particular subject is 2 times the study day of the Day 28 visit – 1, plus the number of questionnaires completed at baseline. Descriptive statistics of the percentage of missing data will be produced.

The above tables will also be produced for each subgroup.

# 5.3. Major Secondary Endpoints

#### 5.3.1. Definition

Formulae to be used for derived variables, including data conversions, are provided in the tables below.

Note that for time-to-event parameters the actual date or date times that the endpoint is met will be used. For the time-to-event parameters the subject will be censored using a time-to value equal to the maximum time across all subjects in the following cases:

- o death,
- o if a subject had not resolved the influenza symptoms at time of hospitalization and/or during hospitalization, and no further data on symptom resolution is available

# 5.3.1.1. Symptoms of Influenza (Flu-iiQ™ Module 1)

| Measurement | Formula |
|---|---|
| Time to resolution of cough (hours) [Time-to-event] | This parameter will be calculated using the symptom of cough included in Module 1 of the Flu-iiQ <sup>TM</sup> . |
| | Cough is considered resolved depending on pre-existence of the symptom. |
| | • The symptom is pre-existing: |
| | <ul> <li>The symptom is considered resolved if post-baseline<br/>severity is equal or lower than the pre-existing severity</li> </ul> |
| | • The symptom is not pre-existing: |
| | <ul> <li>The symptom is considered resolved if its severity is<br/>scored at most mild post-baseline</li> </ul> |
| | The time of resolution is the first of a successive series of 3 recordings in which the symptom for each of the 3 assessments is considered resolved (as defined above). The 3 successive recordings may have |

| | been done over 4 scheduled successive analysis timepoints, in case of |
|---|---|
| | 1 missing in between timepoint. |
| | In case the symptom is not resolved, data will be censored. |
| | Censoring will be done as follows: |
| | Last non-missing record(s) indicate resolution of symptom (but insufficient recordings to meet the time to resolution) |
| | Censoring will be done at the first record of resolution from the last series of recordings of resolution of the symptom |
| | 2) Last non-missing record does not indicate resolution of the symptom |
| | Censoring will be done after the last observation, which is 08:00 on the same day if the last observation was a diary entry from 00:01 until 02:00, 20:00 on the same day if the last observation was a diary entry from 02:01 until 14:00, and 08:00 the next day if the last entry was a diary entry from 14:01 until 00:00. |
| | 3) Additionally, in the following cases the subject will be censored using a time-to equal to the maximum time across all subjects: |
| | o death, |
| | o if a subject had not resolved the symptoms at time of hospitalization and/or during hospitalization, and no further data on symptom resolution is available |
| Time to resolution of sore throat (hours) [Time-to-event] | This parameter is defined similarly as the time to resolution of cough and will be calculated using the symptom of sore throat included in Module 1 of the Flu-iiQ <sup>TM</sup> . |
| Time to resolution of headache (hours) [Time-to-event] | This parameter is defined similarly as the time to resolution of cough and will be calculated using the symptom of headache included in Module 1 of the Flu-iiQ <sup>TM</sup> . |
| Time to resolution of nasal congestion (hours) [Time-to-event] | This parameter is defined similarly as the time to resolution of cough and will be calculated using the symptom of nasal congestion included in Module 1 of the Flu-iiQ <sup>TM</sup> . |
| Time to resolution of<br>feeling feverish<br>(hours) [Time-to-<br>event] | This parameter is defined similarly as the time to resolution of cough and will be calculated using the symptom of feeling feverish included in Module 1 of the Flu-iiQ <sup>TM</sup> . |

| Time to resolution of<br>body aches and pains<br>(hours) [Time-to-<br>event] | This parameter is defined similarly as the time to resolution of cough and will be calculated using the symptom of body aches and pains included in Module 1 of the Flu-iiQ <sup>TM</sup> . |
|---|---|
| Time to resolution of fatigue (hours) [Time-to-event] | This parameter is defined similarly as the time to resolution of cough and will be calculated using the symptom of fatigue included in Module 1 of the Flu-iiQ <sup>TM</sup> . |
| Time to resolution of neck pain (hours) [Time-to-event] | This parameter is defined similarly as the time to resolution of cough and will be calculated using the symptom of neck pain included in Module 1 of the Flu-iiQ <sup>TM</sup> . |
| Time to resolution of interrupted sleep (hours) [Time-to-event] | This parameter is defined similarly as the time to resolution of cough and will be calculated using the symptom of interrupted sleep included in Module 1 of the Flu-iiQ <sup>TM</sup> . |
| Time to resolution of loss of appetite (hours) [Time-to-event] | This parameter is defined similarly as the time to resolution of cough and will be calculated using the symptom of loss of appetite included in Module 1 of the Flu-iiQ <sup>TM</sup> . |
| Composite symptom score for systemic symptoms | The systemic symptoms included in Module 1 of the Flu-iiQ <sup>TM</sup> consist of: headache, feeling feverish, body aches and pains, fatigue, neck pain, interrupted sleep, and loss of appetite. |
| | The subject's composite symptom score for systemic symptoms per datetime is defined as the mean of the severity (0-3 scale) of the non-missing systemic symptoms for each datetime the questionnaire was filled. Note: a higher value is considered a worse value. |
| | If more than 50% of the items to construct a Composite symptom score are missing, the value for that composite score is coded as missing (ie, 4 or more items missing). |
| Composite symptom score for systemic symptoms change from baseline | Composite symptom score for systemic symptoms post-baseline value – composite symptom score for systemic symptoms baseline value. |
| Composite symptom score for respiratory symptoms | The respiratory symptoms included in Module 1 of the Flu-iiQ <sup>TM</sup> consist of: cough, sore throat, and nasal congestion. The subject's composite symptom score for respiratory symptoms per datetime is defined as the mean of the severity (0-3 scale) of the non- |

| | missing respiratory symptoms for each datetime the questionnaire was filled. Note: a higher value is considered a worse value. If more than 50% of the items to construct a Composite symptom score are missing, the value for that composite score is coded as missing (ie, 2 or more items missing). |
|---|---|
| Composite symptom score for respiratory symptoms change from baseline | Composite symptom score for respiratory symptoms post-baseline value – composite symptom score for respiratory symptoms baseline value. |
| Time to resolution of the 7 primary influenza-related symptoms considering improvement from baseline (hours) [Time-to-event] | A symptom is considered resolved depending on pre-existence of the symptom: • the symptom is pre-existing ○ If baseline response > pre-existing response, then the symptom is considered resolved if post-baseline severity is lower than the baseline severity ○ If baseline response ≤ pre-existing response, then the symptom is considered resolved if post-baseline severity is ≤ the pre-existing severity • the symptom is not pre-existing ○ The symptom is considered resolved if its severity is scored at most mild post-baseline The time to resolution will be derived in the same way as the primary endpoint (Section 5.2.1). |

# 5.3.1.2. Other Patient Reported Outcome

| Measurement | Formula |
|---|---|
| Daily activities resumption | Daily activities resumption will be assessed once daily by means of the question 'Over the past 24 hours, how much has influenza interfered with your ability to carry out your daily activities?' |
| | The responses will be dichotomized: 'Not at all' and 'A little bit' will be considered as category "returned to daily activities" and responses 'Somewhat', 'Quite a Bit' and 'Very much' will be considered in category "not returned to daily activities". |
| Time to return to daily activities (hours) [Time-to event] | The time to return to daily activities is defined as the time in hours from initiation of study treatment to the first of a successive series of 2 recordings in which the response is considered as returned to daily |

| | activities. The 2 successive recordings may have been done over 3 scheduled successive analysis timepoints, in case of 1 missing in between timepoint. |
|---|---|
| | In case the return to daily activities is not achieved, data will be censored. |
| | Censoring will be done as follows: |
| | Last non-missing record indicates return to daily activities (but insufficient recordings) |
| | Censoring will be done at the last non-missing record |
| | 2) Last non-missing record does not indicate return to daily activities |
| | Censoring will be done one day (24 hours) after the last non-missing record. |
| | The time to return to daily activities is calculated as: (Date and time of event (actual) or censoring - date and time of first dose of study drug)/3600, rounded to one decimal. |
| Patient Global<br>Impression of Severity<br>of Influenza<br>symptoms | The PGIS captures daily influenza symptom severity from the subjects' perspective per timepoint. Responses will be categorized as: "No Flu symptoms today", "Mild", "Moderate", "Severe" or "Very Severe". |
| Patient global<br>Impression of Change<br>in Influenza<br>symptoms | The PGIC <sup>[3]</sup> is aimed to capture the subject's perceptions of improvement or deterioration in the severity of influenza symptoms compared to when the subject arrived to the investigational site for influenza treatment and is done per timepoint. |
| | Categories are: "Much better", "Somewhat better", "A little better" "About the same", "A little worse", "Somewhat worse" and "Much worse". |
| EQ-5D dimension parameters: Mobility, Self-care, Usual activities, Pain/discomfort, | The EQ-5D <sup>[2]</sup> descriptive system consists of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) with 5 possible levels (no problems (level code = 1), slight problems (level code = 2), moderate problems (level code = 3), severe problems (level code = 4), extreme problems (level code = 5)). Table 7: EQ-5D Dimensions |
| Anxiety/depression | Dimension Level Interpretation |
| | 1 Mobility 1 No problems I have no problems in walking about 2 Slight problems I have slight problems in walking about 3 Moderate problems in walking about I have moderate problems in walking about |
| | 4 Severe problems I have severe problems in walking about 5 Extreme I am unable to walk about problems |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| | 2 C-16 | ٠. | NI | There are mobile and the state of the state |
|---|---|---|---|---|
| | 2 Self-care | 1 | No problems | I have no problems washing or dressing myself |
| | | 3 | Slight problems Moderate | I have slight problems washing or dressing myself I have moderate problems washing or dressing |
| | | 3 | problems | myself |
| | | 4 | Severe problems | I have severe problems washing or dressing |
| | | 4 | Severe problems | myself |
| | | 5 | Extreme problems | I am unable to wash or dress myself |
| | 3 Usual activities | 1 | No problems | I have no problems doing my usual activities |
| | | 2 | Slight problems | I have slight problems doing my usual activities |
| | | 3 | Moderate | I have moderate problems doing my usual |
| | | | problems | activities |
| | | 4 | Severe problems | I have severe problems doing my usual activities |
| | | 5 | Extreme | I am unable to do my usual activities |
| | | | problems | |
| | 4 Pain/discomfort | 1 | No problems | I have no pain or discomfort |
| | | 2 | Slight problems | I have slight pain or discomfort |
| | | 3 | Moderate | I have moderate pain or discomfort |
| | | 1. | problems | |
| | | 4 | Severe problems | I have severe pain or discomfort |
| | | 5 | Extreme problems | I have extreme pain or discomfort |
| | 5 Anxiety/depression | n 1 | No problems | I am not anxious or depressed |
| | 3 Timitety/depression | 2 | Slight problems | I am slightly anxious or depressed |
| | | 3 | Moderate | I am moderately anxious or depressed |
| | | | problems | |
| | | 4 | Severe problems | I am severely anxious or depressed |
| | | 5 | Extreme | I am extremely anxious or depressed |
| | | | problems | |
| EQ-5D visual | FO-5D VAS is | a co1 | ntinuous score | e ranging from 0 (worst health you |
| | - | | | ` ` ` |
| analogue scale (VAS) | can imagine) to | 100 ( | best health yo | ou can imagine). |
| EQ-5D VAS change | EQ-5D VAS pos | t-ba | seline value – | EQ-5D VAS baseline value |
| from baseline | | | | |
| EQ-5D VAS clinically | The change from | ı bas | seline in EQ-5 | 5D VAS will be categorized in two |
| relevant change from | ways: | | | |
| | • | <i>(</i> \ | 7 | |
| baseline | 1. $\leq$ -7, -6 to | | | |
| | 2. $\leq$ -10, -9 t | | | |
| EQ-5D Valuation | EQ-5D Valuation | on i | ndex summa | arizes the information of the 5 |
| index | dimensions of th | e de | scrintive syste | em |
| mach | | | | |
| | _ | | | 3, 4 and 5 to each level of the 5 |
| | dimension | s (se | e table) | |
| | | ` | · · | n patient-time point combination. A |
| | | | | - |
| | | | | of 5 level codes; one level code for |
| | each dimension. The dimensions are ordered as described in the | | | |
| | table above. | | | |
| | | | 125/12 india | ates 'no problems in walking about, |
| | _ | | | - |
| | slight prob | lem | s washing or | dressing myself, unable to do my |
| | • | | | <u> </u> |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| | usual activities, severe pain or discomfort, moderately anxious or depressed'. c. Assign an index value to each health state as defined in Attachment 5 where EQ-5D health state is converted to a single summary index by applying a formula that essentially attaches weights to each of the levels in each dimension. The algorithm is based on the valuation of EQ-5D health states using the UK TTO (=time trade-off method) based value set. |
|---|---|
| EQ-5D Valuation index change from baseline | EQ-5D valuation index post-baseline value – EQ-5D valuation index baseline value |

# 5.3.1.3. Clinical outcomes

| Measurement | Formula |
|---|---|
| Measurement Incidence of treatment-emergent adjudicated influenza complications | The incidence of treatment-emergent adjudicated influenza complications from first intake of study drug until the end of the study will be categorized in a hierarchical fashion. The overall category will consist of any complication. The following subcategories are defined: Pulmonary complications: respiratory failure, primary viral pneumonia, secondary bacterial pneumonia, exacerbations of chronic underlying pulmonary diseases, bronchitis other complications Extrapulmonary complications: Cardiovascular and cerebrovascular disease (eg, myocardial infarction, congestive heart failure, arrhythmia, stroke), Muscular disorders (eg, myositis, rhabdomyolysis), Central nervous system (CNS) involvement, Acute exacerbation of chronic kidney disease, Severe dehydration, |
| | <ul> <li>Acute exacerbation of chronic kidney disease,</li> <li>Severe dehydration,</li> <li>Decompensation of previously controlled diabetes mellitus,</li> <li>Other infections (eg, sinusitis, otitis)</li> <li>Other complications</li> <li>Pulmonary complications including sinusitis and otitis</li> <li>Major / minor complications</li> <li>Infectious / non-infectious complications</li> <li>The complications sinusitis and otitis are determined based on their</li> </ul> |
| Incidence of hospital admission 28 days after treatment initiation. | MedDRA preferred terms as listed in Attachment 1, Table 6, for the protocol terms 'Sinus infection' and 'Ear infection' respectively. Only those terms that are judged to be complications by the adjudication committee will considered for the endpoint 'pulmonary complications including sinusitis and otitis'. Was the subject admitted to the hospital? The following medical encounters are considered as indicating hospitalization: 'Emergency Room', 'Intensive Care Unit', 'Hospice/Palliative Care Unit', and 'Hospital Inpatient Department'. Subjects hospitalized for a preplanned surgery or procedure will not be counted as a hospitalized |

| | subject for this endpoint. If a subject is discharged from hospital and subsequently readmitted, the subject will only be counted once as being admitted. |
|---|---|
| | Categories will be Yes (1) or No (0). |
| Incidence of treatment-emergent adjudicated influenza complications including hospitalization | The incidence of treatment-emergent adjudicated influenza complications from first intake of study drug until the end of the study or hospitalization 28 days after treatment initiation as defined above. Categories will be Yes (1) or No (0). |
| Time to resolution of | It is assumed that all subjects will have fever at baseline. |
| fever (hours) [Time-to event] | The time to resolution of fever is defined as the time in hours from initiation of study treatment to the first of a successive series of 3 recordings for which the fever is resolved (see Table 8). The 3 successive recording may have been done over 4 scheduled successive analysis timepoints, in case of 1 missing in between timepoint. |
| | In case the resolution of fever is not achieved, data will be censored. |
| | Censoring will be done as follows: |
| | Last non-missing record(s) indicate resolution of fever (but insufficient recordings to meet the time to resolution) |
| | Censoring will be done at the first record of resolution of fever from the last series of recordings of resolution of fever |
| | 2) Last non-missing record does not indicate resolution of fever |
| | Censoring will be done after the last observation, which is 08:00 on the same day if the last observation was a diary entry from 00:01 until 02:00, 20:00 on the same day if the last observation was a diary entry from 02:01 until 14:00, and 08:00 the next day if the last entry was a diary entry from 14:01 until 00:00. |
| | Additionally, in the following cases the subject will be censored using a time-to equal to the maximum time across all subjects: |
| | o death, |
| | o if a subject had not resolved the fever at time of hospitalization and/or during hospitalization and no further data on fever resolution is available |

Table 8: Resolution criterion for fever

| Assessment | Resolution Criterion |
|-------------|----------------------------------------------------|
| Temperature | temperature as recorded on the ePRO device <37.0°C |
| | without the use of antipyretics on that day |

The following ATC level 4 codes and generic medication names indicate an antipyretic medication:

- N02BA
- N02BE
- Ibuprofen
- Paracetamol
- Acetylsalicylic acid

If an antipyretic medication misses components of its start and/or stop dates (day and/or month and/or year) the following actions will be taken:

- 1. In case of partial start date
  - If the day is missing, then then the day will be the first day of the month (or the day of first dose whichever is later)
  - If the month is missing the month will be January (or the months of first dose whichever is later)
  - If the year is missing, then the year will be the year of first dose
- 2. In case of partial end date
  - If the day is missing, then the day will be the last day of the month (or the day of last contact with the subject whichever is earlier)
  - If the month is missing, then the month will be December (or the month of last contact with the subject whichever is earlier)
  - If the year is missing, then the year will be the year from the date of last contact with the subject.
- 3. In case of a completely missing start date, the antipyretic will be considered as having started before the trial
- 4. In case of a completely missing end date, the antipyretic medication will be considered as ongoing at the end of the trial.

Antipyretic medication use associated with both the morning and evening temperature recordings for a particular day is also obtained

| | from the subject's diary. If a subject indicates that they used an antipyretic 'today' then the date of this assessment indicates antipyretic use on that whole day. If a subject indicates that they used an antipyretic 'yesterday' then this indicates antipyretic medication use on the whole day before the assessment day. |
|---|---|
| Incidence of all-cause mortality | Did the subject die after first dose of study drug? Categories will be Yes (1) or No (0). |

#### 5.3.1.4. Viral kinetics

The viral culture (TCID<sub>50</sub>) measurements are analyzed using two methods (depending on influenza subtype); ie, NP ELISA and Hemagglutination Inhibition Assay. For analysis purposes the results from the NP ELISA method will be used when available, otherwise the results from the Hemagglutination Inhibition Assay will be used. This will be determined per analysis visit. As a consequence, the series of results of a subject can be a combination of both methods (for example at baseline the NP ELISA result is used and at Day 3 the Hemagglutination Inhibition Assay result is used).

The endpoints listed below will be based on results from nasal mid-turbinate (MT) swabs taken from central testing, excluding data from leftover samples from local virology tests.

| Measurement | Formula |
|---|---|
| Log <sub>10</sub> viral load actual values (Log <sub>10</sub> vp/mL) | Log <sub>10</sub> of the actual values as measured with qRT PCR |
| Viral load negativity | Viral load will be categorized as Negative or Positive: |
| (Log <sub>10</sub> vp/mL) | • Negative (lower than LOD) |
| | <ul> <li>Positive (between LOD and LOQ or quantifiable (above LOQ)).</li> </ul> |
| Viral load<br>categorization (Log10<br>vp/mL) | Viral load will be categorized as Target not detected, Target detected, and Quantifiable: |
| | • Target not detected (lower than LOD) |
| | • Target detected (between LOD and LOQ) |
| | Quantifiable (above LOQ) |
| Log <sub>10</sub> viral load change<br>from baseline (Log <sub>10</sub><br>vp/mL) | Log <sub>10</sub> viral load post-baseline value – log <sub>10</sub> viral load baseline value |

| Log <sub>10</sub> viral titer actual values (Log <sub>10</sub> TCID <sub>50</sub> /mL) | Log <sub>10</sub> of the actual values as measured with viral culture |
|---|---|
| Viral titer negativity | Viral titer will be categorized as Negative or Positive: |
| $(\text{Log}_{10} \text{ TCID}_{50}/\text{mL})$ | Negative (lower than LOQ) |
| | Positive (quantifiable results) |
| Log <sub>10</sub> viral titer change<br>from baseline (Log <sub>10</sub><br>TCID <sub>50</sub> /mL) | Log <sub>10</sub> viral titer post-baseline value – log <sub>10</sub> viral titer baseline value |
| Viral load AUC <sub>0-10d</sub> | Viral load AUC calculated from baseline to Day 10: |
| trapezoidal method | AUC is calculated by the trapezoidal summation rule, based on planned days of sampling, including the timepoints with (imputed) values available: |
| | Sum over i of $(t_{i+1}-t_i)*(Viral\ load_{ti+1}+Viral\ load_{ti})/2$ |
| | The following rules will be applied in the order described below to deal with missing values before calculating the Viral load AUC: |
| | • If the baseline value is missing, then the mean baseline value over all subjects in the ITT-i set will be used. |
| | • If a single or sequential intermediate values (not the baseline value) are missing, then the missing value will be replaced by linear interpolation of the two adjacent values. Note: this is done automatically when applying the trapezoidal summation rule. If the Day 10 value is missing, but there is an assessment after Day 10, then this value will be used to interpolate the value for Day 10. |
| | • If the Day 10 value is missing, and there are no values available after Day 10, then it will be imputed with the last observed post-baseline value (LOCF). |
| | Note: In case no post baseline value is available the AUC will be missing. |
| Viral titer AUC <sub>0-10d</sub> | Viral titer AUC calculated from baseline to Day 10: |
| trapezoidal method | AUC is calculated by the trapezoidal summation rule, based on planned days of sampling, including the timepoints with (imputed) values available: |
| | Sum over i of $(t_{i+1}-t_i)*(Viral\ titer_{ti+1}+Viral\ titer_{ti})/2$ |

| | The following rules will be applied in the order described below to deal with missing values before calculating the Viral titer AUC: |
|---|---|
| | • If the baseline value is missing, then the mean baseline value over all subjects in the ITT-i set will be used. |
| | • If a single or sequential intermediate values (not the baseline value) are missing, then the missing value will be replaced by linear interpolation of the two adjacent values. Note: this is done automatically when applying the trapezoidal summation rule. If the Day 10 value is missing, but there is an assessment after Day 10, then this value will be used to interpolate the value for Day 10. |
| | • If the Day 10 value is missing, and there are no values available after Day 10, then it will be imputed with the last observed post-baseline value (LOCF). |
| | Note: In case no post baseline value is available the AUC will be missing. |
| Time to viral negativity<br>by qRT-PCR (days)<br>[Time-to event] | The time to viral negativity is defined as the time (in days) from first study drug intake until a subject is considered influenza A viral negative. This is the first timepoint of two consecutive timepoints with confirmed negative nasal MT swab ie, the first and next assessment are equal to 'negative' (ignoring missing values). In case the first 'negative' is the last available assessment the subject is considered to have reached viral negativity at this last assessment. If this doesn't occur, a subject will be censored at the time of the last observed non-negative swab + 1 day. Note that for deriving the time to viral negativity by qRT-PCR every subject is considered positive at baseline. |
| Time to viral negativity<br>by viral culture (days)<br>[Time-to event] | The algorithm for Time to viral negativity by viral titer is similar as 'Time to viral negativity by viral load' but viral titer assessments are used instead. |

# 5.3.2. Analysis Methods

#### **Descriptive statistics**

The descriptive statistics that will be shown may include the number of subjects, mean, standard deviation, standard error, 95% CI, median, range, interquartile range, and geometric mean with corresponding 95% CI.

#### Kaplan-Meier analysis, Gehan-Wilcoxon test and Log-rank test

All Time-to event variables will be analyzed using a stratified Gehan-Wilcoxon test, a stratified log-rank test and Kaplan-Meier estimates. A summary table including number of subjects included in the analysis, number of subjects censored, 25th and 75th percentiles and median time-to event, with 95% confidence intervals based on log-log transformation method, and the p-values calculated based on the stratified Gehan-Wilcoxon test and stratified log-rank test will be presented.

The data will be presented graphically using the Kaplan-Meier estimate of the survival function by treatment.

For subgroup analyses, Kaplan-Meier plots will be produced per subgroup and Gehan-Wilcoxon test will be produced for each category of a subgroup.

#### Accelerated failure time (AFT) model

When indicated, time-to event variables will be compared between pimodivir and placebo using an accelerated failure time (AFT) model. The distribution to be used will be determined based on the goodness of fit of the model using Akaike's information criterion and will be selected from the following parametric families: lognormal, log-logistic, or Weibull. The AFT model will include the fixed categorical effects for treatment (with placebo as the reference) and stratification factors. The scale parameter will be the same across groups.

A summary of the final AFT model will include parameter estimates and associated standard errors, estimated accelerated failure time ratios versus placebo and associated 95% confidence intervals, and p-values. The survival curves per treatment group of the accelerated failure time model will also be shown with the Kaplan-Meier plots included in the same output.

For subgroup analyses the survival curves will be shown for each subgroup category separately.

Bootstrapping with replacement, and also considering the actual proportion of subjects in each stratum, will be used to obtain a 100% sample size 10001 times. The median (95% CI) time-to event will be derived from the 10001 bootstrapped samples.

#### Cox Proportional Hazard model

A stratified Cox proportional hazards model will be used adjusted for the stratification factors. The hazard ratio for the comparison of pimodivir versus placebo will be reported together with the 95% confidence interval. A Log-log plot of survival will be added to check the proportional hazard assumption of the Cox proportional hazards model.

For subgroup analyses the Log-log plot of survival will be shown for each subgroup category separately.

#### Logistic regression model

A logistic regression model (applying Firth's penalized likelihood approach) with treatment group and stratification factors as fixed effects, will be used to analyze the binary outcome and to obtain the odds ratios (95% CI) for the comparison of pimodivir versus placebo.

# 5.3.2.1. Symptoms of Influenza (Flu-iiQ<sup>™</sup> Module 1)

#### Composite symptoms scores (systemic symptoms, respiratory symptoms)

The actual composite symptom scores and changes from baseline will be shown descriptively and by mean (SE) plots per analysis visit and timepoint.

# Time to resolution of: cough; sore throat; headache; nasal congestion; feeling feverish; body aches and pains; fatigue; neck pain; interrupted sleep; loss of appetite; the 7 primary influenza-related symptoms considering improvement from baseline

The time to resolution of cough, sore throat, headache, nasal congestion, feeling feverish, body aches and pains, fatigue, neck pain, interrupted sleep, loss of appetite, and the 7 primary influenzarelated symptoms, improvement from baseline will be analyzed by Kaplan-Meier analysis, Gehan-Wilcoxon test, log-rank test, AFT model, and Cox proportional hazards model.

The AFT and Cox models will include the fixed categorical effects for treatment (with placebo as the reference) and stratification factors and the baseline symptom score as a continuous variable.

If the baseline symptom score is missing, then the baseline score will be imputed as the median score from all subjects in the ITT-i set.

#### 5.3.2.2. Other Patient Reported Outcome

#### Time to return to daily activities

Time to return to daily activities will be analyzed by Kaplan-Meier analysis, Gehan-Wilcoxon test, log-rank test, AFT model, and Cox proportional hazards model.

The AFT and Cox models will include the fixed categorical effects for treatment (with placebo as the reference) and stratification factors.

#### Patient global Impression parameters and daily activities resumption

The subject's perception of severity and change of influenza symptoms (PGIS and PGIC) and the daily activities resumption will be tabulated per parameter and per category by analysis timepoint using frequency tabulations.

# EQ-5D dimensions

Tabulations of the number (and percentage) of subjects per parameter, response and timepoint will be shown per treatment group.

# **EQ-5D VAS, EQ-5D Valuation index**

The actual values and changes from baseline will be shown descriptively and by mean (SE) plots per analysis visit.

The proportion of subjects with a clinically relevant change from baseline of 7 or more (decrease or increase) and of 10 or more (decrease or increase) will be provided for each post-baseline assessment.

#### Missing data

- 1. If for a questionnaire one (or more) dimensions of the descriptive system are missing then
  - The EQ-5D VAS will be included in the analysis
  - The valuation index will not be included in the analysis
  - The non-missing dimensions of EQ-5D descriptive system will be included in the analysis
    of the separate dimensions
- 2. If for a questionnaire the EQ-5D VAS is missing then
  - the EQ-5D descriptive system and valuation index will be included in the analysis if complete (otherwise see 1)

#### 5.3.2.3. Clinical Outcomes

Incidence of treatment-emergent adjudicated influenza complications, hospital admission rate, incidence of treatment-emergent adjudicated influenza complications including hospital admission, and incidence of all-cause mortality

The number and percentage of subjects in each parameter category and subcategory will be tabulated and listed. All subjects in the applicable analysis set will be counted for the denominator of the proportion.

The occurrence (yes/no) for hospital admission rate, incidence of treatment-emergent adjudicated influenza complications including hospital admission, and incidence of all-cause mortality will be analyzed using logistic regression as described above (Section 5.3.2).

The occurrence (yes/no) of influenza complications will be analyzed using logistic regression as described above, for each of the following categories:

- the overall influenza complications
- the pulmonary complications,
- the extrapulmonary complications
- the pulmonary complications including sinusitis and otitis
- the infectious complications
- the non-infectious complications
- the major complications
- the minor complications

#### Time to resolution of fever

Time to resolution of fever will be analyzed similarly as time to return to daily activities.

A subgroup analysis will be done based on the subset of subjects with fever at baseline (temperature  $\geq$ 37.0°C) as recorded as part of the on-site vital signs assessment.

Temperature recordings made by the subject on the ePRO device lower than 34°C or higher than 43°C will not be included in the analysis.

#### 5.3.2.4. Viral kinetics

#### Viral load and viral titer over time

The actual values and change from baseline of the viral load and viral titer over time will be shown descriptively and by mean (SE) plots per analysis timepoint.

Individual AUCs from baseline to Day 10 for both viral load and viral titer will be calculated using the trapezoid method and summarized using descriptive statistics.

Viral load negativity, viral load categorization, and viral titer negativity will be summarized using frequency tabulations (n and %) at each analysis visit.

■ *Difference in mean viral load AUC calculated from baseline to Day 10:* 

Post-baseline mean viral load values up to and including Day 10 will be analyzed using a restricted maximum likelihood based repeated measures approach. Analyses will include the fixed, categorical effects of treatment, strata, visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline viral load and baseline viral load -by-visit interaction. The following list of covariance structures will be applied in the model fit, in the specified order, and the first correlation structure to yield convergence will be applied in the analysis:

- Unstructured [UN]
- Ante-dependence [ANTE(1)]
- Heterogenous Toeplitz [TOEPH]
- Heterogeneous CS [CSH]
- $\blacksquare$  Heterogeneous AR(1) [ARH(1)]
- Toeplitz [TOEP]

The Kenward-Roger approximation will be used to estimate denominator degrees of freedom.

The model above will be used to estimate the difference in the viral AUCs for pimodivir versus placebo.

Post-baseline mean viral titer values up to and including Day 10 will be analyzed as described above for the post-baseline mean viral load values.

A least squares means  $\pm 95\%$  CI plot will also be provided for the estimated viral load and estimated viral titer over time.

#### Time to viral negativity by viral load and by viral titer

The time to viral negativity will be analyzed by Kaplan-Meier analysis, Gehan-Wilcoxon test, logrank test, AFT model, and Cox proportional hazards model.

The AFT and Cox models will include the fixed categorical effects for treatment (with placebo as the reference) and stratification factors and the baseline viral load, or viral titer, as a continuous variable.

# 5.4. Exploratory Endpoints

#### 5.4.1. Definition

Formulae to be used for derived variables, including data conversions, are provided in the tables below. Note that for time to event variables the actual date times will be used.

# 5.4.1.1. Impact of Influenza (Flu-iiQ™ Modules 2, 3, 4)

| Composite impact score | Per datetime and per module (modules 2, 3 and 4) of the FLU-iiQ <sup>TM</sup> questionnaire a composite impact score will be calculated as the mean of the non-missing items in each module respectively on a 0-3 scale. |
|---|---|
| | If more than 50% of the items to construct a Composite impact score are missing, then the value for that composite impact score for that individual and time point is coded as missing (ie, 4 or more items missing for module 2, 3 or more items missing for module 3, 3 or more items missing for module 4). |
| Composite impact | For each module (modules 2, 3 and 4) of the Flu-iiQ <sup>TM</sup> questionnaire: |
| score change from baseline | Composite impact score post-baseline value – composite impact score baseline value |
| Time to<br>normalization of<br>impact on daily<br>activities (hours) | Time to normalization of impact on daily activities is based on module 2 of the FLU-iiQ <sup>TM</sup> questionnaire, and is defined as the time in hours from the first dose of investigational product until the first one of a successive series of 3 recordings where all scores in the FLU-iiQ <sup>TM</sup> module are reported as "no difficulty". |
| | The 3 successive recordings may have been done over 4 scheduled successive analysis timepoints, in case of 1 missing in between timepoint. |
| | Censoring will be done similar to the time to resolution of influenza symptoms. |
| Time to<br>normalization of<br>impact on emotions<br>(hours) | The algorithm for time to normalization of impact on emotions is similar to 'Time to normalization of impact on daily activities'. Module 3: emotional impact is used and recordings should report "not at all" to define resolution. |
| Time to<br>normalization of<br>impact on others<br>(hours) | The algorithm for time to normalization of impact on others is similar to 'Time to resumption of normalization of impact on daily activities'. Module 4: impact on others is used and recordings should report "not at all concerned" to define resolution. |

# 5.4.2. Analysis Methods

# 5.4.2.1. Impact of Influenza (Flu-iiQ™ Modules 2, 3, 4)

#### **Composite impact scores**

The actual composite impact scores and changes from baseline will be shown descriptively and by mean (SE) plots per analysis visit and timepoint.

# <u>Time to resumption of normal activities for usual activities, for emotional impact, for impact on others</u>

The times to resumption of normal activities will be analyzed similarly as the time to resolution of the individual symptoms of influenza.

#### 6. TASTE AND SWALLOWABILITY

#### 6.1. Definition

Taste and swallowability will only be assessed for adolescents in this study.

The acceptability of the taste will be derived from the responses to the overall question on taste, dichotomizing the responses 'None' and 'Weak' as acceptable and responses 'Moderate' or 'Strong' as unacceptable.

For the swallowability, a dichotomization of the responses will be made of 'slightly difficult' or worse vs. 'neither difficult nor easy' or better.

# 6.2. Analysis Methods

Taste and swallowability questionnaire results will be summarized for the safety set per tablet intake (first and last intake of the study drug) by means of frequency tabulations of the actual responses. Additionally, the number of subjects (%) will be presented by response category (including dichotomization) for swallowability and taste separately.

#### 7. SAFETY

All safety analyses will be done on the Safety Set.

#### 7.1. Adverse Events

#### 7.1.1. Definitions

#### **Coding of AE**

The verbatim terms used in the eCRF by investigators to identify AEs will be coded using the Medical Dictionary for Regulatory Activities. Events are looked at on the level of their preferred term.

#### **Treatment-emergent AE**

Pre-treatment AEs are defined as AEs that were reported or worsened after signing the ICF up to the start of study drug dosing. Treatment-emergent AEs (TEAE) are defined as AEs that were reported or worsened on or after the start of study drug dosing and up to and including the end of the follow-up phase.

An AE, at the preferred term level, is considered treatment-emergent if:

- An AE starts after or at first dose of study drug and
  - o The AE was not present prior to first dose of study drug
  - O An AE was present prior to first dose of study drug:
    - The same AE (based on preferred term) started 2 or more days after the end date of the AE present prior to first dose
    - The same AE (based on preferred term) starts at the end date or the day after the end date of the AE present prior to the first dose and new AE has worsened, ie an increase in toxicity grade or changed to an SAE
- The start date of the AE is missing
- The start time of the AE is missing, and the AE was not present the day before first dose of study drug, and the start date of the AE is the same as the start date of first dose of study drug
- The day is missing of the AE start date but month and year are the same as month and year of first dose of study drug
- The month is missing of the AE start date but year is the same as year of first dose of study drug

#### **Phase allocation of AE**

Adverse events present in the SDTM database are allocated to phases based on their start date and time. If the start date and time of an event falls between (or on) the start and stop date and time of a phase, the AE is attributed to that phase (treatment-emergent principle).

Rule: phase start datetime  $\leq$  AE start datetime  $\leq$  phase stop datetime.

Incomplete AE dates and or times (ie, time and/or day and/or month and/or year missing):

- In case of partial AE start dates and or times, the events are allocated to the phases using the available partial information on start and end datetime; no imputation will be done. If, for instance, for the AE start date only month and year are available, these data are compared to the month and year information of the phases. This rule may lead to multiplication of the event as a consequence of its assignment to multiple phases.
- In case of a completely missing AE start date, the event is allocated to the first active treatment phase, except if the end date of the AE falls before the start of this active treatment phase.
- In case of a completely missing AE end date, the following rules apply:
  - in case the date is identified as unknown the date will remain missing;
  - in case the date is not flagged as unknown the date is assumed to be the cut-off date of the analysis for subjects still ongoing in the study, and the end date of the last phase for subjects who discontinue or completed the study.

#### Examples:

Screening phase: start date: 02JAN2017 - stop date: 28JAN2017 Treatment phase: start date: 29JAN2017 - stop date: 12AUG2017

- 1) Adverse event: start date: JAN2017- stop date: 15JUL2017
  As the AE start date only has information about month and year, only this information will be used from the phases and therefore the AE will be assigned to the screening phase as well as to the treatment phase.
- 2) Adverse event: start date: JAN2017- stop date 27JAN2017 As the AE stops before or at the start of the treatment phase, it is only assigned to the Screening phase.

*Remarks:* In addition to the date information, time information is taken into account to allocate AEs to phases.

#### **Adverse events**

The variables attributed to adverse events are

- AE term (verbatim and MedDRA preferred term and system organ class)
- Onset datetime, End datetime and duration of AE
- Serious AE (Yes/No), if yes classification will be listed
- Toxicity grade (Mild, Moderate, Severe, Potentially life-threatening)
- Action taken with study treatment (Dose not changed, Dose interrupted, Drug withdrawn, Not applicable, Unknown)
- Relation to study treatment (Not related, Doubtful, Possible, Probable, Very likely)
- Outcome of AE
- AE leading to death (Yes/No)
- Concomitant treatment taken for AE (Yes/No)

- Influenza-related complication (Yes/No)
- Required hospitalization/prolonged hospitalization (Yes/No)

#### **Anticipated Events**

An anticipated event is an AE (serious or non-serious) that commonly occurs as a consequence of the underlying disease or condition under investigation (disease related) or background regimen.

For the purposes of this study the following events will be considered anticipated events. (see Attachment 1 for the classification of AEs into Anticipated Events and Anticipated Event Groups):

- Pneumonia
- Bronchitis
- Sinus infections
- Ear infections
- Worsening of asthma, asthma attack
- COPD exacerbation
- Complications of sickle cell disease, sickle cell crisis
- Complications of diabetes mellitus, diabetic ketoacidosis
- Acute respiratory distress syndrome (ARDS)

#### **Influenza-related complications**

The categories of influenza-related complications are defined in the efficacy Section 5.3.1.3.

Note: the investigator's categorization and assessment of complications may be overruled by the Adjudication Committee.

#### **Confirmed diarrhea events**

Additional details required to confirm a diarrhea event, including number of loose stools episodes per day and stool consistency, will be collected for subjects who report a diarrhea type event.

A confirmed diarrhea event is defined as three or more loose stools episodes per day with a consistency of 'loose' or 'watery'.

# 7.1.2. Analysis Methods

#### **Treatment-emergent adverse events**

There will be no formal statistical testing unless indicated otherwise.

A summary will be provided for the following TEAEs per phase (Treatment phase, Follow-up phase) and for the combination of Treatment and Follow-up phases:

- any adverse events,
- serious adverse events,
- deaths due to AE,
- adverse events by worst toxicity grade,
- AEs of worst grade 3 or 4
- AEs of worst grade 3

- AEs of worst grade 4
- AEs at least possibly related to study drug,
- AEs for which study drug was temporarily stopped,
- AEs for which study drug was permanently stopped,
- AEs leading to study discontinuation
- serious adverse events that were at least possibly related to study drug.
- adjudicated influenza related complications
- COVID-19 AEs
- COVID-19 serious adverse events
- COVID-19 non-serious adverse events

The adverse events will be shown by MedDRA system organ class and preferred term, in order of descending frequency in the pimodivir group. For each AE, the percentage of subjects who experience at least 1 occurrence of the given event will be summarized by treatment group and per phase (Treatment phase, Follow-up phase) and for the combination of Treatment and Follow-up phases. Incidence tabulations will be provided for the following categories:

- any adverse events
- serious adverse events
- AEs at least possibly related to study drug
- AEs for which study drug was temporarily stopped
- AEs for which study drug was permanently stopped
- AEs leading to study discontinuation
- serious adverse events that were at least possibly related to study drug
- AEs related to COVID-19 infection
- Serious adverse events related to COVID-19 infection
- AEs related to COVID-19 infection leading to death

and in addition for treatment emergent adverse events with incidence of at least 5% in any treatment group.

In order to fulfil requirements for the plain language summary document and presentations for EudraCT the following adverse event categories will be shown by MedDRA system organ class and preferred term per phase (Treatment phase, Follow-up phase) and for the combination of Treatment and Follow-up phases. No tabulations by subgroups will be provided for these categories:

- deaths due to AEs that were at least possibly related to study drug
- AEs for which study drug was permanently stopped that were at least possibly related to study drug

- non-serious AEs that were at least possibly related to study drug
- any non-serious AEs

AEs leading to death, SAEs, AEs leading to dose interruption or permanent stop of study drug, AEs related to COVID-19 infection will be listed separately. All AEs will be listed in an individual subject data listing, including pre-treatment AEs. All listings will be provided for the safety set.

The duration (in days) of an AE is calculated based on the AE start date and AE end date as:

```
AE duration = AE end date – AE start date + 1
```

Note that the AE duration will only be calculated when the start date and end date is fully known, in case of partial or missing start and end dates the AE duration will be missing.

#### **Anticipated Events**

Frequency tabulations of anticipated events and anticipated event grouped terms will be shown for treatment phase, follow-up phase and for the combination of treatment and follow-up phases. The tabulation will show per treatment the number (%) of subjects with serious, non-serious and total anticipated events and anticipated event grouped terms and a one-sided p-value of Fisher exact test for anticipated events and anticipated event grouped terms. Note that the Fisher exact test will only be provided for the occurrence of events for the combination of treatment and follow-up phases.

A listing of the anticipated events will be added.

More details on the anticipated events analysis can be found in the Anticipated Events Safety Monitoring plan.

#### **Influenza-related complications**

Adverse Events adjudicated as influenza-related complications will be tabulated by category and adverse event, for treatment phase and follow-up phase and for the combination of treatment and follow-up phases.

Adverse events investigator-assessed as influenza-related complications will also be tabulated by category and adverse event, for treatment phase and follow-up phase and for the combination of treatment and follow-up phases. A listing showing the AEs reported as influenza-related complications and complication information will be made linking the information to the AE listing.

#### **Confirmed diarrhea events**

The number and percentage of subjects who experience at least 1 occurrence of confirmed diarrhea events will be summarized by treatment group and per phase (Treatment phase, Follow-up phase) and for the combination of Treatment and Follow-up phases.

For all subjects that complete the additional diarrhea form, a cross-tabulation of number of loose stools episodes per day (categorized as 1, 2, 3 or more) versus stool consistency will be produced by treatment group and per phase (Treatment phase, Follow-up phase) and for the combination of

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

62

Treatment and Follow-up phases. If a subject has more than 1 diarrhea event per phase, then the worst response from all events in that phase will be tabulated.

Descriptive statistics will be produced by treatment group for the number of days from first dose of study drug to onset of first diarrhea event and for total duration of diarrhea events. A frequency tabulation will be produced by treatment group for the number of days from last dose of study drug to resolution of last diarrhea event.

Frequency tabulations will be produced by treatment group and per phase (Treatment phase, Follow-up phase) and for the combination of Treatment and Follow-up phases for the severity grade of the diarrhea event and for whether any concomitant medication was used to treat the diarrhea event.

No tabulations by subgroups will be provided.

All information recorded on the specific diarrhea form will be listed.

#### 7.2. Clinical Laboratory Tests

#### 7.2.1. Definitions

Laboratory parameters of hematology, serum chemistry and urinalysis will be investigated: all analyses will be done on SI-converted values as available in the database.

# Imputations of numerical values expressed as characters

In case a laboratory test result is censored (no numeric value is available, but only a verbatim term), the following rules are applied:

- '<x' or '>x': a numeric value will be imputed by the cut-off value decreased or increased with one unit respectively
- ' $\leq$ x' or ' $\geq$ x': imputation by x.

#### **Toxicity grades and abnormalities for laboratory parameters:**

The laboratory abnormalities will be determined according to the criteria specified in the WHO grading table<sup>[6]</sup> (see Attachment 2), available toxicity grades in the laboratory raw data will not be used. In case no toxicity grades are defined for a test, the abnormalities (above/below normal range) will be used.

In determining toxicity grades/abnormalities for each subject the following rules are applied:

- Worst grades/abnormalities are determined over the whole observational period, for treatment phase, follow-up phase and combination of treatment and follow-up phase separately, and including all post-baseline scheduled and unscheduled measurements of that phase.
- The abnormalities "abnormally low" and "abnormally high" are considered equally important, ie, if a subject has as well an abnormally low as an abnormally high value post-

baseline, both abnormalities are shown in the tables. (This implies that the sum of the percentages can be more than 100%)

• If, for a specific test, the grading list provides distinct limits for abnormally low (=hypo) values as well as for abnormally high (=hyper) values, this test should be repeated for hyper and hypo limits separately in cross-tabulations.

#### Treatment-emergent definition for toxicity grades and abnormalities

An abnormality (toxicity grade or abnormality based on normal ranges) will be considered treatment-emergent if it is worse than the baseline abnormality. If the baseline abnormality is missing, the abnormality is always considered as treatment-emergent. A shift from "abnormally low" at baseline to "abnormally high" post-baseline (or vice versa) is also treatment-emergent.

#### 7.2.2. Analysis Methods

Actual values and changes from baseline will be summarized by treatment group at each scheduled time point, including the safety follow-up visit, the Day 28 final study visit and the last study visit.

A tabulation of the toxicities/abnormalities per timepoint will be presented. This table will also show the number and percentage of subjects per toxicity/abnormality, the number and percentage of subjects per treatment-emergent abnormality, and the cumulative number of subjects per treatment-emergent abnormality per post-baseline timepoint, including the safety follow-up visit, the Day 28 final study visit and the last study visit.

Additionally, a tabulation of the worst toxicity/abnormality will be presented. This table will show the number and percentage of subjects per worst toxicity/abnormality per phase (Treatment phase, Follow-up phase) and for the combination of Treatment and Follow-up phases.

A cross-tabulation of the worst toxicity/abnormality versus baseline will be presented per phase (treatment, follow-up and combination treatment + follow-up). This table will also show the number and percentage of subjects per worst toxicity/abnormality, the number and percentage of subjects per treatment-emergent worst toxicity/abnormality, and the cumulative number of subjects per treatment-emergent toxicity/abnormality.

For tabulations of hyperglycaemia, the results will also be presented for the subgroup of subjects that had been fasting for at least 10 hours.

Mean  $\pm$  SE graphs over time for the actual values and changes from baseline will be generated for all tests performed.

A listing of abnormal individual subject hematology and clinical chemistry values from scheduled and unscheduled time points will be provided. This listing will include all other time points for the corresponding subject/parameter.

Grade 3 or higher toxicity laboratory values will be listed separately.

Frequency tables (n %) will be produced for the categorical urinalysis parameters by treatment group at each scheduled timepoint, including the safety follow-up visit, the Day 28 final study visit and the last study visit.

All urinalysis results will be listed.

#### 7.3. Vital Signs

Systolic and Diastolic blood pressure, temperature, pulse rate, respiratory rate will be included in the analysis.

#### 7.3.1. Definitions

Vital Signs abnormalities will be determined according to the WHO grading scale<sup>[6]</sup> and the boundaries defined in Attachment 3.

Worst abnormalities are determined over the whole observational period and for each trial phase separately (treatment phase, follow-up phase and combination of treatment and follow-up phases), including all post-baseline scheduled and unscheduled measurements of that phase.

An abnormality (based on normal ranges) will be considered treatment-emergent if it is worse than the baseline abnormality. If the baseline abnormality is missing, the abnormality is always considered as treatment-emergent. A shift from "abnormally low" at baseline to "abnormally high" post-baseline (or vice versa) is also treatment-emergent.

Assessments taken while the subject was not in a supine position will not be included in descriptive statistics but will be considered in determining worst case values.

# 7.3.2. Analysis Methods

Actual values and changes from baseline will be summarized by treatment group at each scheduled timepoint, including the safety follow-up visit, the Day 28 final study visit and the last study visit.

A tabulation of the abnormalities per timepoint will be presented. This table will also show the number and percentage of subjects per abnormality, the number and percentage of subjects per treatment-emergent abnormality, and the cumulative number of subjects per treatment-emergent abnormality per post-baseline timepoint, including the safety follow-up visit, the Day 28 final study visit and the last study visit.

Additionally, a tabulation of the worst abnormality will be presented. This table will show the number and percentage of subjects per worst abnormality.

A cross-tabulation of the worst abnormality versus baseline will be presented per phase (treatment, follow-up and the combination treatment and follow-up phase). This table will also show the number and percentage of subjects per worst abnormality, the number and percentage of subjects per treatment-emergent worst abnormality, and the cumulative number of subjects per treatment-emergent abnormality.

Mean  $\pm$  SE graphs over time for the actual values and changes from baseline will be generated for all tests performed.

Vital signs data for subjects having at least one treatment-emergent abnormality will be listed.

#### 7.4. Physical examinations

Abnormal physical examination results will be listed.

#### 7.5. Electrocardiogram

PR duration, QT duration, QRS duration, Heart Rate and QTc intervals using Bazett's correction formula and Fridericia's correction formula will be investigated. QTc values will be used as reported, they will not be recalculated. If the ECG is performed in triplicate, then the mean of the non-missing ECG recordings will be used as the value for each specific parameter and timepoint.

#### 7.5.1. Definitions

ECG abnormalities will be determined according to the boundaries defined in Attachment 4.

An abnormality (based on normal ranges) will be considered treatment-emergent if it is worse than the baseline abnormality. If the baseline abnormality is missing, the abnormality is always considered as treatment-emergent. A shift from "abnormally low" at baseline to "abnormally high" post-baseline (or vice versa) is also treatment-emergent.

Assessments taken while the subject was not in a supine position will not be included in descriptive statistics but will be considered in determining worst case values.

# 7.5.2. Analysis Methods

Actual values and changes from baseline will be summarized by treatment group at each scheduled timepoint, including the safety follow-up visit, the Day 28 final study visit and the last study visit.

A tabulation of the abnormalities per timepoint will be presented. This table will also show the number and percentage of subjects per abnormality, the number and percentage of subjects per treatment-emergent abnormality, and the cumulative number of subjects per treatment-emergent abnormality per post-baseline timepoint, including the safety follow-up visit, the Day 28 final study visit and the last study visit.

A cross-tabulation of the worst abnormalities versus baseline will be presented per phase (treatment, follow-up and the combination treatment and follow-up phase). This table will also show the number and percentage of subjects per worst abnormality the number and percentage of subjects per treatment-emergent worst abnormality, and the cumulative number of subjects per treatment-emergent abnormality.

Mean  $\pm$  SE graphs over time for the actual values and changes from baseline will be generated for all tests performed.

A frequency tabulation of the QT/QTc change categories at Day 28, safety follow-up visit and last study visit versus baseline will be presented.

ECG data for subjects having at least one treatment-emergent abnormality will be listed.

#### 8. RESISTANCE

#### 8.1. Viral Phenotype

The pimodivir  $EC_{50}$  and oseltamivir  $IC_{50}$  with their fold change values will be analyzed at baseline and at all post-baseline visits with available data (FC = fold change in  $EC_{50}$  (IC<sub>50</sub>) value).

FC is calculated as the EC50 (or IC50) of the subject's influenza strain divided by the EC50 (or IC50) of a reference strain. If the patient EC50 (or IC50) is censored, the fold change value gets the same censor, eg, patient EC50 = >20 nM, reference EC50 = 4nM, Fold Change value >5.

The following output will be provided:

- Emerging phenotypic resistance: descriptive statistics for FC in EC<sub>50</sub> and IC<sub>50</sub> value for pimodivir and oseltamivir respectively at baseline and at all post-baseline visits with available data. The number (%) of subjects by treatment arm with censored phenotype data (by lower and upper bound) at baseline and at all post-baseline visits with available data will also be shown.
- Descriptive statistics for fold change ratio of all post-baseline visits with available data versus baseline including geometric mean and 95% CI.
- A listing showing viral load data together with phenotype data (EC<sub>50</sub>, IC<sub>50</sub> and fold change values) per subject and influenza subtype for all available time points including screening/baseline.

#### 8.2. Viral Genotype

Assessment of viral sequences will be done to determine amino-acid substitutions that may be associated with resistance to pimodivir and to other influenza antivirals if present as part of the SOC. To that end, genotypic data for PB2, PB1, PA, NA, HA and optionally other genome segments of the influenza virus will be gathered.

All positions in the gathered regions will be analyzed for all samples, overall and by influenza subtype.

The gathered regions most relevant for pimodivir are PB2, PB1 and PA, those for neuraminidase inhibitors (NAI) (including oseltamivir) are NA and HA

The following 12 amino-acid positions in PB2 are of interest: 306, 323, 324, 325, 337, 357, 363, 376, 378, 404, 406, 431, and 510.

The following mutations in NA, associated with resistance to oseltamivir, are of interest:

- For subtype H1N1: D199N, I223R, H275Y, and N295S
- For subtype H3N2: E119V, H274Y, R292K, and N294S

The list of positions of interest might be updated during the analysis.

A mutation is treatment-emerging at a specific (post-baseline) time-point if the amino-acid of the

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

considered position is absent at screening/baseline and present at that timepoint.

The baseline is the collection of all polymorphisms present at any timepoint up to the first intake of study drug. A table with an overview of the time points underlying the "baseline" will be generated.

Data will be summarized using frequency tabulations (n and %). Displays and individual mutations should be presented for each genome segment separately (ie, PB1, PB2, PA, NA and HA separately). The following output will be provided:

- Baseline polymorphisms: number (%) of subjects with available genotype data, with any baseline polymorphism, and the number of subjects per polymorphism, for all polymorphisms, per treatment arm.
- Baseline polymorphisms: number (%) of subjects with any baseline polymorphism and with specific baseline polymorphisms at the positions of interest.
- Frequency tabulations for the presence of all emerging mutations overall post-baseline.
- Frequency tabulations for the presence of all emerging mutations overall post-baseline at positions of interest.
- Listing for genotype data per subject for all available timepoints including screening/baseline including viral load data (include influenza subtype and influenza subtype category). A patient profile will be created including this data supplemented with the phenotypic data.

#### 9. PHARMACOKINETICS/PHARMACODYNAMICS

Blood samples for PK assessments of pimodivir will be collected from all subjects at the Day 3 and Day 6 visits.

Descriptive statistics of pimodivir plasma concentration over time will be tabulated for the PK analysis set.

#### 9.1. Pharmacokinetics

Based on the individual plasma concentration-time data from all subjects, exposure parameters of pimodivir will be derived using population PK modelling. The following exposure parameters will be derived for the samples collected at Day 3 and Day 6:  $AUC_{12h}$ ,  $C_{trough}$ , and, if feasible,  $C_{max}$ , and  $T_{max}$ .

Descriptive statistics, including arithmetic mean, standard deviation, geometric mean, coefficient of variation, median, minimum, maximum, and interquartile range will be calculated at Day 3 and Day 6 for all available parameters for the PK analysis set.

# 9.2. Pharmacokinetic/Pharmacodynamic Relationships

Pharmacokinetic/Pharmacodynamic relationships will be analyzed for the PD analysis set.

The exposure parameters  $AUC_{12h}$  and  $C_{trough}$  will be categorized into quartiles for the Day 3 visit, only  $C_{trough}$  will be categorized into quartiles for the Day 6 visit. Relationships of these parameters with the primary and selected secondary efficacy endpoints will be explored as follows.

Kaplan-Meier estimates for the time to resolution of the 7 primary influenza-related symptoms will be produced per each quartile for each exposure parameter.

The number and percentage of subjects with treatment-emergent adjudicated influenza complications will be tabulated for each quartile for each exposure parameter.

The number and percentage of subjects admitted to hospital within 28 days after treatment initiation will be tabulated for each quartile for each exposure parameter.

Kaplan-Meier estimates for the time to return to daily activities and for the time to resolution of fever will be produced per each quartile for each exposure parameter.

Relationships of AUC<sub>12h</sub> with safety will be explored as follows. The number and percentage of subjects with the following treatment-emergent adverse events by AUC<sub>12h</sub> quartile will be tabulated:

- Any AE
- AEs of worst grade 3 or 4
- Deaths due to AE
- Serious AEs
- AEs for which study drug was permanently stopped
- AEs at least possibly related to study drug
- Confirmed diarrhea events

A cross-tabulation of the worst treatment-emergent toxicity grades versus AUC<sub>12h</sub> quartile will be presented for the laboratory parameters AST, ALT, and total bilirubin.

Separate tables will be produced for the worst treatment-emergent toxicity grades at Day 3 and overall.

#### 10. HEALTH ECONOMICS

The following medical resource utilization data will be explored

#### 10.1. Definitions

| Measurement | Formula |
|---|---|
| Number of medical care encounters | Medical care encounters, including surgeries and other selected procedures (inpatient and outpatient), as recorded on the eCRF. The number of medical care encounters is derived as the frequency of the medical encounters other than those mandated in the protocol (eCRF). |
| Number of outpatient medical care encounters | Similar to the description for number of medical care encounters, but only for outpatient medical care encounters, as recorded on the eCRF (Hospital Outpatient Department, Laboratory Department, Medical Practitioner Office, Home Care). |
| Frequency of visits of outpatient medical care encounters | Frequency of visits will be provided per outpatient medical encounter type (Hospital Outpatient Department, Laboratory Department, Medical Practitioner Office or Home Care) as reported on the eCRF. |
| Type of practitioner for hospital outpatient department encounters | Type of practitioner will be provided for Hospital Outpatient Department encounters as reported on the eCRF. |

# 10.2. Analysis Methods

Frequency tabulations of medical care encounters and outpatient medical care encounters will be provided per type of medical encounter and for any medical encounter.

Frequency tabulations of the frequency of visits will be provided, per the following medical encounter types:

- Hospital Outpatient Department,
- Laboratory Department,
- Medical Practitioner Office,
- Home Care

Frequency tabulations of the type of practitioner will be provided for the Hospital Outpatient Department.

#### **REFERENCES**

- 1. Guideline, I. H. T. The clinical evaluation of QT/QTc interval prolongation and proarrhythmic potential for non-antiarrhythmic drugs E14. Recommended for adoption at Step; 2006; 4.
- 2. Herdman M, Gudex C, Lloyd A, Janssen MF, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Quality of Life Research. 2011;20:1727-36
- 3. Hurst H, Bolton J. Assessing the clinical significance of change scores recorded on subjective outcome measures. J. Manipulative Physiol Ther. 2004;27:26-35.
- 4. Jaeschke R, Singer J, Guyatt GH. Measurement of health status. Ascertaining the minimal clinically important difference. Control Clin Trials. 1989;10(4):407-415.
- 5. United Nations publication, Standard Country or Area Codes for Statistical Use (M49 standard), https://unstats.un.org/unsd/methodology/m49/
- 6. World Health Organization. "WHO toxicity grading scale for determining the severity of adverse events."; 2003

#### **ATTACHMENTS**

#### ATTACHMENT 1. : ANTICIPATED EVENTS AND ANTICIPATED EVENT GROUPS

Table 9 shows an overview of the anticipated event groups with group number.

Table 10 indicates which adverse event preferred terms (MedDRA PT) are Anticipated Events (AnE) and Closely Related Medical Events (ME) based on MedDRA Version 18.1. These adverse events will be classified as an Anticipated Event according to the protocol term and are grouped into Anticipated Event Groups.

**Table 9: Anticipated Event groups** 

| Group Number | Grouped Term |
|--------------|-----------------------------|
| Group 1 | Infections and infestations |
| Group 2 | Diabetic complications |

Table 10: Anticipated Events (AnE) and Closely Related Medical Events (ME).

| Protocol Term | AnE | ME | MedDRA PT * | MedDRA | Grouped Term | Group |
|---|---|---|---|---|---|---|
| | | | | Code* | | Number |
| Pneumonia | $\boxtimes$ | | Pneumonia | 10035664 | Infections and infestations | 1 |
| Pneumonia | | $\boxtimes$ | Enterobacter pneumonia | 10054218 | Infections and infestations | 1 |
| Pneumonia | | $\boxtimes$ | Pneumonia haemophilus | 10035702 | Infections and infestations | 1 |
| Pneumonia | | $\boxtimes$ | Pneumonia staphylococcal | 10035734 | Infections and infestations | 1 |
| Pneumonia | | $\boxtimes$ | Pneumonia streptococcal | 10035735 | Infections and infestations | 1 |
| Bronchitis | $\boxtimes$ | | Bronchitis | 10006451 | Infections and infestations | 1 |
| Bronchitis | | $\boxtimes$ | Bronchitis bacterial | 10061736 | Infections and infestations | 1 |
| Bronchitis | | $\boxtimes$ | Bronchitis haemophilus | 10006460 | Infections and infestations | 1 |
| Sinus infection | $\boxtimes$ | | Sinusitis <sup>1</sup> | 10040753 | Infections and infestations | 1 |
| Sinus infection | | $\boxtimes$ | Acute sinusitis <sup>1</sup> | 10001076 | Infections and infestations | 1 |
| Sinus infection | | $\boxtimes$ | Chronic sinusitis <sup>1</sup> | 10009137 | Infections and infestations | 1 |
| Sinus infection | | $\boxtimes$ | Viral sinusitis | 10051513 | Infections and infestations | 1 |
| Ear infection | $\boxtimes$ | | Ear infection | 10014011 | Infections and infestations | 1 |
| Ear infection | | $\boxtimes$ | Middle ear effusion | 10062545 | Infections and infestations | 1 |
| Ear infection | | $\boxtimes$ | Otitis externa | 10033072 | Infections and infestations | 1 |
| Ear infection | | $\boxtimes$ | Otitis media | 10033078 | Infections and infestations | 1 |
| Ear infection | | | Otitis media acute | 10033079 | Infections and infestations | 1 |

CONFIDENTIAL – FOIA Exemptions Apply in U.S. Approved, Date: 1 July 2020
| Protocol Term | AnE | ME | MedDRA PT * | MedDRA<br>Code* | Grouped Term | Group<br>Number |
|---|---|---|---|---|---|---|
| Worsening of asthma, asthma attack <sup>2</sup> | | $\boxtimes$ | Asthma | 10003553 | NA | |
| Worsening of asthma, asthma attack <sup>2</sup> | | $\boxtimes$ | Asthmatic crisis | 10064823 | NA | |
| Worsening of asthma, asthma attack <sup>2</sup> | | $\boxtimes$ | Status asthmaticus | 10041961 | NA | |
| COPD exacerbation <sup>3</sup> | $\boxtimes$ | | Chronic obstructive pulmonary disease | 10009033 | NA | |
| COPD exacerbation <sup>3</sup> | | $\boxtimes$ | Emphysema | 10014561 | NA | |
| Complications of sickle cell disease, sickle cell crisis <sup>4</sup> | | $\boxtimes$ | Sickle cell anaemia | 10040641 | NA | |
| Complications of sickle cell disease, sickle cell crisis <sup>4</sup> | | $\boxtimes$ | Sickle cell anaemia with crisis | 10040642 | NA | |
| Complications of sickle cell disease, sickle cell crisis <sup>4</sup> | | $\boxtimes$ | Acute chest syndrome | 10051895 | NA | |
| Complications of sickle cell disease, sickle cell crisis <sup>4</sup> | | $\boxtimes$ | Ischaemic stroke | 10061256 | NA | |
| Complications of sickle cell disease, sickle cell crisis <sup>4</sup> | | | Embolic stroke | 10014498 | NA | |
| Complications of sickle cell disease, sickle cell crisis <sup>4</sup> | | $\boxtimes$ | Deep vein thrombosis | 10051055 | NA | |
| Complications of sickle cell disease, sickle cell crisis <sup>4</sup> | | | Pulmonary embolism | 10037377 | NA | |
| Complications of diabetes mellitus, diabetic ketoacidosis <sup>4</sup> | | | Diabetic complication | 10061104 | Diabetic complications | 2 |
| Complications of diabetes mellitus, diabetic ketoacidosis <sup>4</sup> | | | Diabetic ketoacidosis | 10012671 | Diabetic complications | 2 |
| Complications of diabetes mellitus, diabetic ketoacidosis <sup>4</sup> | | $\boxtimes$ | Diabetes mellitus <sup>5</sup> | 10012601 | Diabetic complications | 2 |
| Complications of diabetes mellitus, diabetic ketoacidosis <sup>4</sup> | | $\boxtimes$ | Diabetic ketoacidotic hyperglycaemic coma | 10012672 | Diabetic complications | 2 |
| Complications of diabetes mellitus, diabetic ketoacidosis <sup>4</sup> | | $\boxtimes$ | Hypoglycaemia | 10020993 | Diabetic complications | 2 |
| Complications of diabetes mellitus, diabetic ketoacidosis <sup>4</sup> | | | Diabetic metabolic decompensation | 10012655 | Diabetic complications | 2 |
| Acute Respiartory Distress Syndrome (ARDS) | | | Acute respiratory distress syndrome | 10001052 | NA | |
| Acute Respiartory Distress Syndrome (ARDS) | | $\boxtimes$ | Acute respiratory failure <sup>6</sup> | 10001053 | NA | |

- <sup>1</sup> Infectious etiology only
- <sup>2</sup> Please note that asthma aggravated codes to a PT of asthma. These PTs will be considered as anticipated events <u>only</u> if the subjects have documented those conditions (such as: asthma, COPD, Sickle cell disease, or diabetes) before enrolling the study.
- <sup>3</sup> Please note that chronic obstructive airways disease exacerbated codes to a PT of chronic obstructive pulmonary disease. These PTs will be considered as anticipated events only if the subjects have documented those conditions (such as: asthma, COPD, Sickle cell disease, or diabetes) before enrolling the study.
- <sup>4</sup> These PTs will be considered as anticipated events only if the subjects have documented those conditions (such as: asthma, COPD, Sickle cell disease, or diabetes) before enrolling the study.
- <sup>5</sup> Please note that diabetes mellitus aggravated and diabetes mellitus exacerbated codes to a PT of diabetes mellitus.
- <sup>6</sup> This event will be considered anticipated only if it occurs in the context of ARDS

# ATTACHMENT 2. : WHO TOXICITY GRADING SCALE FOR DETERMINING THE SEVERITY OF ADVERSE EVENTS (FEB 2003)

**ABBREVIATIONS** (used in the table):

ULN = Upper Limit of Normal LLN = Lower Limit of Normal

 $R_x = Therapy$  IV = Intravenous

 $FEV_1$  = forced expiratory volume in 1 second

#### **ESTIMATING SEVERITY GRADE**

For abnormalities NOT found elsewhere in the Toxicity Tables use the scale below to estimate grade of severity:

| GRADE 1 | Mild | Transient or mild discomfort (<48 hours); no medical intervention/therapy required. |
|---|---|---|
| GRADE 2 | Moderate | Mild to moderate limitation in activity; some assistance may be needed; no or minimal medical intervention/ therapy required. |
| GRADE 3 | Severe | Marked limitation in activity; some assistance usually required; medical intervention/therapy required; hospitalizations possible. |
| GRADE 4 | Potentially life-<br>threatening <sup>a</sup> | Extreme limitation in activity; significant assistance required; significant medical intervention/therapy required; hospitalization or hospice care probable. |

a Revised by the sponsor

#### **COMMENTS REGARDING THE USE OF THESE TABLES**

- For parameters not included in the following Toxicity Tables, sites should refer to the "Guide For Estimating Severity Grade" located above.
- Criteria are generally grouped by body system. Some protocols may have additional protocol-specific grading criteria, which will supersede the use of these tables for specified criteria.

| Item | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|------------|---------|---------|---------|---------|
| Hematology | | | | |

| ItemGrade 1Hemoglobin9.5-10.5 grAbsolute1,000-1,500Neutrophil Count1,000-1,500Platelets75,000-99,0Prothrombin Time (PT)≥1.01 toActivated Partial Thromboplastin Time (aPTT)≥1.01 toFibrinogen≥0.75 toLLNEibrin Split Product20-40 mcg/sMethemoglobin5.0-9.9%Liver Enzymes≥1.25 toAST (SGOT)≥1.25 toULNULNGamma-glutamyltransferaseULNAlkaline≥1.25 toPhosphataseULNAmylase≥1.1 to ≤1.ChemistriesHyponatremia130-135 m | $0/\text{mm}^{3}$ $000/\text{mm}^{3}$ $\leq 1.25 \text{ x}$ $\leq 1.66 \text{ x}$ $\leq 0.99 \text{ x}$ | Grade 2 8.0-9.4 gm/dL 750-999/mm³ 50,000-74,999/mm³ >1.25 to ≤1.50 x ULN >1.66 to ≤2.33 x ULN ≥0.50 to <0.75 x LLN | Grade 3 6.5-7.9 gm/dL 500-749/mm³ 20,000-49,999/mm³ >1.50 to ≤3.00 x ULN >2.33 to ≤3.00 x ULN ≥0.25 to <0.50 x | Grade 4 <6.5 gm/dL <500/mm³ <20,000/mm³ >3.00 x ULN >3.00 x ULN |
|---|---|---|---|---|
| Absolute Neutrophil Count Platelets Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) Fibrin Split Product Methemoglobin Liver Enzymes AST (SGOT) ALT (SGPT) ALT (SGPT) Alkaline Phosphatase Hyponatremia 1,000-1,500 21.01 to ULN ≥1.01 to ULN ≥1.01 to ULN ≥0.75 to LLN ≥0.75 to LLN ≥1.25 to ULN ≥1.25 to ULN Altaline ≥1.25 to ULN Alkaline ≥1.25 to Phosphatase Hyponatremia 130-135 mi | $0/\text{mm}^{3}$ $000/\text{mm}^{3}$ $\leq 1.25 \text{ x}$ $\leq 1.66 \text{ x}$ $\leq 0.99 \text{ x}$ | 750-999/mm³ 50,000-74,999/mm³ >1.25 to ≤1.50 x ULN >1.66 to ≤2.33 x ULN ≥0.50 to <0.75 x LLN | 500-749/mm <sup>3</sup> 20,000-49,999/mm <sup>3</sup> >1.50 to ≤3.00 x ULN >2.33 to ≤3.00 x ULN ≥0.25 to <0.50 x | <500/mm³ <20,000/mm³ >3.00 x ULN >3.00 x ULN |
| Neutrophil Count Platelets 75,000-99,9 Prothrombin Time (PT) ≥1.01 to ULN Activated Partial Thromboplastin Time (aPTT) ≥1.01 to ULN Fibrinogen ≥0.75 to LLN Fibrin Split Product 20-40 mcg/striple Methemoglobin 5.0-9.9% Liver Enzymes AST (SGOT) ≥1.25 to ULN ALT (SGPT) ≥1.25 to ULN Gamma-glutamyltransferase ULN Alkaline ≥1.25 to ULN Amylase ≥1.1 to ≤1. Chemistries Hyponatremia 130-135 m² | $ \begin{array}{c cccc} 0000/\text{mm}^{3} & \\ \leq 1.25 & x \\ \leq 1.66 & x \\ \leq 0.99 & x \end{array} $ | 50,000-74,999/mm³ >1.25 to ≤1.50 x ULN >1.66 to ≤2.33 x ULN ≥0.50 to <0.75 x LLN | 20,000-49,999/mm³ >1.50 to ≤3.00 x ULN >2.33 to ≤3.00 x ULN ≥0.25 to <0.50 x | <20,000/mm³<br>>3.00 x ULN<br>>3.00 x ULN |
| Platelets 75,000-99,0 Prothrombin Time (PT) ≥1.01 to ULN Activated Partial Thromboplastin Time (aPTT) ≥1.01 to ULN Fibrinogen ≥0.75 to LLN Fibrin Split Product Methemoglobin 5.0-9.9% Liver Enzymes AST (SGOT) ≥1.25 to ULN ALT (SGPT) ≥1.25 to ULN Gamma-glutamyltransferase ULN Alkaline Phosphatase ∪LN Amylase ≥1.1 to ≤1. Chemistries Hyponatremia 130-135 m. | ≤1.25 x<br>≤1.66 x<br>≤0.99 x | $>1.25$ to $\le 1.50$ x<br>ULN<br>$>1.66$ to $\le 2.33$ x<br>ULN<br>$\ge 0.50$ to $< 0.75$ x LLN | >1.50 to ≤3.00 x<br>ULN<br>>2.33 to ≤3.00 x<br>ULN<br>≥0.25 to <0.50 x | >3.00 x ULN<br>>3.00 x ULN |
| Prothrombin Time (PT) ULN Activated Partial ≥1.01 to ULN Thromboplastin ULN Time (aPTT) Fibrinogen ≥0.75 to LLN Fibrin Split Product 20-40 meg/ Methemoglobin 5.0-9.9% Liver Enzymes AST (SGOT) ≥1.25 to ULN ALT (SGPT) ≥1.25 to ULN Gamma- ≥1.25 to ULN Alkaline ≥1.25 to ULN Alkaline ≥1.25 to ULN Amylase ≥1.1 to ≤1. Chemistries Hyponatremia 130-135 m | ≤1.25 x<br>≤1.66 x<br>≤0.99 x | $>1.25$ to $\le 1.50$ x<br>ULN<br>$>1.66$ to $\le 2.33$ x<br>ULN<br>$\ge 0.50$ to $< 0.75$ x LLN | >1.50 to ≤3.00 x<br>ULN<br>>2.33 to ≤3.00 x<br>ULN<br>≥0.25 to <0.50 x | >3.00 x ULN<br>>3.00 x ULN |
| (PT) ULN Activated Partial Thromboplastin Time (aPTT) ≥1.01 to ULN Fibrinogen ≥0.75 to LLN Fibrin Split Product 20-40 mcg/s Methemoglobin 5.0-9.9% Liver Enzymes AST (SGOT) ≥1.25 to ULN ALT (SGPT) ≥1.25 to ULN Gamma-glutamyltransferase ULN Alkaline ≥1.25 to ULN Amylase ≥1.1 to ≤1. Chemistries Hyponatremia 130-135 m² | ≤1.66 x<br>≤0.99 x | ULN $>1.66$ to $\le 2.33$ x ULN $\ge 0.50$ to $< 0.75$ x LLN | ULN >2.33 to ≤3.00 x ULN<br>≥0.25 to <0.50 x | >3.00 x ULN |
| Activated Partial Thromboplastin Time (aPTT) ≥1.01 to ULN Fibrinogen ≥0.75 to LLN Fibrin Split Product 20-40 mcg/20-40 mc | ≤0.99 x | >1.66 to ≤2.33 x<br>ULN<br>≥0.50 to <0.75 x LLN | >2.33 to ≤3.00 x<br>ULN<br>≥0.25 to <0.50 x | |
| Thromboplastin Time (aPTT) Fibrinogen ≥0.75 to LLN Fibrin Split Product Methemoglobin Liver Enzymes AST (SGOT) ALT (SGPT) Gamma- glutamyltransferase Alkaline Phosphatase Hyponatremia LUN ULN 21.25 to ULN ≥1.25 to ULN ≥1.25 to ULN ≥1.25 to ULN ≥1.25 to ULN ≥1.25 to ULN Alkaline ≥1.25 to ILN Amylase ≥1.1 to ≤1. | ≤0.99 x | ULN<br>≥0.50 to <0.75 x LLN | ULN ≥0.25 to <0.50 x | |
| Time (aPTT) Fibrinogen ≥0.75 to LLN Fibrin Split Product Methemoglobin Liver Enzymes AST (SGOT) ALT (SGPT) ALT (SGPT) Solution | | ≥0.50 to <0.75 x LLN | ≥0.25 to <0.50 x | <0.25 x L I N |
| Fibrin Split Product 20-40 mcg/Methemoglobin 5.0-9.9% Liver Enzymes AST (SGOT) $\geq$ 1.25 to ULN ALT (SGPT) $\geq$ 1.25 to ULN Gamma- $\geq$ 1.25 to ULN Alkaline $\geq$ 1.25 to Phosphatase ULN Amylase $\geq$ 1.1 to $\leq$ 1. Chemistries Hyponatremia 130-135 m | | | | <0.25 x I I N |
| Fibrin Split Product Methemoglobin 5.0-9.9% Liver Enzymes AST (SGOT) ALT (SGPT) Gamma- glutamyltransferase Alkaline Phosphatase Phosphatase Chemistries Hyponatremia 20-40 mcg/ 20-40 mcg/ 21.25 to ULN ≥1.25 to ULN ≥1.25 to ULN ≥1.25 to ULN 130-135 m | /mL | 41.50 mag/1 | | ·0.23 A LLIN |
| Methemoglobin 5.0-9.9% Liver Enzymes ≥1.25 to ULN ALT (SGPT) ≥1.25 to ULN Gamma-glutamyltransferase ∪LN Alkaline ≥1.25 to ULN Phosphatase ∪LN Amylase ≥1.1 to ≤1. Chemistries Hyponatremia 130-135 m² | /mL | 41.50 mag/T | LLN | |
| Liver EnzymesAST (SGOT) $\geq 1.25$ to<br>ULNALT (SGPT) $\geq 1.25$ to<br>ULNGamma-<br>glutamyltransferase $\geq 1.25$ to<br>ULNAlkaline $\geq 1.25$ to<br>PhosphataseULNAmylase $\geq 1.1$ to $\leq 1$ .ChemistriesHyponatremia $130-135$ m² | | 41-50 mcg/mL | 51-60 mcg/mL | >60 mcg/mL |
| $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | | 10.0-14.9% | 15.0-19.9% | >20.0% |
| $\begin{array}{c c} & ULN \\ \hline ALT (SGPT) & \geq 1.25 \text{ to} \\ \hline ULN \\ \hline Gamma- & \geq 1.25 \text{ to} \\ \hline glutamyltransferase & ULN \\ \hline Alkaline & \geq 1.25 \text{ to} \\ \hline Phosphatase & ULN \\ \hline Amylase & \geq 1.1 \text{ to} \leq 1. \\ \hline \hline \textbf{Chemistries} \\ \hline \\ Hyponatremia & 130-135 \text{ m} \\ \hline \end{array}$ | | | | |
| $ \begin{array}{c cccc} ALT (SGPT) & \geq 1.25 & to \\ ULN & \\ \hline Gamma- & \geq 1.25 & to \\ glutamyltransferase & ULN \\ \hline Alkaline & \geq 1.25 & to \\ Phosphatase & ULN \\ \hline Amylase & \geq 1.1 & to \leq 1. \\ \hline \hline \textbf{Chemistries} & \\ \hline Hyponatremia & 130-135 & m. \\ \hline \end{array} $ | ≤2.50 x | $>2.50$ to $\le 5.00$ x | $>5.00$ to $\le 10.00$ x | >10.00 x ULN |
| Gamma- glutamyltransferase $\ge 1.25$ to glutamyltransferase ULN Alkaline Phosphatase ULN Amylase $\ge 1.25$ to ULN $\ge 1.25$ to Phosphatase ULN $\ge 1.1$ to $\le 1$ . Chemistries Hyponatremia | | ULN | ULN | |
| | ≤2.50 x | $>2.50$ to $\le 5.00$ x | $>5.00$ to $\le 10.00$ x | >10.00 x ULN |
| glutamyltransferase Alkaline Phosphatase ULN Amylase ≥1.25 to ULN Δmylase ≥1.1 to ≤1. Chemistries Hyponatremia 130-135 m | 12.50 | ULN | ULN | . 10.00 |
| Alkaline Phosphatase ULN Amylase ≥1.1 to ≤1. Chemistries Hyponatremia 130-135 m | ≤2.50 x | $>2.50$ to $\le 5.00$ x | >5.00 to ≤10.00 x | >10.00 x ULN |
| Phosphatase ULN Amylase ≥1.1 to ≤1. Chemistries Hyponatremia 130-135 m² | <2.50 ··· | ULN >2.50 to ≤5.00 x | ULN<br>>5.00 to ≤10.00 x | >10.00 x ULN |
| Amylase ≥1.1 to ≤1. Chemistries Hyponatremia 130-135 m | ≥2.30 X | 22.30 to ≤3.00 x<br>ULN | ULN 53.00 to ≤10.00 x | ≥10.00 X ULN |
| Chemistries Hyponatremia 130-135 m | 5 v III N | >1.5 to $\leq$ 2.0 x ULN | >2.0 to ≤5.0 x ULN | >5.0 x ULN |
| Hyponatremia 130-135 m | 3 A OLIV | - 1.5 to _2.0 A CEIV | > 2.0 to _3.0 A CEIV | > 5.0 X CEIV |
| | Ea/L | 123-129 mEq/L | 116-122 mEq/L | <116 mEq/L or |
| Hypernatremia 146-150 m | 242 | 120 129 11124 2 | 110 1 <b>22</b> 11154/2 | mental status |
| Hypernatremia 146-150 m | | | | changes or |
| Hypernatremia 146-150 m | | | | seizures |
| Trypermaticina 140 150 m | Eq/L | 151-157 mEq/L | 158-165 mEq/L | >165 mEq/L or |
| | | | | mental status |
| | | | | changes or |
| | | | | seizures |
| Hypokalemia 3.0-3.4 mE | q/L | 2.5-2.9 mEq/L | 2.0-2.4 mEq/L or | <2.0 mEq/L or |
| | | | intensive | paresis or ileus or |
| | | | replacement Rx | life-threatening |
| | | | required or | arrhythmia |
| | | | hospitalization | |
| Hymanical 5.6.60 E | a/I | 6.1.6.5 mgE = /I | required | >7.0 mE-/I |
| Hyperkalemia 5.6-6.0 mE | q/L | 6.1-6.5 mEq/L | 6.6-7.0 mEq/L | >7.0 mEq/L or life-threatening |
| | | | | arrhythmia |
| Hypoglycemia 55-64 mg/d | | 40-54 mg/dL | 30-39 mg/dL | <30 mg/dL or |
| 11,pogrycenna 33-04 mg/C | 1T. | 10 James all | JO J MIS UL | mental status |
| | iL | | | changes or coma |
| Hyperglycemia 116-160 m | iL | 161-250 mg/dL | 251-500 mg/dL | _ |
| (note if fasting) | | - | I | ketoacidosis or |
| Hyperglycemia 116-160 m, (note if fasting) | 1L | 161-250 mg/dL | 251-500 mg/dL | J |

| Item | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Hypocalcemia | 8.4-7.8 mg/dL | 7.7-7.0 mg/dL | 6.9-6.1 mg/dL | <6.1 mg/dL or |
| (corrected for | | | | life-threatening |
| albumin) | | | | arrhythmia or |
| | | | | tetany |
| Hypercalcemia | 10.6-11.5 mg/dL | 11.6-12.5 mg/dL | 12.6-13.5 mg/dL | >13.5 mg/dL or |
| (corrected for | | | | life-threatening |
| albumin) | | | | arrhythmia |
| Hypomagnesemia | 1.4-1.2 mEq/L | 1.1-0.9 mEq/L | 0.8-0.6 mEq/L | <0.6 mEq/L or |
| | | | | life-threatening |
| | | | | arrhythmia |
| Hypophosphatemia | 2.0-2.4 mg/dL | 1.5-1.9 mg/dL or | 1.0-1.4 mg/dL | <1.0 mg/dL or |
| | | replacement Rx | intensive Rx or | life-threatening |
| | | required | hospitalization | arrhythmia |
| | | | required | |
| Hyperbilirubinemia | ≥1.1 to ≤1.5 x ULN | >1.5 to ≤2.5 x ULN | >2.5 to ≤5.0 x ULN | >5.0 x ULN |
| BUN | $\geq 1.25$ to $\leq 2.50$ x | $>2.50$ to $\le 5.00$ x | $>5.00$ to $\le 10.00$ x | >10.00 x ULN |
| CDIA | ULN | ULN | ULN | . 20 |
| CPK* | 3 to <6 x ULN | 6 to <10 x ULN | 10 to <20 x ULN | ≥20 x ULN |
| Creatinine | ≥1.1 to ≤1.5 x ULN | $>1.5$ to $\le 3.0$ x ULN | >3.0 to ≤6.0 x ULN | >6.0 x ULN or |
| Τ' ψ | 11. 15 1131 | 1.5.4. 2.0. 11131 | 20 | required dialysis |
| Lipase* | 1.1 to <1.5 x ULN | 1.5 to <3.0 x ULN | 3.0 to <5.0 x ULN | ≥5.0 x ULN |
| • | Division of AIDS (DAII | (DS) Table for Grading t | ne Severity of Adult an | d Pediatric Adverse |
| Events, version 2.0, N | November 2014. | | | |
| Urinalysis Proteinuria | 1+ or <0.3% or <3g/L | 2-3+ or 0.3-1.0% or | 4+ or >1.0% or | nephrotic |
| Proteinuria | | 3-10 g/L or | >10 g/L or | * . |
| | or 200 mg – 1 gm | 1-2 gm loss/day | 2-3.5 gm loss/day | syndrome or >3.5 gm loss/day |
| | loss/day | 1-2 gill loss/day | 2-3.5 gm ioss/day | > 5.5 giii ioss/day |
| Hematuria | microscopic only | gross, no clots | gross + clots | obstructive or |
| Tremataria | initerescopie omy | gross, no cross | gross · Gross | required |
| | | | | transfusion |
| Cardiac Dysfunction | 1 | | | |
| Cardiac Rhythm | - | asymptomatic, | recurrent/persistent; | requires Rx |
| | | transient signs, no | • | 1 |
| | | Rx required | • | |
| Hypertension | transient inc. | recurrent, chronic, | requires acute Rx; | requires |
| - | >20 mm; no Rx | > 20 mm, Rx | no hospitalization | hospitalization |
| | | required | | |
| Hypotension | transient orthostatic | symptoms | requires IV fluids; | requires |
| | hypotension, no Rx | correctable with oral | no hospitalization | hospitalization |
| | | fluids Rx | required | |
| Pericarditis | minimal effusion | mild/moderate | symptomatic | tamponade; |
| | | asymptomatic | effusion; pain; ECG | pericardiocentesis |
| | | effusion, no Rx | changes | or surgery |
| | | | | required |
| Hemorrhage, Blood | microscopic/occult | mild, no transfusion | gross blood loss; | massive blood |
| Loss | | | 1-2 units transfused | loss; >3 units |
| | | | | transfused |

Respiratory

| Item | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Cough | transient; no Rx | treatment associated cough; local Rx | uncontrolled | - |
| Bronchospasm,<br>Acute | transient; no Rx<br><80-70% FEV <sub>1</sub><br>(or peak flow) | | no normalization with bronchodilator; FEV <sub>1</sub> 25-50% (or peak flow retractions) | cyanosis: FEV <sub>1</sub> <25% (or peak flow) or intubated |
| Gastrointestinal | | | | |
| Stomatitis | mild discomfort; no limits on activity | some limits on eating/drinking | eating/talking very limited | requires IV fluids |
| Nausea | mild discomfort;<br>maintains<br>reasonable intake | moderate discomfort;<br>intake decreased<br>significantly; some<br>activity limited | severe discomfort;<br>no significant<br>intake; activities<br>limited | minimal fluid<br>intake |
| Vomiting | transient emesis | occasional/moderate<br>vomiting | orthostatic<br>hypotension or IV<br>fluids required | hypotensive shock<br>or hospitalization<br>required for IV<br>fluid therapy |
| Constipation | mild | moderate | severe | distensions<br>w/vomiting |
| Diarrhea | transient 3-4 loose<br>stools/day | 5-7 loose stools/day | orthostatic<br>hypotension or<br>>7 loose stools/day<br>or required IV fluids | hypotensive shock<br>or hospitalization<br>for IV fluid<br>therapy required |
| Neuro & Neuromus | cular | | | |
| Neuro-Cerebellar | slight<br>incoordination<br>dysdiadochokinesis | intention tremor,<br>dysmetria, slurred<br>speech; nystagmus | locomotor ataxia | incapacitated |
| Mood | mild anxiety or<br>depression | moderate anxiety or<br>depression and Rx<br>required | severe anxiety or<br>depression or mania;<br>needs assistance | acute psychosis;<br>incapacitated,<br>requires<br>hospitalization |
| Neuro Control<br>(ADL = activities of<br>daily living) | mild difficulty concentrating; no Rx; mild confusion/agitation; ADL unaffected | moderate<br>confusion/agitation<br>some limitation of<br>ADL; minimal Rx | severe<br>confusion/agitation<br>needs assistance for<br>ADL; Rx required | toxic psychosis;<br>hospitalization |
| Muscle Strength | subjective weakness<br>no objective<br>symptoms/ signs | mild objective<br>signs/symptoms no<br>decrease in function | objective weakness function limited | paralysis |
| Other Parameters | | | | |
| Fever: oral, >12 hours | 37.7-38.5 °C or 100.0-101.5 °F | 38.6-39.5 °C or<br>101.6-102.9 °F | 39.6-40.5 °C or<br>103-105 °F | >40.5 °C or<br>>105 °F |
| Headache | mild, no Rx | transient, moderate;<br>Rx required | severe; responds to<br>initial narcotic<br>therapy | intractable;<br>required repeated<br>narcotic therapy |
| Fatigue | no decrease in ADL | normal activity<br>decreased 25-50% | normal activity<br>decreased >50%<br>can't work | unable to care for self |

| Item | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Allergic Reaction | pruritus without rash | localized urticaria | generalized<br>urticaria;<br>angioedema | anaphylaxis |
| Local Reaction | tenderness or<br>erythema | induration <10 cm or<br>phlebitis or<br>inflammation | induration >10 cm<br>or ulceration | necrosis |
| Mucocutaneous | Erythema; pruritus | diffuse,<br>maculopapular rash,<br>dry desquamation | vesiculation, moist<br>desquamation, or<br>ulceration | exfoliative dermatitis, mucous membrane involvement, or erythema multiforme or suspected Stevens-Johnson or necrosis requiring surgery |

## ATTACHMENT 3. : WHO GRADING SCALE VITAL SIGNS

The following abnormalities are defined for vital signs:

| Abnormality Code | Pulse | SBP* | |
|---|---|---|---|
| Abnormalities on actual ve | alues | | |
| Abnormally low | < 45 bpm | ≤ 50 mmHg | ≤ 90 mmHg |
| Grade 1 or mild | | > 90 mmHg - < 100 mmHg | > 140 mmHg - < 160 mmHg |
| Grade 2 or moderate | - | $\geq 100 \text{ mmHg} - < 110 \text{ mmHg}$ | $\geq$ 160 mmHg - < 180 mmHg |
| Grade 3 or severe | - | ≥ 110 mmHg | ≥ 180 mmHg |
| Abnormally high | ≥ 120 bpm | - | - |

<sup>\*</sup> The classification of AEs related to hypotension and hypertension will be done according to the WHO grading scale

| | Vital Signs p | arameter |
|---|---|---|
| Abnormality Code | Temperature (°C/°F) | |
| Grade 1 or mild | 37.7 - 38.5 °C or<br>100.0 - 101.5 °F | 17-20 |
| Grade 2 or moderate | 38.6 - 39.5 °C or<br>101.6 - 102.9 °F | 21-25 |
| Grade 3 or severe | 39.6 - 40.5 °C or<br>103.0 - 105.0 °F | >25 |
| Grade 4 or potentially life-threatening | >40.5°C or<br>>105.0°F | |

#### ATTACHMENT 4. : ECG ABNORMALITIES

The following abnormalities are defined for ECG:

| | ECG parameter | | | |
|---|---|---|---|---|
| Abnormality Code | HR | PR | QRS | QTcorrected |
| Abnormalities on actual values | | | | |
| Abnormally low | < 45 bpm | < 110 ms | - | - |
| Abnormally high | ≥ 120 bpm | > 220 ms | ≥ 120 ms | - |
| Borderline prolonged QT (males) | - | - | - | $450 \text{ ms} < \text{QTc} \le 480 \text{ ms}$ |
| Borderline prolonged QT (females) | - | - | - | $470 \text{ ms} < \text{QTc} \le 480 \text{ ms}$ |
| Prolonged QT | - | - | - | $480 \text{ ms} < \text{QTc} \le 500 \text{ ms}$ |
| Pathologically prolonged QT | - | - | - | QTc > 500 ms |
| Abnormalities on changes from baseline ( $\Delta QTc$ ) | | | | |
| Normal QTc change | - | - | - | $\Delta QTc < 30 \text{ ms}$ |
| Borderline QTc change | - | - | - | $30 \text{ ms} \leq \Delta QTc \leq 60 \text{ ms}$ |
| Abnormally high QTc change | - | - | - | $\Delta QTc > 60 \text{ ms}$ |

## ATTACHMENT 5. : EQ-5D VALUATION INDEX

| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
|---|---|---|---|---|---|---|---|
| 11111 | 1 | 11242 | 0,498 | 11423 | 0,606 | 11554 | 0,018 |
| 11112 | 0,879 | 11243 | 0,484 | 11424 | 0,437 | 11555 | -0,066 |
| 11113 | 0,848 | 11244 | 0,323 | 11425 | 0,26 | 12111 | 0,846 |
| 11114 | 0,635 | 11245 | 0,157 | 11431 | 0,653 | 12111 | 0,779 |
| 11115 | 0,414 | 11251 | 0,235 | 11432 | 0,596 | 12113 | 0,761 |
| 11113 | 0,837 | 11251 | 0,179 | 11433 | 0,582 | 12114 | 0,548 |
| 11121 | 0,768 | 11252 | 0,179 | 11434 | 0,412 | 12114 | 0,327 |
| 11122 | 0,768 | 11253 | 0,184 | 11434 | 0,412 | 12113 | 0,737 |
| 11123 | 0,537 | 11254 | -0,001 | 11433 | 0,230 | 12121 | 0,678 |
| 11124 | 0,337 | 11311 | 0,883 | 11441 | 0,473 | 12122 | 0,663 |
| 11131 | 0,796 | 11312 | 0,827 | 11443 | 0,404 | 12124 | 0,45<br>0,229 |
| 11132 | 0,74 | 11313 | 0,812 | 11444 | 0,27 | 12125 | |
| 11133 | 0,725 | 11314 | 0,599 | 11445 | 0,131 | 12131 | 0,709 |
| 11134 | 0,512 | 11315 | 0,378 | 11451 | 0,209 | 12132 | 0,653 |
| 11135 | 0,291 | 11321 | 0,785 | 11452 | 0,153 | 12133 | 0,638 |
| 11141 | 0,584 | 11322 | 0,728 | 11453 | 0,138 | 12134 | 0,425 |
| 11142 | 0,527 | 11323 | 0,714 | 11454 | 0,057 | 12135 | 0,204 |
| 11143 | 0,513 | 11324 | 0,501 | 11455 | -0,027 | 12141 | 0,497 |
| 11144 | 0,352 | 11325 | 0,28 | 11511 | 0,556 | 12142 | 0,441 |
| 11145 | 0,186 | 11331 | 0,76 | 11512 | 0,5 | 12143 | 0,426 |
| 11151 | 0,264 | 11332 | 0,704 | 11513 | 0,485 | 12144 | 0,266 |
| 11152 | 0,208 | 11333 | 0,689 | 11514 | 0,404 | 12145 | 0,099 |
| 11153 | 0,193 | 11334 | 0,476 | 11515 | 0,32 | 12151 | 0,177 |
| 11154 | 0,112 | 11335 | 0,255 | 11521 | 0,458 | 12152 | 0,121 |
| 11155 | 0,028 | 11341 | 0,548 | 11522 | 0,401 | 12153 | 0,106 |
| 11211 | 0,906 | 11342 | 0,491 | 11523 | 0,387 | 12154 | 0,025 |
| 11212 | 0,837 | 11343 | 0,477 | 11524 | 0,306 | 12155 | -0,059 |
| 11213 | 0,819 | 11344 | 0,316 | 11525 | 0,222 | 12211 | 0,806 |
| 11214 | 0,606 | 11345 | 0,15 | 11531 | 0,433 | 12212 | 0,748 |
| 11215 | 0,385 | 11351 | 0,228 | 11532 | 0,377 | 12213 | 0,733 |
| 11221 | 0,795 | 11352 | 0,172 | 11533 | 0,362 | 12214 | 0,52 |
| 11222 | 0,736 | 11353 | 0,157 | 11534 | 0,281 | 12215 | 0,299 |
| 11223 | 0,721 | 11354 | 0,076 | 11535 | 0,197 | 12221 | 0,706 |
| 11224 | 0,508 | 11355 | -0,008 | 11541 | 0,328 | 12222 | 0,649 |
| 11225 | 0,287 | 11411 | 0,776 | 11542 | 0,272 | 12223 | 0,634 |
| 11231 | 0,767 | 11412 | 0,719 | 11543 | 0,257 | 12224 | 0,421 |
| 11232 | 0,711 | 11413 | 0,705 | 11544 | 0,176 | 12225 | 0,2 |
| 11233 | 0,696 | 11414 | 0,535 | 11545 | 0,092 | 12231 | 0,681 |
| 11234 | 0,483 | 11415 | 0,359 | 11551 | 0,17 | 12232 | 0,624 |
| 11235 | 0,262 | 11421 | 0,677 | 11552 | 0,114 | 12233 | 0,61 |
| 11241 | 0,555 | 11422 | 0,621 | 11553 | 0,099 | 12234 | 0,397 |
| 12235 | 0,176 | 12424 | 0,35 | 13113 | 0,744 | 13252 | 0,075 |

| - | | | | | | | |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 12241 | 0,468 | 12425 | 0,174 | 13114 | 0,531 | 13253 | 0,06 |
| 12242 | 0,412 | 12431 | 0,566 | 13115 | 0,31 | 13254 | -0,021 |
| 12243 | 0,397 | 12432 | 0,51 | 13121 | 0,717 | 13255 | -0,105 |
| 12244 | 0,237 | 12433 | 0,495 | 13122 | 0,66 | 13311 | 0,779 |
| 12245 | 0,071 | 12434 | 0,325 | 13123 | 0,646 | 13312 | 0,723 |
| 12251 | 0,149 | 12435 | 0,149 | 13124 | 0,433 | 13313 | 0,708 |
| 12252 | 0,092 | 12441 | 0,389 | 13125 | 0,212 | 13314 | 0,495 |
| 12253 | 0,078 | 12442 | 0,332 | 13131 | 0,692 | 13315 | 0,274 |
| 12254 | -0,003 | 12443 | 0,318 | 13132 | 0,636 | 13321 | 0,681 |
| 12255 | -0,088 | 12444 | 0,184 | 13133 | 0,621 | 13322 | 0,624 |
| 12311 | 0,796 | 12445 | 0,044 | 13134 | 0,408 | 13323 | 0,61 |
| 12312 | 0,74 | 12451 | 0,122 | 13135 | 0,187 | 13324 | 0,397 |
| 12313 | 0,725 | 12452 | 0,066 | 13141 | 0,48 | 13325 | 0,176 |
| 12314 | 0,512 | 12453 | 0,051 | 13142 | 0,423 | 13331 | 0,656 |
| 12315 | 0,291 | 12454 | -0,03 | 13143 | 0,409 | 13332 | 0,6 |
| 12321 | 0,698 | 12455 | -0,114 | 13144 | 0,248 | 13333 | 0,585 |
| 12322 | 0,642 | 12511 | 0,469 | 13145 | 0,082 | 13334 | 0,372 |
| 12323 | 0,627 | 12512 | 0,413 | 13151 | 0,16 | 13335 | 0,151 |
| 12324 | 0,414 | 12513 | 0,398 | 13152 | 0,104 | 13341 | 0,444 |
| 12325 | 0,193 | 12514 | 0,317 | 13153 | 0,089 | 13342 | 0,387 |
| 12331 | 0,673 | 12515 | 0,233 | 13154 | 0,008 | 13343 | 0,373 |
| 12332 | 0,617 | 12521 | 0,371 | 13155 | -0,076 | 13344 | 0,212 |
| 12333 | 0,602 | 12522 | 0,315 | 13211 | 0,786 | 13345 | 0,046 |
| 12334 | 0,389 | 12523 | 0,3 | 13212 | 0,73 | 13351 | 0,124 |
| 12335 | 0,168 | 12524 | 0,219 | 13213 | 0,715 | 13352 | 0,068 |
| 12341 | 0,461 | 12525 | 0,135 | 13214 | 0,502 | 13353 | 0,053 |
| 12342 | 0,405 | 12531 | 0,346 | 13215 | 0,281 | 13354 | -0,028 |
| 12343 | 0,39 | 12532 | 0,29 | 13221 | 0,688 | 13355 | -0,112 |
| 12344 | 0,23 | 12533 | 0,275 | 13222 | 0,631 | 13411 | 0,672 |
| 12345 | 0,063 | 12534 | 0,194 | 13223 | 0,617 | 13412 | 0,615 |
| 12351 | 0,141 | 12535 | 0,11 | 13224 | 0,404 | 13413 | 0,601 |
| 12352 | 0,085 | 12541 | 0,241 | 13225 | 0,183 | 13414 | 0,431 |
| 12353 | 0,07 | 12542 | 0,185 | 13231 | 0,663 | 13415 | 0,255 |
| 12354 | -0,011 | 12543 | 0,17 | 13232 | 0,607 | 13421 | 0,573 |
| 12355 | -0,095 | 12544 | 0,089 | 13233 | 0,592 | 13422 | 0,517 |
| 12411 | 0,689 | 12545 | 0,005 | 13234 | 0,379 | 13423 | 0,502 |
| 12412 | 0,633 | 12551 | 0,083 | 13235 | 0,158 | 13424 | 0,333 |
| 12413 | 0,618 | 12552 | 0,027 | 13241 | 0,451 | 13425 | 0,156 |
| 12414 | 0,448 | 12553 | 0,012 | 13242 | 0,394 | 13431 | 0,549 |
| 12415 | 0,272 | 12554 | -0,069 | 13243 | 0,38 | 13432 | 0,492 |
| 12421 | 0,591 | 12555 | -0,153 | 13244 | 0,219 | 13433 | 0,478 |
| 12422 | 0,534 | 13111 | 0,815 | 13245 | 0,053 | 13434 | 0,308 |
| 12423 | 0,52 | 13112 | 0,759 | 13251 | 0,131 | 13435 | 0,132 |
| | , | | , | | , | | , |
| 13441 | 0,371 | 14125 | 0,185 | 14314 | 0,435 | 14453 | 0,007 |

| - | | | | | | | |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 13442 | 0,315 | 14131 | 0,6 | 14315 | 0,247 | 14454 | -0,074 |
| 13443 | 0,3 | 14132 | 0,544 | 14321 | 0,588 | 14455 | -0,158 |
| 13444 | 0,166 | 14133 | 0,529 | 14322 | 0,532 | 14511 | 0,425 |
| 13445 | 0,027 | 14134 | 0,348 | 14323 | 0,517 | 14512 | 0,369 |
| 13451 | 0,105 | 14135 | 0,16 | 14324 | 0,337 | 14513 | 0,354 |
| 13452 | 0,049 | 14141 | 0,414 | 14325 | 0,149 | 14514 | 0,273 |
| 13453 | 0,034 | 14142 | 0,357 | 14331 | 0,564 | 14515 | 0,189 |
| 13454 | -0,047 | 14143 | 0,343 | 14332 | 0,508 | 14521 | 0,327 |
| 13455 | -0,131 | 14144 | 0,202 | 14333 | 0,493 | 14522 | 0,27 |
| 13511 | 0,452 | 14145 | 0,055 | 14334 | 0,312 | 14523 | 0,256 |
| 13512 | 0,396 | 14151 | 0,133 | 14335 | 0,124 | 14524 | 0,175 |
| 13513 | 0,381 | 14152 | 0,077 | 14341 | 0,378 | 14525 | 0,091 |
| 13514 | 0,3 | 14153 | 0,062 | 14342 | 0,321 | 14531 | 0,302 |
| 13515 | 0,216 | 14154 | -0,019 | 14343 | 0,307 | 14532 | 0,246 |
| 13521 | 0,354 | 14155 | -0,103 | 14344 | 0,166 | 14533 | 0,231 |
| 13522 | 0,297 | 14211 | 0,694 | 14345 | 0,019 | 14534 | 0,15 |
| 13523 | 0,283 | 14212 | 0,638 | 14351 | 0,097 | 14535 | 0,066 |
| 13524 | 0,202 | 14213 | 0,623 | 14352 | 0,041 | 14541 | 0,197 |
| 13525 | 0,118 | 14214 | 0,442 | 14353 | 0,026 | 14542 | 0,141 |
| 13531 | 0,329 | 14215 | 0,254 | 14354 | -0,055 | 14543 | 0,126 |
| 13532 | 0,273 | 14221 | 0,596 | 14355 | -0,139 | 14544 | 0,045 |
| 13533 | 0,258 | 14222 | 0,539 | 14411 | 0,601 | 14545 | -0,039 |
| 13534 | 0,177 | 14223 | 0,525 | 14412 | 0,545 | 14551 | 0,039 |
| 13535 | 0,093 | 14224 | 0,344 | 14413 | 0,53 | 14552 | -0,017 |
| 13541 | 0,224 | 14225 | 0,156 | 14414 | 0,382 | 14553 | -0,032 |
| 13542 | 0,168 | 14231 | 0,571 | 14415 | 0,228 | 14554 | -0,113 |
| 13543 | 0,153 | 14232 | 0,515 | 14421 | 0,502 | 14555 | -0,197 |
| 13544 | 0,072 | 14233 | 0,5 | 14422 | 0,446 | 15111 | 0,436 |
| 13545 | -0,012 | 14234 | 0,319 | 14423 | 0,431 | 15112 | 0,38 |
| 13551 | 0,066 | 14235 | 0,131 | 14424 | 0,283 | 15113 | 0,365 |
| 13552 | 0,01 | 14241 | 0,385 | 14425 | 0,13 | 15114 | 0,284 |
| 13553 | -0,005 | 14242 | 0,328 | 14431 | 0,478 | 15115 | 0,2 |
| 13554 | -0,086 | 14243 | 0,314 | 14432 | 0,422 | 15121 | 0,338 |
| 13555 | -0,17 | 14244 | 0,173 | 14433 | 0,407 | 15122 | 0,281 |
| 14111 | 0,723 | 14245 | 0,026 | 14434 | 0,259 | 15123 | 0,267 |
| 14112 | 0,667 | 14251 | 0,104 | 14435 | 0,105 | 15124 | 0,186 |
| 14113 | 0,652 | 14252 | 0,048 | 14441 | 0,318 | 15125 | 0,102 |
| 14114 | 0,471 | 14253 | 0,033 | 14442 | 0,262 | 15131 | 0,313 |
| 14115 | 0,283 | 14254 | -0,048 | 14443 | 0,247 | 15132 | 0,257 |
| 14121 | 0,624 | 14255 | -0,132 | 14444 | 0,126 | 15133 | 0,242 |
| 14122 | 0,568 | 14311 | 0,687 | 14445 | 0 | 15134 | 0,161 |
| 14123 | 0,553 | 14312 | 0,631 | 14451 | 0,078 | 15135 | 0,077 |
| 14124 | 0,373 | 14313 | 0,616 | 14452 | 0,022 | 15141 | 0,208 |
| | • | | , | | , | | • |
| 15142 | 0,152 | 15331 | 0,277 | 21115 | 0,357 | 21254 | 0,026 |

| | | | | | 5,000,000,000 | 1 11141 ) 515 1 141 | |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 15143 | 0,137 | 15332 | 0,221 | 21121 | 0,767 | 21255 | -0,058 |
| 15144 | 0,056 | 15333 | 0,206 | 21122 | 0,708 | 21311 | 0,826 |
| 15145 | -0,028 | 15334 | 0,125 | 21123 | 0,693 | 21312 | 0,77 |
| 15151 | 0,05 | 15335 | 0,041 | 21124 | 0,48 | 21313 | 0,755 |
| 15152 | -0,006 | 15341 | 0,172 | 21125 | 0,259 | 21314 | 0,542 |
| 15153 | -0,021 | 15342 | 0,116 | 21131 | 0,739 | 21315 | 0,321 |
| 15154 | -0,102 | 15343 | 0,101 | 21132 | 0,683 | 21321 | 0,728 |
| 15155 | -0,186 | 15344 | 0,02 | 21133 | 0,668 | 21322 | 0,671 |
| 15211 | 0,407 | 15345 | -0,064 | 21134 | 0,455 | 21323 | 0,657 |
| 15212 | 0,351 | 15351 | 0,014 | 21135 | 0,234 | 21324 | 0,444 |
| 15213 | 0,336 | 15352 | -0,042 | 21141 | 0,527 | 21325 | 0,223 |
| 15214 | 0,255 | 15353 | -0,057 | 21142 | 0,47 | 21331 | 0,703 |
| 15215 | 0,171 | 15354 | -0,138 | 21143 | 0,456 | 21332 | 0,647 |
| 15221 | 0,309 | 15355 | -0,222 | 21144 | 0,296 | 21333 | 0,632 |
| 15222 | 0,252 | 15411 | 0,381 | 21145 | 0,129 | 21334 | 0,419 |
| 15223 | 0,238 | 15412 | 0,325 | 21151 | 0,207 | 21335 | 0,198 |
| 15224 | 0,157 | 15413 | 0,31 | 21152 | 0,151 | 21341 | 0,491 |
| 15225 | 0,073 | 15414 | 0,229 | 21153 | 0,136 | 21342 | 0,434 |
| 15231 | 0,284 | 15415 | 0,145 | 21154 | 0,055 | 21343 | 0,42 |
| 15232 | 0,228 | 15421 | 0,282 | 21155 | -0,029 | 21344 | 0,26 |
| 15233 | 0,213 | 15422 | 0,226 | 21211 | 0,836 | 21345 | 0,093 |
| 15234 | 0,132 | 15423 | 0,211 | 21212 | 0,778 | 21351 | 0,171 |
| 15235 | 0,048 | 15424 | 0,13 | 21213 | 0,762 | 21352 | 0,115 |
| 15241 | 0,179 | 15425 | 0,046 | 21214 | 0,549 | 21353 | 0,1 |
| 15242 | 0,123 | 15431 | 0,258 | 21215 | 0,328 | 21354 | 0,019 |
| 15243 | 0,108 | 15432 | 0,202 | 21221 | 0,735 | 21355 | -0,065 |
| 15244 | 0,027 | 15433 | 0,187 | 21222 | 0,679 | 21411 | 0,719 |
| 15245 | -0,057 | 15434 | 0,106 | 21223 | 0,664 | 21412 | 0,663 |
| 15251 | 0,021 | 15435 | 0,022 | 21224 | 0,451 | 21413 | 0,648 |
| 15252 | -0,035 | 15441 | 0,153 | 21225 | 0,23 | 21414 | 0,478 |
| 15253 | -0,05 | 15442 | 0,097 | 21231 | 0,71 | 21415 | 0,302 |
| 15254 | -0,131 | 15443 | 0,082 | 21232 | 0,654 | 21421 | 0,62 |
| 15255 | -0,215 | 15544 | -0,038 | 21233 | 0,639 | 21422 | 0,564 |
| 15311 | 0,4 | 15545 | -0,122 | 21234 | 0,426 | 21423 | 0,549 |
| 15312 | 0,344 | 15551 | -0,044 | 21235 | 0,205 | 21424 | 0,38 |
| 15313 | 0,329 | 15552 | -0,1 | 21241 | 0,498 | 21425 | 0,204 |
| 15314 | 0,248 | 15553 | -0,115 | 21242 | 0,442 | 21431 | 0,596 |
| 15315 | 0,164 | 15554 | -0,196 | 21243 | 0,427 | 21432 | 0,54 |
| 15321 | 0,302 | 15555 | -0,28 | 21244 | 0,267 | 21433 | 0,525 |
| 15322 | 0,245 | 21111 | 0,877 | 21245 | 0,1 | 21434 | 0,355 |
| 15323 | 0,231 | 21112 | 0,809 | 21251 | 0,178 | 21435 | 0,179 |
| 15324 | 0,15 | 21113 | 0,791 | 21252 | 0,122 | 21441 | 0,419 |
| 15325 | 0,066 | 21114 | 0,578 | 21253 | 0,107 | 21442 | 0,362 |
| 21443 | 0,348 | 22132 | 0,596 | 22321 | 0,641 | 22455 | -0,17 |

| | | | | | | <u>J</u> | |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 21444 | 0,213 | 22133 | 0,582 | 22322 | 0,585 | 22511 | 0,413 |
| 21445 | 0,074 | 22134 | 0,369 | 22323 | 0,57 | 22512 | 0,356 |
| 21451 | 0,152 | 22135 | 0,148 | 22324 | 0,357 | 22513 | 0,342 |
| 21452 | 0,096 | 22141 | 0,44 | 22325 | 0,136 | 22514 | 0,261 |
| 21453 | 0,081 | 22142 | 0,384 | 22331 | 0,617 | 22515 | 0,177 |
| 21454 | 0 | 22143 | 0,369 | 22332 | 0,56 | 22521 | 0,314 |
| 21455 | -0,084 | 22144 | 0,209 | 22333 | 0,546 | 22522 | 0,258 |
| 21511 | 0,499 | 22145 | 0,043 | 22334 | 0,333 | 22523 | 0,243 |
| 21512 | 0,443 | 22151 | 0,121 | 22335 | 0,112 | 22524 | 0,162 |
| 21513 | 0,428 | 22152 | 0,064 | 22341 | 0,404 | 22525 | 0,078 |
| 21514 | 0,347 | 22153 | 0,05 | 22342 | 0,348 | 22531 | 0,29 |
| 21515 | 0,263 | 22154 | -0,031 | 22343 | 0,333 | 22532 | 0,233 |
| 21521 | 0,401 | 22155 | -0,115 | 22344 | 0,173 | 22533 | 0,219 |
| 21522 | 0,344 | 22211 | 0,747 | 22345 | 0,007 | 22534 | 0,138 |
| 21523 | 0,33 | 22212 | 0,691 | 22351 | 0,085 | 22535 | 0,054 |
| 21524 | 0,249 | 22213 | 0,676 | 22352 | 0,028 | 22541 | 0,185 |
| 21525 | 0,165 | 22214 | 0,463 | 22353 | 0,014 | 22542 | 0,128 |
| 21531 | 0,376 | 22215 | 0,242 | 22354 | -0,067 | 22543 | 0,114 |
| 21532 | 0,32 | 22221 | 0,648 | 22355 | -0,151 | 22544 | 0,033 |
| 21533 | 0,305 | 22222 | 0,592 | 22411 | 0,632 | 22545 | -0,051 |
| 21534 | 0,224 | 22223 | 0,577 | 22412 | 0,576 | 22551 | 0,027 |
| 21535 | 0,14 | 22224 | 0,364 | 22413 | 0,561 | 22552 | -0,03 |
| 21541 | 0,271 | 22225 | 0,143 | 22414 | 0,392 | 22553 | -0,044 |
| 21542 | 0,215 | 22231 | 0,624 | 22415 | 0,216 | 22554 | -0,125 |
| 21543 | 0,2 | 22232 | 0,567 | 22421 | 0,534 | 22555 | -0,209 |
| 21544 | 0,119 | 22233 | 0,553 | 22422 | 0,477 | 23111 | 0,758 |
| 21545 | 0,035 | 22234 | 0,34 | 22423 | 0,463 | 23112 | 0,702 |
| 21551 | 0,113 | 22235 | 0,119 | 22424 | 0,293 | 23113 | 0,687 |
| 21552 | 0,057 | 22241 | 0,411 | 22425 | 0,117 | 23114 | 0,474 |
| 21553 | 0,042 | 22242 | 0,355 | 22431 | 0,509 | 23115 | 0,253 |
| 21554 | -0,039 | 22243 | 0,34 | 22432 | 0,453 | 23121 | 0,66 |
| 21555 | -0,123 | 22244 | 0,18 | 22433 | 0,438 | 23122 | 0,603 |
| 22111 | 0,778 | 22245 | 0,014 | 22434 | 0,269 | 23123 | 0,589 |
| 22112 | 0,72 | 22251 | 0,092 | 22435 | 0,093 | 23124 | 0,376 |
| 22113 | 0,705 | 22252 | 0,035 | 22441 | 0,332 | 23125 | 0,155 |
| 22114 | 0,492 | 22253 | 0,021 | 22442 | 0,276 | 23131 | 0,635 |
| 22115 | 0,271 | 22254 | -0,06 | 22443 | 0,261 | 23132 | 0,579 |
| 22121 | 0,678 | 22255 | -0,144 | 22444 | 0,127 | 23133 | 0,564 |
| 22122 | 0,621 | 22311 | 0,74 | 22445 | -0,013 | 23134 | 0,351 |
| 22123 | 0,606 | 22312 | 0,683 | 22451 | 0,066 | 23135 | 0,13 |
| 22124 | 0,393 | 22313 | 0,669 | 22452 | 0,009 | 23141 | 0,423 |
| 22125 | 0,172 | 22314 | 0,456 | 22453 | -0,005 | 23142 | 0,366 |
| 22131 | 0,653 | 22315 | 0,235 | 22454 | -0,086 | 23143 | 0,352 |
| | , | | , | | • | | * |
| 23144 | 0,192 | 23333 | 0,528 | 23522 | 0,24 | 24155 | -0,16 |

| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
|---|---|---|---|---|---|---|---|
| 23145 | 0,025 | 23334 | 0,315 | 23523 | 0,226 | 24211 | 0,637 |
| 23151 | 0,103 | 23335 | 0,094 | 23524 | 0,145 | 24212 | 0,581 |
| 23152 | 0,047 | 23341 | 0,387 | 23525 | 0,061 | 24213 | 0,566 |
| 23153 | 0,032 | 23342 | 0,33 | 23531 | 0,272 | 24214 | 0,385 |
| 23154 | -0,049 | 23343 | 0,316 | 23532 | 0,216 | 24215 | 0,198 |
| 23155 | -0,133 | 23344 | 0,156 | 23533 | 0,201 | 24221 | 0,539 |
| 23211 | 0,729 | 23345 | -0,011 | 23534 | 0,12 | 24222 | 0,482 |
| 23212 | 0,673 | 23351 | 0,067 | 23535 | 0,036 | 24223 | 0,468 |
| 23213 | 0,658 | 23352 | 0,011 | 23541 | 0,167 | 24224 | 0,287 |
| 23214 | 0,445 | 23353 | -0,004 | 23542 | 0,111 | 24225 | 0,099 |
| 23215 | 0,224 | 23354 | -0,085 | 23543 | 0,096 | 24231 | 0,514 |
| 23221 | 0,631 | 23355 | -0,169 | 23544 | 0,015 | 24232 | 0,458 |
| 23222 | 0,575 | 23411 | 0,615 | 23545 | -0,069 | 24233 | 0,443 |
| 23223 | 0,56 | 23412 | 0,559 | 23551 | 0,009 | 24234 | 0,262 |
| 23224 | 0,347 | 23413 | 0,544 | 23552 | -0,047 | 24235 | 0,075 |
| 23225 | 0,126 | 23414 | 0,374 | 23553 | -0,062 | 24241 | 0,328 |
| 23231 | 0,606 | 23415 | 0,198 | 23554 | -0,143 | 24242 | 0,272 |
| 23232 | 0,55 | 23421 | 0,516 | 23555 | -0,227 | 24243 | 0,257 |
| 23233 | 0,535 | 23422 | 0,46 | 24111 | 0,666 | 24244 | 0,116 |
| 23234 | 0,322 | 23423 | 0,445 | 24112 | 0,61 | 24245 | -0,03 |
| 23235 | 0,101 | 23424 | 0,276 | 24113 | 0,595 | 24251 | 0,048 |
| 23241 | 0,394 | 23425 | 0,1 | 24114 | 0,414 | 24252 | -0,009 |
| 23242 | 0,338 | 23431 | 0,492 | 24115 | 0,227 | 24253 | -0,023 |
| 23243 | 0,323 | 23432 | 0,436 | 24121 | 0,568 | 24254 | -0,104 |
| 23244 | 0,163 | 23433 | 0,421 | 24122 | 0,511 | 24255 | -0,188 |
| 23245 | -0,004 | 23434 | 0,251 | 24123 | 0,497 | 24311 | 0,63 |
| 23251 | 0,074 | 23435 | 0,075 | 24124 | 0,316 | 24312 | 0,574 |
| 23252 | 0,018 | 23441 | 0,315 | 24125 | 0,128 | 24313 | 0,559 |
| 23253 | 0,003 | 23442 | 0,258 | 24131 | 0,543 | 24314 | 0,378 |
| 23254 | -0,078 | 23443 | 0,244 | 24132 | 0,487 | 24315 | 0,191 |
| 23255 | -0,162 | 23444 | 0,109 | 24133 | 0,472 | 24321 | 0,532 |
| 23311 | 0,722 | 23445 | -0,03 | 24134 | 0,291 | 24322 | 0,475 |
| 23312 | 0,666 | 23451 | 0,048 | 24135 | 0,104 | 24323 | 0,461 |
| 23313 | 0,651 | 23452 | -0,008 | 24141 | 0,357 | 24324 | 0,28 |
| 23314 | 0,438 | 23453 | -0,023 | 24142 | 0,3 | 24325 | 0,092 |
| 23315 | 0,217 | 23454 | -0,104 | 24143 | 0,286 | 24331 | 0,507 |
| 23321 | 0,624 | 23455 | -0,188 | 24144 | 0,145 | 24332 | 0,451 |
| 23322 | 0,567 | 23511 | 0,395 | 24145 | -0,002 | 24333 | 0,436 |
| 23323 | 0,553 | 23512 | 0,339 | 24151 | 0,077 | 24334 | 0,255 |
| 23324 | 0,34 | 23513 | 0,324 | 24152 | 0,02 | 24335 | 0,068 |
| 23325 | 0,119 | 23514 | 0,243 | 24153 | 0,006 | 24341 | 0,321 |
| 23331 | 0,599 | 23515 | 0,159 | 24154 | -0,076 | 24342 | 0,264 |
| 23332 | 0,543 | 23521 | 0,297 | 24155 | -0,16 | 24343 | 0,25 |
| | , - | | | | , - | | , |
| 24344 | 0,109 | 24533 | 0,175 | 25222 | 0,196 | 25411 | 0,324 |

| - | | | | | 2 1001211 | 1 11141 ) 515 1 141 | |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 24345 | -0,038 | 24534 | 0,094 | 25223 | 0,181 | 25412 | 0,268 |
| 24351 | 0,041 | 24535 | 0,01 | 25224 | 0,1 | 25413 | 0,253 |
| 24352 | -0,016 | 24541 | 0,14 | 25225 | 0,016 | 25414 | 0,172 |
| 24353 | -0,031 | 24542 | 0,084 | 25231 | 0,227 | 25415 | 0,088 |
| 24354 | -0,112 | 24543 | 0,069 | 25232 | 0,171 | 25421 | 0,226 |
| 24355 | -0,196 | 24544 | -0,012 | 25233 | 0,156 | 25422 | 0,169 |
| 24411 | 0,544 | 24545 | -0,096 | 25234 | 0,075 | 25423 | 0,155 |
| 24412 | 0,488 | 24551 | -0,018 | 25235 | -0,009 | 25424 | 0,074 |
| 24413 | 0,473 | 24552 | -0,074 | 25241 | 0,122 | 25425 | -0,01 |
| 24414 | 0,325 | 24553 | -0,089 | 25242 | 0,066 | 25431 | 0,201 |
| 24415 | 0,172 | 24554 | -0,17 | 25243 | 0,051 | 25432 | 0,145 |
| 24421 | 0,446 | 24555 | -0,254 | 25244 | -0,03 | 25433 | 0,13 |
| 24422 | 0,389 | 25111 | 0,379 | 25245 | -0,114 | 25434 | 0,049 |
| 24423 | 0,375 | 25112 | 0,323 | 25251 | -0,036 | 25435 | -0,035 |
| 24424 | 0,227 | 25113 | 0,308 | 25252 | -0,092 | 25441 | 0,096 |
| 24425 | 0,073 | 25114 | 0,227 | 25253 | -0,107 | 25442 | 0,04 |
| 24431 | 0,421 | 25115 | 0,143 | 25254 | -0,188 | 25443 | 0,025 |
| 24432 | 0,365 | 25121 | 0,281 | 25255 | -0,272 | 25444 | -0,056 |
| 24433 | 0,35 | 25122 | 0,224 | 25311 | 0,343 | 25445 | -0,14 |
| 24434 | 0,202 | 25123 | 0,21 | 25312 | 0,287 | 25451 | -0,062 |
| 24435 | 0,049 | 25124 | 0,129 | 25313 | 0,272 | 25452 | -0,118 |
| 24441 | 0,262 | 25125 | 0,045 | 25314 | 0,191 | 25453 | -0,133 |
| 24442 | 0,205 | 25131 | 0,256 | 25315 | 0,107 | 25454 | -0,214 |
| 24443 | 0,191 | 25132 | 0,2 | 25321 | 0,245 | 25455 | -0,298 |
| 24444 | 0,069 | 25133 | 0,185 | 25322 | 0,188 | 25511 | 0,285 |
| 24445 | -0,057 | 25134 | 0,104 | 25323 | 0,174 | 25512 | 0,229 |
| 24451 | 0,022 | 25135 | 0,02 | 25324 | 0,093 | 25513 | 0,214 |
| 24452 | -0,035 | 25141 | 0,151 | 25325 | 0,009 | 25514 | 0,133 |
| 24453 | -0,05 | 25142 | 0,095 | 25331 | 0,22 | 25515 | 0,049 |
| 24454 | -0,131 | 25143 | 0,08 | 25332 | 0,164 | 25521 | 0,187 |
| 24455 | -0,215 | 25144 | -0,001 | 25333 | 0,149 | 25522 | 0,13 |
| 24511 | 0,369 | 25145 | -0,085 | 25334 | 0,068 | 25523 | 0,116 |
| 24512 | 0,312 | 25151 | -0,007 | 25335 | -0,016 | 25524 | 0,035 |
| 24513 | 0,298 | 25152 | -0,063 | 25341 | 0,115 | 25525 | -0,049 |
| 24514 | 0,217 | 25153 | -0,078 | 25342 | 0,059 | 25531 | 0,162 |
| 24515 | 0,133 | 25154 | -0,159 | 25343 | 0,044 | 25532 | 0,106 |
| 24521 | 0,27 | 25155 | -0,243 | 25344 | -0,037 | 25533 | 0,091 |
| 24522 | 0,214 | 25211 | 0,35 | 25345 | -0,121 | 25534 | 0,01 |
| 24523 | 0,199 | 25212 | 0,294 | 25351 | -0,043 | 25535 | -0,074 |
| 24524 | 0,118 | 25213 | 0,279 | 25352 | -0,099 | 25541 | 0,057 |
| 24525 | 0,034 | 25214 | 0,198 | 25353 | -0,114 | 25542 | 0,001 |
| 24531 | 0,246 | 25215 | 0,114 | 25354 | -0,195 | 25543 | -0,014 |
| 24532 | 0,189 | 25221 | 0,252 | 25355 | -0,279 | 25544 | -0,095 |
| 25545 | -0,179 | 31234 | 0,414 | 31423 | 0,537 | 32112 | 0,707 |

| | | | | | Statistical | Analysis i lai | 1 030230721 1 |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 25551 | -0,101 | 31235 | 0,193 | 31424 | 0,368 | 32113 | 0,692 |
| 25552 | -0,157 | 31241 | 0,486 | 31425 | 0,191 | 32114 | 0,479 |
| 25553 | -0,172 | 31242 | 0,429 | 31431 | 0,584 | 32115 | 0,258 |
| 25554 | -0,253 | 31243 | 0,415 | 31432 | 0,527 | 32121 | 0,665 |
| 25555 | -0,337 | 31244 | 0,254 | 31433 | 0,513 | 32122 | 0,609 |
| 31111 | 0,85 | 31245 | 0,088 | 31434 | 0,343 | 32123 | 0,594 |
| 31112 | 0,794 | 31251 | 0,166 | 31435 | 0,167 | 32124 | 0,381 |
| 31113 | 0,779 | 31252 | 0,11 | 31441 | 0,406 | 32125 | 0,16 |
| 31114 | 0,566 | 31253 | 0,095 | 31442 | 0,35 | 32131 | 0,64 |
| 31115 | 0,345 | 31254 | 0,014 | 31443 | 0,335 | 32132 | 0,584 |
| 31121 | 0,752 | 31255 | -0,07 | 31444 | 0,201 | 32133 | 0,569 |
| 31122 | 0,695 | 31311 | 0,814 | 31445 | 0,062 | 32134 | 0,356 |
| 31123 | 0,681 | 31312 | 0,758 | 31451 | 0,14 | 32135 | 0,135 |
| 31124 | 0,468 | 31313 | 0,743 | 31452 | 0,084 | 32141 | 0,428 |
| 31125 | 0,247 | 31314 | 0,53 | 31453 | 0,069 | 32142 | 0,372 |
| 31131 | 0,727 | 31315 | 0,309 | 31454 | -0,012 | 32143 | 0,357 |
| 31132 | 0,671 | 31321 | 0,716 | 31455 | -0,096 | 32144 | 0,197 |
| 31133 | 0,656 | 31322 | 0,659 | 31511 | 0,487 | 32145 | 0,03 |
| 31134 | 0,443 | 31323 | 0,645 | 31512 | 0,431 | 32151 | 0,108 |
| 31135 | 0,222 | 31324 | 0,432 | 31513 | 0,416 | 32152 | 0,052 |
| 31141 | 0,515 | 31325 | 0,211 | 31514 | 0,335 | 32153 | 0,037 |
| 31142 | 0,458 | 31331 | 0,691 | 31515 | 0,251 | 32154 | -0,044 |
| 31143 | 0,444 | 31332 | 0,635 | 31521 | 0,389 | 32155 | -0,128 |
| 31144 | 0,283 | 31333 | 0,62 | 31522 | 0,332 | 32211 | 0,735 |
| 31145 | 0,117 | 31334 | 0,407 | 31523 | 0,318 | 32212 | 0,678 |
| 31151 | 0,195 | 31335 | 0,186 | 31524 | 0,237 | 32213 | 0,664 |
| 31152 | 0,139 | 31341 | 0,479 | 31525 | 0,153 | 32214 | 0,451 |
| 31153 | 0,124 | 31342 | 0,422 | 31531 | 0,364 | 32215 | 0,23 |
| 31154 | 0,043 | 31343 | 0,408 | 31532 | 0,308 | 32221 | 0,636 |
| 31155 | -0,041 | 31344 | 0,247 | 31533 | 0,293 | 32222 | 0,58 |
| 31211 | 0,821 | 31345 | 0,081 | 31534 | 0,212 | 32223 | 0,565 |
| 31212 | 0,765 | 31351 | 0,159 | 31535 | 0,128 | 32224 | 0,352 |
| 31213 | 0,75 | 31352 | 0,103 | 31541 | 0,259 | 32225 | 0,131 |
| 31214 | 0,537 | 31353 | 0,088 | 31542 | 0,203 | 32231 | 0,612 |
| 31215 | 0,316 | 31354 | 0,007 | 31543 | 0,188 | 32232 | 0,555 |
| 31221 | 0,723 | 31355 | -0,077 | 31544 | 0,107 | 32233 | 0,541 |
| 31222 | 0,666 | 31411 | 0,707 | 31545 | 0,023 | 32234 | 0,328 |
| 31223 | 0,652 | 31412 | 0,65 | 31551 | 0,101 | 32235 | 0,107 |
| 31224 | 0,439 | 31413 | 0,636 | 31552 | 0,045 | 32241 | 0,399 |
| 31225 | 0,218 | 31414 | 0,466 | 31553 | 0,03 | 32242 | 0,343 |
| 31231 | 0,698 | 31415 | 0,29 | 31554 | -0,051 | 32243 | 0,328 |
| 31232 | 0,642 | 31421 | 0,608 | 31555 | -0,135 | 32244 | 0,168 |
| 31233 | 0,627 | 31422 | 0,552 | 32111 | 0,763 | 32245 | 0,002 |
| 32251 | 0,08 | 32435 | 0,08 | 33124 | 0,364 | 33313 | 0,639 |

| - | | | | | 5,44,15,41,441 | 1 11101 ) 010 1 101 | |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 32252 | 0,023 | 32441 | 0,32 | 33125 | 0,143 | 33314 | 0,426 |
| 32253 | 0,009 | 32442 | 0,263 | 33131 | 0,623 | 33315 | 0,205 |
| 32254 | -0,072 | 32443 | 0,249 | 33132 | 0,567 | 33321 | 0,612 |
| 32255 | -0,157 | 32444 | 0,115 | 33133 | 0,552 | 33322 | 0,555 |
| 32311 | 0,727 | 32445 | -0,025 | 33134 | 0,339 | 33323 | 0,541 |
| 32312 | 0,671 | 32451 | 0,053 | 33135 | 0,118 | 33324 | 0,328 |
| 32313 | 0,656 | 32452 | -0,003 | 33141 | 0,411 | 33325 | 0,107 |
| 32314 | 0,443 | 32453 | -0,018 | 33142 | 0,354 | 33331 | 0,587 |
| 32315 | 0,222 | 32454 | -0,099 | 33143 | 0,34 | 33332 | 0,531 |
| 32321 | 0,629 | 32455 | -0,183 | 33144 | 0,179 | 33333 | 0,516 |
| 32322 | 0,573 | 32511 | 0,4 | 33145 | 0,013 | 33334 | 0,303 |
| 32323 | 0,558 | 32512 | 0,344 | 33151 | 0,091 | 33335 | 0,082 |
| 32324 | 0,345 | 32513 | 0,329 | 33152 | 0,035 | 33341 | 0,375 |
| 32325 | 0,124 | 32514 | 0,248 | 33153 | 0,02 | 33342 | 0,318 |
| 32331 | 0,604 | 32515 | 0,164 | 33154 | -0,061 | 33343 | 0,304 |
| 32332 | 0,548 | 32521 | 0,302 | 33155 | -0,145 | 33344 | 0,143 |
| 32333 | 0,533 | 32522 | 0,246 | 33211 | 0,717 | 33345 | -0,023 |
| 32334 | 0,32 | 32523 | 0,231 | 33212 | 0,661 | 33351 | 0,055 |
| 32335 | 0,099 | 32524 | 0,15 | 33213 | 0,646 | 33352 | -0,001 |
| 32341 | 0,392 | 32525 | 0,066 | 33214 | 0,433 | 33353 | -0,016 |
| 32342 | 0,336 | 32531 | 0,277 | 33215 | 0,212 | 33354 | -0,097 |
| 32343 | 0,321 | 32532 | 0,221 | 33221 | 0,619 | 33355 | -0,181 |
| 32344 | 0,161 | 32533 | 0,206 | 33222 | 0,562 | 33411 | 0,603 |
| 32345 | -0,006 | 32534 | 0,125 | 33223 | 0,548 | 33412 | 0,546 |
| 32351 | 0,072 | 32535 | 0,041 | 33224 | 0,335 | 33413 | 0,532 |
| 32352 | 0,016 | 32541 | 0,172 | 33225 | 0,114 | 33414 | 0,362 |
| 32353 | 0,001 | 32542 | 0,116 | 33231 | 0,594 | 33415 | 0,186 |
| 32354 | -0,08 | 32543 | 0,101 | 33232 | 0,538 | 33421 | 0,504 |
| 32355 | -0,164 | 32544 | 0,02 | 33233 | 0,523 | 33422 | 0,448 |
| 32411 | 0,62 | 32545 | -0,064 | 33234 | 0,31 | 33423 | 0,433 |
| 32412 | 0,564 | 32551 | 0,014 | 33235 | 0,089 | 33424 | 0,264 |
| 32413 | 0,549 | 32552 | -0,042 | 33241 | 0,382 | 33425 | 0,087 |
| 32414 | 0,379 | 32553 | -0,057 | 33242 | 0,325 | 33431 | 0,48 |
| 32415 | 0,203 | 32554 | -0,138 | 33243 | 0,311 | 33432 | 0,423 |
| 32421 | 0,522 | 32555 | -0,222 | 33244 | 0,15 | 33433 | 0,409 |
| 32422 | 0,465 | 33111 | 0,746 | 33245 | -0,016 | 33434 | 0,239 |
| 32423 | 0,451 | 33112 | 0,69 | 33251 | 0,062 | 33435 | 0,063 |
| 32424 | 0,281 | 33113 | 0,675 | 33252 | 0,006 | 33441 | 0,302 |
| 32425 | 0,105 | 33114 | 0,462 | 33253 | -0,009 | 33442 | 0,246 |
| 32431 | 0,497 | 33115 | 0,241 | 33254 | -0,09 | 33443 | 0,231 |
| 32432 | 0,441 | 33121 | 0,648 | 33255 | -0,174 | 33444 | 0,097 |
| 32433 | 0,426 | 33122 | 0,591 | 33311 | 0,71 | 33445 | -0,042 |
| 32434 | 0,256 | 33123 | 0,577 | 33312 | 0,654 | 33451 | 0,036 |
| 33452 | -0,02 | 34141 | 0,345 | 34325 | 0,08 | 34514 | 0,204 |

| - | | | | | 2 4441241241 | 1 11101 ) 010 1 1011 | . 00 020 0 . 21 23 |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 33453 | -0,035 | 34142 | 0,288 | 34331 | 0,495 | 34515 | 0,12 |
| 33454 | -0,116 | 34143 | 0,274 | 34332 | 0,439 | 34521 | 0,258 |
| 33455 | -0,2 | 34144 | 0,133 | 34333 | 0,424 | 34522 | 0,201 |
| 33511 | 0,383 | 34145 | -0,014 | 34334 | 0,243 | 34523 | 0,187 |
| 33512 | 0,327 | 34151 | 0,064 | 34335 | 0,055 | 34524 | 0,106 |
| 33513 | 0,312 | 34152 | 0,008 | 34341 | 0,309 | 34525 | 0,022 |
| 33514 | 0,231 | 34153 | -0,007 | 34342 | 0,252 | 34531 | 0,233 |
| 33515 | 0,147 | 34154 | -0,088 | 34343 | 0,238 | 34532 | 0,177 |
| 33521 | 0,285 | 34155 | -0,172 | 34344 | 0,097 | 34533 | 0,162 |
| 33522 | 0,228 | 34211 | 0,625 | 34345 | -0,05 | 34534 | 0,081 |
| 33523 | 0,214 | 34212 | 0,569 | 34351 | 0,028 | 34535 | -0,003 |
| 33524 | 0,133 | 34213 | 0,554 | 34352 | -0,028 | 34541 | 0,128 |
| 33525 | 0,049 | 34214 | 0,373 | 34353 | -0,043 | 34542 | 0,072 |
| 33531 | 0,26 | 34215 | 0,185 | 34354 | -0,124 | 34543 | 0,057 |
| 33532 | 0,204 | 34221 | 0,527 | 34355 | -0,208 | 34544 | -0,024 |
| 33533 | 0,189 | 34222 | 0,47 | 34411 | 0,532 | 34545 | -0,108 |
| 33534 | 0,108 | 34223 | 0,456 | 34412 | 0,476 | 34551 | -0,03 |
| 33535 | 0,024 | 34224 | 0,275 | 34413 | 0,461 | 34552 | -0,086 |
| 33541 | 0,155 | 34225 | 0,087 | 34414 | 0,313 | 34553 | -0,101 |
| 33542 | 0,099 | 34231 | 0,502 | 34415 | 0,159 | 34554 | -0,182 |
| 33543 | 0,084 | 34232 | 0,446 | 34421 | 0,433 | 34555 | -0,266 |
| 33544 | 0,003 | 34233 | 0,431 | 34422 | 0,377 | 35111 | 0,367 |
| 33545 | -0,081 | 34234 | 0,25 | 34423 | 0,362 | 35112 | 0,311 |
| 33551 | -0,003 | 34235 | 0,062 | 34424 | 0,214 | 35113 | 0,296 |
| 33552 | -0,059 | 34241 | 0,316 | 34425 | 0,061 | 35114 | 0,215 |
| 33553 | -0,074 | 34242 | 0,259 | 34431 | 0,409 | 35115 | 0,131 |
| 33554 | -0,155 | 34243 | 0,245 | 34432 | 0,353 | 35121 | 0,269 |
| 33555 | -0,239 | 34244 | 0,104 | 34433 | 0,338 | 35122 | 0,212 |
| 34111 | 0,654 | 34245 | -0,043 | 34434 | 0,19 | 35123 | 0,198 |
| 34112 | 0,598 | 34251 | 0,035 | 34435 | 0,036 | 35124 | 0,117 |
| 34113 | 0,583 | 34252 | -0,021 | 34441 | 0,249 | 35125 | 0,033 |
| 34114 | 0,402 | 34253 | -0,036 | 34442 | 0,193 | 35131 | 0,244 |
| 34115 | 0,214 | 34254 | -0,117 | 34443 | 0,178 | 35132 | 0,188 |
| 34121 | 0,555 | 34255 | -0,201 | 34444 | 0,057 | 35133 | 0,173 |
| 34122 | 0,499 | 34311 | 0,618 | 34445 | -0,069 | 35134 | 0,092 |
| 34123 | 0,484 | 34312 | 0,562 | 34451 | 0,009 | 35135 | 0,008 |
| 34124 | 0,304 | 34313 | 0,547 | 34452 | -0,047 | 35141 | 0,139 |
| 34125 | 0,116 | 34314 | 0,366 | 34453 | -0,062 | 35142 | 0,083 |
| 34131 | 0,531 | 34315 | 0,178 | 34454 | -0,143 | 35143 | 0,068 |
| 34132 | 0,475 | 34321 | 0,519 | 34455 | -0,227 | 35144 | -0,013 |
| 34133 | 0,46 | 34322 | 0,463 | 34511 | 0,356 | 35145 | -0,097 |
| 34134 | 0,279 | 34323 | 0,448 | 34512 | 0,3 | 35151 | -0,019 |
| 34135 | 0,091 | 34324 | 0,268 | 34513 | 0,285 | 35152 | -0,075 |
| 35153 | -0,09 | 35342 | 0,047 | 35531 | 0,15 | 41215 | 0,299 |

| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
|---|---|---|---|---|---|---|---|
| 35154 | -0,171 | 35343 | 0,032 | 35532 | 0,094 | 41221 | 0,686 |
| 35155 | -0,255 | 35344 | -0,049 | 35533 | 0,079 | 41222 | 0,629 |
| 35211 | 0,338 | 35345 | -0,133 | 35534 | -0,002 | 41223 | 0,615 |
| 35212 | 0,282 | 35351 | -0,055 | 35535 | -0,086 | 41224 | 0,411 |
| 35213 | 0,267 | 35352 | -0,111 | 35541 | 0,045 | 41225 | 0,2 |
| 35214 | 0,186 | 35353 | -0,126 | 35542 | -0,011 | 41231 | 0,661 |
| 35215 | 0,102 | 35354 | -0,207 | 35543 | -0,026 | 41232 | 0,605 |
| 35221 | 0,24 | 35355 | -0,291 | 35544 | -0,107 | 41233 | 0,59 |
| 35222 | 0,183 | 35411 | 0,312 | 35545 | -0,191 | 41234 | 0,387 |
| 35223 | 0,169 | 35412 | 0,256 | 35551 | -0,113 | 41235 | 0,176 |
| 35224 | 0,088 | 35413 | 0,241 | 35552 | -0,169 | 41241 | 0,456 |
| 35225 | 0,004 | 35414 | 0,16 | 35553 | -0,184 | 41242 | 0,4 |
| 35231 | 0,215 | 35415 | 0,076 | 35554 | -0,265 | 41243 | 0,385 |
| 35232 | 0,159 | 35421 | 0,213 | 35555 | -0,349 | 41244 | 0,231 |
| 35233 | 0,144 | 35422 | 0,157 | 41111 | 0,813 | 41245 | 0,07 |
| 35234 | 0,063 | 35423 | 0,142 | 41112 | 0,757 | 41251 | 0,149 |
| 35235 | -0,021 | 35424 | 0,061 | 41113 | 0,742 | 41252 | 0,092 |
| 35241 | 0,11 | 35425 | -0,023 | 41114 | 0,539 | 41253 | 0,078 |
| 35242 | 0,054 | 35431 | 0,189 | 41115 | 0,327 | 41254 | -0,004 |
| 35243 | 0,039 | 35432 | 0,133 | 41121 | 0,714 | 41255 | -0,088 |
| 35244 | -0,042 | 35433 | 0,118 | 41122 | 0,658 | 41311 | 0,777 |
| 35245 | -0,126 | 35434 | 0,037 | 41123 | 0,643 | 41312 | 0,721 |
| 35251 | -0,048 | 35435 | -0,047 | 41124 | 0,44 | 41313 | 0,706 |
| 35252 | -0,104 | 35441 | 0,084 | 41125 | 0,229 | 41314 | 0,503 |
| 35253 | -0,119 | 35442 | 0,028 | 41131 | 0,69 | 41315 | 0,291 |
| 35254 | -0,2 | 35443 | 0,013 | 41132 | 0,634 | 41321 | 0,678 |
| 35255 | -0,284 | 35444 | -0,068 | 41133 | 0,619 | 41322 | 0,622 |
| 35311 | 0,331 | 35445 | -0,152 | 41134 | 0,416 | 41323 | 0,607 |
| 35312 | 0,275 | 35451 | -0,074 | 41135 | 0,204 | 41324 | 0,404 |
| 35313 | 0,26 | 35452 | -0,13 | 41141 | 0,485 | 41325 | 0,193 |
| 35314 | 0,179 | 35453 | -0,145 | 41142 | 0,429 | 41331 | 0,654 |
| 35315 | 0,095 | 35454 | -0,226 | 41143 | 0,414 | 41332 | 0,598 |
| 35321 | 0,233 | 35455 | -0,31 | 41144 | 0,26 | 41333 | 0,583 |
| 35322 | 0,176 | 35511 | 0,273 | 41145 | 0,099 | 41334 | 0,38 |
| 35323 | 0,162 | 35512 | 0,217 | 41151 | 0,177 | 41335 | 0,168 |
| 35324 | 0,081 | 35513 | 0,202 | 41152 | 0,121 | 41341 | 0,449 |
| 35325 | -0,004 | 35514 | 0,121 | 41153 | 0,106 | 41342 | 0,393 |
| 35331 | 0,208 | 35515 | 0,037 | 41154 | 0,025 | 41343 | 0,378 |
| 35332 | 0,152 | 35521 | 0,175 | 41155 | -0,059 | 41344 | 0,224 |
| 35333 | 0,137 | 35522 | 0,118 | 41211 | 0,784 | 41345 | 0,063 |
| 35334 | 0,056 | 35523 | 0,104 | 41212 | 0,728 | 41351 | 0,141 |
| 35335 | -0,028 | 35524 | 0,023 | 41213 | 0,713 | 41352 | 0,085 |
| 35341 | 0,103 | 35525 | -0,062 | 41214 | 0,51 | 41353 | 0,07 |
| | , - | | , | | , | | , |
| 41354 | -0,011 | 41543 | 0,17 | 42232 | 0,518 | 42421 | 0,491 |

| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
|---|---|---|---|---|---|---|---|
| 41355 | -0,095 | 41544 | 0,089 | 42233 | 0,504 | 42422 | 0,434 |
| 41411 | 0,676 | 41545 | 0,005 | 42234 | 0,3 | 42423 | 0,42 |
| 41412 | 0,62 | 41551 | 0,083 | 42235 | 0,089 | 42424 | 0,257 |
| 41413 | 0,605 | 41552 | 0,027 | 42241 | 0,37 | 42425 | 0,087 |
| 41414 | 0,442 | 41553 | 0,012 | 42242 | 0,313 | 42431 | 0,466 |
| 41415 | 0,272 | 41554 | -0,069 | 42243 | 0,299 | 42432 | 0,41 |
| 41421 | 0,577 | 41555 | -0,153 | 42244 | 0,144 | 42433 | 0,395 |
| 41422 | 0,521 | 42111 | 0,726 | 42245 | -0,016 | 42434 | 0,232 |
| 41423 | 0,506 | 42112 | 0,67 | 42251 | 0,062 | 42435 | 0,063 |
| 41424 | 0,343 | 42113 | 0,655 | 42252 | 0,006 | 42441 | 0,294 |
| 41425 | 0,174 | 42114 | 0,452 | 42253 | -0,009 | 42442 | 0,238 |
| 41431 | 0,553 | 42115 | 0,241 | 42254 | -0,09 | 42443 | 0,223 |
| 41432 | 0,497 | 42121 | 0,628 | 42255 | -0,174 | 42444 | 0,093 |
| 41433 | 0,482 | 42122 | 0,572 | 42311 | 0,69 | 42445 | -0,042 |
| 41434 | 0,319 | 42123 | 0,557 | 42312 | 0,634 | 42451 | 0,036 |
| 41435 | 0,149 | 42124 | 0,353 | 42313 | 0,619 | 42452 | -0,021 |
| 41441 | 0,381 | 42125 | 0,142 | 42314 | 0,416 | 42453 | -0,035 |
| 41442 | 0,325 | 42131 | 0,603 | 42315 | 0,205 | 42454 | -0,116 |
| 41443 | 0,31 | 42132 | 0,547 | 42321 | 0,592 | 42455 | -0,2 |
| 41444 | 0,18 | 42133 | 0,532 | 42322 | 0,536 | 42511 | 0,383 |
| 41445 | 0,044 | 42134 | 0,329 | 42323 | 0,521 | 42512 | 0,326 |
| 41451 | 0,122 | 42135 | 0,118 | 42324 | 0,317 | 42513 | 0,312 |
| 41452 | 0,066 | 42141 | 0,399 | 42325 | 0,106 | 42514 | 0,231 |
| 41453 | 0,051 | 42142 | 0,342 | 42331 | 0,567 | 42515 | 0,147 |
| 41454 | -0,03 | 42143 | 0,328 | 42332 | 0,511 | 42521 | 0,284 |
| 41455 | -0,114 | 42144 | 0,173 | 42333 | 0,496 | 42522 | 0,228 |
| 41511 | 0,469 | 42145 | 0,013 | 42334 | 0,293 | 42523 | 0,213 |
| 41512 | 0,413 | 42151 | 0,091 | 42335 | 0,082 | 42524 | 0,132 |
| 41513 | 0,398 | 42152 | 0,034 | 42341 | 0,363 | 42525 | 0,048 |
| 41514 | 0,317 | 42153 | 0,02 | 42342 | 0,306 | 42531 | 0,26 |
| 41515 | 0,233 | 42154 | -0,061 | 42343 | 0,292 | 42532 | 0,203 |
| 41521 | 0,371 | 42155 | -0,145 | 42344 | 0,137 | 42533 | 0,189 |
| 41522 | 0,315 | 42211 | 0,698 | 42345 | -0,023 | 42534 | 0,108 |
| 41523 | 0,3 | 42212 | 0,641 | 42351 | 0,055 | 42535 | 0,024 |
| 41524 | 0,219 | 42213 | 0,627 | 42352 | -0,002 | 42541 | 0,155 |
| 41525 | 0,135 | 42214 | 0,423 | 42353 | -0,016 | 42542 | 0,098 |
| 41531 | 0,346 | 42215 | 0,212 | 42354 | -0,097 | 42543 | 0,084 |
| 41532 | 0,29 | 42221 | 0,599 | 42355 | -0,181 | 42544 | 0,003 |
| 41533 | 0,275 | 42222 | 0,543 | 42411 | 0,589 | 42545 | -0,081 |
| 41534 | 0,194 | 42223 | 0,528 | 42412 | 0,533 | 42551 | -0,003 |
| 41535 | 0,11 | 42224 | 0,325 | 42413 | 0,518 | 42552 | -0,06 |
| 41541 | 0,241 | 42225 | 0,113 | 42414 | 0,355 | 42553 | -0,074 |
| 41542 | 0,185 | 42231 | 0,575 | 42415 | 0,186 | 42554 | -0,155 |
| 42555 | -0,239 | 43244 | 0,127 | 43433 | 0,378 | 44122 | 0,467 |

| | | | | | 5,000,000,000 | 1 11141 ) 515 1 141 | |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 43111 | 0,709 | 43245 | -0,034 | 43434 | 0,215 | 44123 | 0,452 |
| 43112 | 0,653 | 43251 | 0,045 | 43435 | 0,045 | 44124 | 0,278 |
| 43113 | 0,638 | 43252 | -0,012 | 43441 | 0,277 | 44125 | 0,098 |
| 43114 | 0,435 | 43253 | -0,027 | 43442 | 0,221 | 44131 | 0,499 |
| 43115 | 0,223 | 43254 | -0,108 | 43443 | 0,206 | 44132 | 0,442 |
| 43121 | 0,61 | 43255 | -0,192 | 43444 | 0,076 | 44133 | 0,428 |
| 43122 | 0,554 | 43311 | 0,673 | 43445 | -0,06 | 44134 | 0,254 |
| 43123 | 0,539 | 43312 | 0,617 | 43451 | 0,018 | 44135 | 0,074 |
| 43124 | 0,336 | 43313 | 0,602 | 43452 | -0,038 | 44141 | 0,318 |
| 43125 | 0,125 | 43314 | 0,399 | 43453 | -0,053 | 44142 | 0,262 |
| 43131 | 0,586 | 43315 | 0,187 | 43454 | -0,134 | 44143 | 0,247 |
| 43132 | 0,53 | 43321 | 0,574 | 43455 | -0,218 | 44144 | 0,11 |
| 43133 | 0,515 | 43322 | 0,518 | 43511 | 0,365 | 44145 | -0,032 |
| 43134 | 0,312 | 43323 | 0,503 | 43512 | 0,309 | 44151 | 0,047 |
| 43135 | 0,1 | 43324 | 0,3 | 43513 | 0,294 | 44152 | -0,01 |
| 43141 | 0,381 | 43325 | 0,089 | 43514 | 0,213 | 44153 | -0,024 |
| 43142 | 0,325 | 43331 | 0,55 | 43515 | 0,129 | 44154 | -0,105 |
| 43143 | 0,31 | 43332 | 0,494 | 43521 | 0,267 | 44155 | -0,189 |
| 43144 | 0,156 | 43333 | 0,479 | 43522 | 0,211 | 44211 | 0,593 |
| 43145 | -0,005 | 43334 | 0,276 | 43523 | 0,196 | 44212 | 0,536 |
| 43151 | 0,073 | 43335 | 0,064 | 43524 | 0,115 | 44213 | 0,522 |
| 43152 | 0,017 | 43341 | 0,345 | 43525 | 0,031 | 44214 | 0,348 |
| 43153 | 0,002 | 43342 | 0,289 | 43531 | 0,242 | 44215 | 0,168 |
| 43154 | -0,079 | 43343 | 0,274 | 43532 | 0,186 | 44221 | 0,494 |
| 43155 | -0,163 | 43344 | 0,12 | 43533 | 0,171 | 44222 | 0,438 |
| 43211 | 0,68 | 43345 | -0,041 | 43534 | 0,09 | 44223 | 0,423 |
| 43212 | 0,624 | 43351 | 0,037 | 43535 | 0,006 | 44224 | 0,249 |
| 43213 | 0,609 | 43352 | -0,019 | 43541 | 0,137 | 44225 | 0,069 |
| 43214 | 0,406 | 43353 | -0,034 | 43542 | 0,081 | 44231 | 0,47 |
| 43215 | 0,195 | 43354 | -0,115 | 43543 | 0,066 | 44232 | 0,413 |
| 43221 | 0,582 | 43355 | -0,199 | 43544 | -0,015 | 44233 | 0,399 |
| 43222 | 0,525 | 43411 | 0,572 | 43545 | -0,099 | 44234 | 0,225 |
| 43223 | 0,511 | 43412 | 0,516 | 43551 | -0,021 | 44235 | 0,045 |
| 43224 | 0,307 | 43413 | 0,501 | 43552 | -0,077 | 44241 | 0,289 |
| 43225 | 0,096 | 43414 | 0,338 | 43553 | -0,092 | 44242 | 0,233 |
| 43231 | 0,557 | 43415 | 0,168 | 43554 | -0,173 | 44243 | 0,218 |
| 43232 | 0,501 | 43421 | 0,473 | 43555 | -0,257 | 44244 | 0,082 |
| 43233 | 0,486 | 43422 | 0,417 | 44111 | 0,622 | 44245 | -0,06 |
| 43234 | 0,283 | 43423 | 0,402 | 44112 | 0,565 | 44251 | 0,018 |
| 43235 | 0,072 | 43424 | 0,239 | 44113 | 0,551 | 44252 | -0,039 |
| 43241 | 0,352 | 43425 | 0,07 | 44114 | 0,377 | 44253 | -0,053 |
| 43242 | 0,296 | 43431 | 0,449 | 44115 | 0,197 | 44254 | -0,134 |
| 43243 | 0,281 | 43432 | 0,393 | 44121 | 0,523 | 44255 | -0,218 |
| 44311 | 0,586 | 44445 | -0,087 | 45134 | 0,074 | 45323 | 0,144 |

| | | | | | | <u> </u> | |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 44312 | 0,529 | 44451 | -0,009 | 45135 | -0,01 | 45324 | 0,063 |
| 44313 | 0,515 | 44452 | -0,065 | 45141 | 0,121 | 45325 | -0,021 |
| 44314 | 0,341 | 44453 | -0,08 | 45142 | 0,065 | 45331 | 0,19 |
| 44315 | 0,161 | 44454 | -0,16 | 45143 | 0,05 | 45332 | 0,134 |
| 44321 | 0,487 | 44455 | -0,245 | 45144 | -0,031 | 45333 | 0,119 |
| 44322 | 0,431 | 44511 | 0,339 | 45145 | -0,115 | 45334 | 0,038 |
| 44323 | 0,416 | 44512 | 0,282 | 45151 | -0,037 | 45335 | -0,046 |
| 44324 | 0,242 | 44513 | 0,268 | 45152 | -0,093 | 45341 | 0,085 |
| 44325 | 0,062 | 44514 | 0,187 | 45153 | -0,108 | 45342 | 0,029 |
| 44331 | 0,463 | 44515 | 0,103 | 45154 | -0,189 | 45343 | 0,014 |
| 44332 | 0,406 | 44521 | 0,24 | 45155 | -0,273 | 45344 | -0,067 |
| 44333 | 0,392 | 44522 | 0,184 | 45211 | 0,321 | 45345 | -0,151 |
| 44334 | 0,218 | 44523 | 0,169 | 45212 | 0,264 | 45351 | -0,073 |
| 44335 | 0,038 | 44524 | 0,088 | 45213 | 0,25 | 45352 | -0,129 |
| 44341 | 0,282 | 44525 | 0,004 | 45214 | 0,169 | 45353 | -0,144 |
| 44342 | 0,226 | 44531 | 0,216 | 45215 | 0,085 | 45354 | -0,225 |
| 44343 | 0,211 | 44532 | 0,159 | 45221 | 0,222 | 45355 | -0,309 |
| 44344 | 0,074 | 44533 | 0,145 | 45222 | 0,166 | 45411 | 0,294 |
| 44345 | -0,068 | 44534 | 0,064 | 45223 | 0,151 | 45412 | 0,238 |
| 44351 | 0,011 | 44535 | -0,02 | 45224 | 0,07 | 45413 | 0,223 |
| 44352 | -0,046 | 44541 | 0,111 | 45225 | -0,014 | 45414 | 0,142 |
| 44353 | -0,06 | 44542 | 0,054 | 45231 | 0,198 | 45415 | 0,058 |
| 44354 | -0,141 | 44543 | 0,04 | 45232 | 0,141 | 45421 | 0,196 |
| 44355 | -0,225 | 44544 | -0,041 | 45233 | 0,127 | 45422 | 0,139 |
| 44411 | 0,504 | 44545 | -0,126 | 45234 | 0,046 | 45423 | 0,125 |
| 44412 | 0,448 | 44551 | -0,047 | 45235 | -0,039 | 45424 | 0,044 |
| 44413 | 0,433 | 44552 | -0,104 | 45241 | 0,092 | 45425 | -0,04 |
| 44414 | 0,29 | 44553 | -0,118 | 45242 | 0,036 | 45431 | 0,171 |
| 44415 | 0,142 | 44554 | -0,199 | 45243 | 0,021 | 45432 | 0,115 |
| 44421 | 0,406 | 44555 | -0,283 | 45244 | -0,06 | 45433 | 0,1 |
| 44422 | 0,35 | 45111 | 0,349 | 45245 | -0,144 | 45434 | 0,019 |
| 44423 | 0,335 | 45112 | 0,293 | 45251 | -0,066 | 45435 | -0,065 |
| 44424 | 0,192 | 45113 | 0,278 | 45252 | -0,122 | 45441 | 0,066 |
| 44425 | 0,043 | 45114 | 0,197 | 45253 | -0,137 | 45442 | 0,01 |
| 44431 | 0,381 | 45115 | 0,113 | 45254 | -0,218 | 45443 | -0,005 |
| 44432 | 0,325 | 45121 | 0,251 | 45255 | -0,302 | 45444 | -0,086 |
| 44433 | 0,31 | 45122 | 0,195 | 45311 | 0,313 | 45445 | -0,17 |
| 44434 | 0,167 | 45123 | 0,18 | 45312 | 0,257 | 45451 | -0,092 |
| 44435 | 0,019 | 45124 | 0,099 | 45313 | 0,242 | 45452 | -0,148 |
| 44441 | 0,226 | 45125 | 0,015 | 45314 | 0,161 | 45453 | -0,163 |
| 44442 | 0,169 | 45131 | 0,226 | 45315 | 0,077 | 45454 | -0,244 |
| 44443 | 0,155 | 45132 | 0,17 | 45321 | 0,215 | 45455 | -0,328 |
| 44444 | 0,036 | 45133 | 0,155 | 45322 | 0,159 | 45511 | 0,255 |
| 45512 | 0,199 | 51151 | -0,05 | 51335 | -0,059 | 51524 | -0,009 |

| - | | | | | 5,441,541,541 | 1 111111 / 212 1 1111 | |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 45513 | 0,184 | 51152 | -0,106 | 51341 | 0,072 | 51525 | -0,093 |
| 45514 | 0,103 | 51153 | -0,121 | 51342 | 0,016 | 51531 | 0,119 |
| 45515 | 0,019 | 51154 | -0,202 | 51343 | 0,001 | 51532 | 0,063 |
| 45521 | 0,157 | 51155 | -0,286 | 51344 | -0,08 | 51533 | 0,048 |
| 45522 | 0,101 | 51211 | 0,307 | 51345 | -0,164 | 51534 | -0,033 |
| 45523 | 0,086 | 51212 | 0,251 | 51351 | -0,086 | 51535 | -0,117 |
| 45524 | 0,005 | 51213 | 0,236 | 51352 | -0,142 | 51541 | 0,014 |
| 45525 | -0,079 | 51214 | 0,155 | 51353 | -0,157 | 51542 | -0,042 |
| 45531 | 0,132 | 51215 | 0,071 | 51354 | -0,238 | 51543 | -0,057 |
| 45532 | 0,076 | 51221 | 0,209 | 51355 | -0,322 | 51544 | -0,138 |
| 45533 | 0,061 | 51222 | 0,152 | 51411 | 0,281 | 51545 | -0,222 |
| 45534 | -0,02 | 51223 | 0,138 | 51412 | 0,225 | 51551 | -0,144 |
| 45535 | -0,104 | 51224 | 0,057 | 51413 | 0,21 | 51552 | -0,2 |
| 45541 | 0,027 | 51225 | -0,027 | 51414 | 0,129 | 51553 | -0,215 |
| 45542 | -0,029 | 51231 | 0,184 | 51415 | 0,045 | 51554 | -0,296 |
| 45543 | -0,044 | 51232 | 0,128 | 51421 | 0,182 | 51555 | -0,38 |
| 45544 | -0,125 | 51233 | 0,113 | 51422 | 0,126 | 52111 | 0,249 |
| 45545 | -0,209 | 51234 | 0,032 | 51423 | 0,111 | 52112 | 0,193 |
| 45551 | -0,131 | 51235 | -0,052 | 51424 | 0,03 | 52113 | 0,178 |
| 45552 | -0,187 | 51241 | 0,079 | 51425 | -0,054 | 52114 | 0,097 |
| 45553 | -0,202 | 51242 | 0,023 | 51431 | 0,158 | 52115 | 0,013 |
| 45554 | -0,283 | 51243 | 0,008 | 51432 | 0,102 | 52121 | 0,151 |
| 45555 | -0,367 | 51244 | -0,073 | 51433 | 0,087 | 52122 | 0,095 |
| 51111 | 0,336 | 51245 | -0,157 | 51434 | 0,006 | 52123 | 0,08 |
| 51112 | 0,28 | 51251 | -0,079 | 51435 | -0,078 | 52124 | -0,001 |
| 51113 | 0,265 | 51252 | -0,135 | 51441 | 0,053 | 52125 | -0,085 |
| 51114 | 0,184 | 51253 | -0,15 | 51442 | -0,003 | 52131 | 0,126 |
| 51115 | 0,1 | 51254 | -0,231 | 51443 | -0,018 | 52132 | 0,07 |
| 51121 | 0,238 | 51255 | -0,315 | 51444 | -0,099 | 52133 | 0,055 |
| 51122 | 0,181 | 51311 | 0,3 | 51445 | -0,183 | 52134 | -0,026 |
| 51123 | 0,167 | 51312 | 0,244 | 51451 | -0,105 | 52135 | -0,11 |
| 51124 | 0,086 | 51313 | 0,229 | 51452 | -0,161 | 52141 | 0,021 |
| 51125 | 0,002 | 51314 | 0,148 | 51453 | -0,176 | 52142 | -0,035 |
| 51131 | 0,213 | 51315 | 0,064 | 51454 | -0,257 | 52143 | -0,05 |
| 51132 | 0,157 | 51321 | 0,202 | 51455 | -0,341 | 52144 | -0,131 |
| 51133 | 0,142 | 51322 | 0,145 | 51511 | 0,242 | 52145 | -0,215 |
| 51134 | 0,061 | 51323 | 0,131 | 51512 | 0,186 | 52151 | -0,137 |
| 51135 | -0,023 | 51324 | 0,05 | 51513 | 0,171 | 52152 | -0,193 |
| 51141 | 0,108 | 51325 | -0,035 | 51514 | 0,09 | 52153 | -0,208 |
| 51142 | 0,052 | 51331 | 0,177 | 51515 | 0,006 | 52154 | -0,289 |
| 51143 | 0,037 | 51332 | 0,121 | 51521 | 0,144 | 52155 | -0,373 |
| 51144 | -0,044 | 51333 | 0,106 | 51522 | 0,087 | 52211 | 0,221 |
| 51145 | -0,128 | 51334 | 0,025 | 51523 | 0,073 | 52212 | 0,164 |
| 52213 | 0,15 | 52352 | -0,229 | 52541 | -0,073 | 53225 | -0,131 |

| - | | | | | 5 (40) 5 (10) | 1 11141 ) 515 1 141 | |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 52214 | 0,069 | 52353 | -0,244 | 52542 | -0,129 | 53231 | 0,08 |
| 52215 | -0,016 | 52354 | -0,325 | 52543 | -0,144 | 53232 | 0,024 |
| 52221 | 0,122 | 52355 | -0,409 | 52544 | -0,225 | 53233 | 0,009 |
| 52222 | 0,066 | 52411 | 0,194 | 52545 | -0,309 | 53234 | -0,072 |
| 52223 | 0,051 | 52412 | 0,138 | 52551 | -0,231 | 53235 | -0,156 |
| 52224 | -0,03 | 52413 | 0,123 | 52552 | -0,287 | 53241 | -0,025 |
| 52225 | -0,114 | 52414 | 0,042 | 52553 | -0,302 | 53242 | -0,081 |
| 52231 | 0,098 | 52415 | -0,042 | 52554 | -0,383 | 53243 | -0,096 |
| 52232 | 0,041 | 52421 | 0,096 | 52555 | -0,467 | 53244 | -0,177 |
| 52233 | 0,027 | 52422 | 0,04 | 53111 | 0,232 | 53245 | -0,261 |
| 52234 | -0,054 | 52423 | 0,025 | 53112 | 0,176 | 53251 | -0,183 |
| 52235 | -0,139 | 52424 | -0,056 | 53113 | 0,161 | 53252 | -0,239 |
| 52241 | -0,008 | 52425 | -0,14 | 53114 | 0,08 | 53253 | -0,254 |
| 52242 | -0,064 | 52431 | 0,071 | 53115 | -0,004 | 53254 | -0,335 |
| 52243 | -0,079 | 52432 | 0,015 | 53121 | 0,134 | 53255 | -0,419 |
| 52244 | -0,16 | 52433 | 0 | 53122 | 0,077 | 53311 | 0,196 |
| 52245 | -0,244 | 52434 | -0,081 | 53123 | 0,063 | 53312 | 0,14 |
| 52251 | -0,166 | 52435 | -0,165 | 53124 | -0,019 | 53313 | 0,125 |
| 52252 | -0,222 | 52441 | -0,034 | 53125 | -0,103 | 53314 | 0,044 |
| 52253 | -0,237 | 52442 | -0,09 | 53131 | 0,109 | 53315 | -0,04 |
| 52254 | -0,317 | 52443 | -0,105 | 53132 | 0,053 | 53321 | 0,098 |
| 52255 | -0,402 | 52444 | -0,186 | 53133 | 0,038 | 53322 | 0,041 |
| 52311 | 0,213 | 52445 | -0,27 | 53134 | -0,043 | 53323 | 0,027 |
| 52312 | 0,157 | 52451 | -0,192 | 53135 | -0,127 | 53324 | -0,055 |
| 52313 | 0,142 | 52452 | -0,248 | 53141 | 0,004 | 53325 | -0,139 |
| 52314 | 0,061 | 52453 | -0,263 | 53142 | -0,052 | 53331 | 0,073 |
| 52315 | -0,023 | 52454 | -0,344 | 53143 | -0,067 | 53332 | 0,017 |
| 52321 | 0,115 | 52455 | -0,428 | 53144 | -0,148 | 53333 | 0,002 |
| 52322 | 0,059 | 52511 | 0,155 | 53145 | -0,232 | 53334 | -0,079 |
| 52323 | 0,044 | 52512 | 0,099 | 53151 | -0,154 | 53335 | -0,163 |
| 52324 | -0,037 | 52513 | 0,084 | 53152 | -0,21 | 53341 | -0,032 |
| 52325 | -0,121 | 52514 | 0,003 | 53153 | -0,225 | 53342 | -0,088 |
| 52331 | 0,09 | 52515 | -0,081 | 53154 | -0,306 | 53343 | -0,103 |
| 52332 | 0,034 | 52521 | 0,057 | 53155 | -0,39 | 53344 | -0,184 |
| 52333 | 0,019 | 52522 | 0,001 | 53211 | 0,203 | 53345 | -0,268 |
| 52334 | -0,062 | 52523 | -0,014 | 53212 | 0,147 | 53351 | -0,19 |
| 52335 | -0,146 | 52524 | -0,095 | 53213 | 0,132 | 53352 | -0,246 |
| 52341 | -0,015 | 52525 | -0,179 | 53214 | 0,051 | 53353 | -0,261 |
| 52342 | -0,071 | 52531 | 0,032 | 53215 | -0,033 | 53354 | -0,342 |
| 52343 | -0,086 | 52532 | -0,024 | 53221 | 0,105 | 53355 | -0,426 |
| 52344 | -0,167 | 52533 | -0,039 | 53222 | 0,048 | 53411 | 0,177 |
| 52345 | -0,251 | 52534 | -0,12 | 53223 | 0,034 | 53412 | 0,121 |
| 52351 | -0,173 | 52535 | -0,204 | 53224 | -0,047 | 53413 | 0,106 |
| 53414 | 0,025 | 53553 | -0,319 | 54242 | -0,108 | 54431 | 0,027 |

| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
|---|---|---|---|---|---|---|---|
| 53415 | -0,059 | 53554 | -0,4 | 54243 | -0,123 | 54432 | -0,029 |
| 53421 | 0,078 | 53555 | -0,484 | 54244 | -0,204 | 54433 | -0,044 |
| 53422 | 0,022 | 54111 | 0,205 | 54245 | -0,288 | 54434 | -0,125 |
| 53423 | 0,007 | 54112 | 0,149 | 54251 | -0,21 | 54435 | -0,209 |
| 53424 | -0,074 | 54113 | 0,134 | 54252 | -0,266 | 54441 | -0,078 |
| 53425 | -0,158 | 54114 | 0,053 | 54253 | -0,281 | 54442 | -0,134 |
| 53431 | 0,054 | 54115 | -0,031 | 54254 | -0,362 | 54443 | -0,149 |
| 53432 | -0,002 | 54121 | 0,107 | 54255 | -0,446 | 54444 | -0,23 |
| 53433 | -0,017 | 54122 | 0,05 | 54311 | 0,169 | 54445 | -0,314 |
| 53434 | -0,098 | 54123 | 0,036 | 54312 | 0,113 | 54451 | -0,236 |
| 53435 | -0,182 | 54124 | -0,045 | 54313 | 0,098 | 54452 | -0,292 |
| 53441 | -0,051 | 54125 | -0,129 | 54314 | 0,017 | 54453 | -0,307 |
| 53442 | -0,107 | 54131 | 0,082 | 54315 | -0,067 | 54454 | -0,388 |
| 53443 | -0,122 | 54132 | 0,026 | 54321 | 0,071 | 54455 | -0,472 |
| 53444 | -0,203 | 54133 | 0,011 | 54322 | 0,014 | 54511 | 0,111 |
| 53445 | -0,287 | 54134 | -0,07 | 54323 | 0 | 54512 | 0,055 |
| 53451 | -0,209 | 54135 | -0,154 | 54324 | -0,081 | 54513 | 0,04 |
| 53452 | -0,265 | 54141 | -0,023 | 54325 | -0,165 | 54514 | -0,041 |
| 53453 | -0,28 | 54142 | -0,079 | 54331 | 0,046 | 54515 | -0,125 |
| 53454 | -0,361 | 54143 | -0,094 | 54332 | -0,01 | 54521 | 0,013 |
| 53455 | -0,445 | 54144 | -0,175 | 54333 | -0,025 | 54522 | -0,044 |
| 53511 | 0,138 | 54145 | -0,259 | 54334 | -0,106 | 54523 | -0,058 |
| 53512 | 0,082 | 54151 | -0,181 | 54335 | -0,19 | 54524 | -0,139 |
| 53513 | 0,067 | 54152 | -0,237 | 54341 | -0,059 | 54525 | -0,223 |
| 53514 | -0,014 | 54153 | -0,252 | 54342 | -0,115 | 54531 | -0,012 |
| 53515 | -0,098 | 54154 | -0,333 | 54343 | -0,13 | 54532 | -0,068 |
| 53521 | 0,04 | 54155 | -0,417 | 54344 | -0,211 | 54533 | -0,083 |
| 53522 | -0,017 | 54211 | 0,176 | 54345 | -0,295 | 54534 | -0,164 |
| 53523 | -0,032 | 54212 | 0,12 | 54351 | -0,217 | 54535 | -0,248 |
| 53524 | -0,113 | 54213 | 0,105 | 54352 | -0,273 | 54541 | -0,117 |
| 53525 | -0,197 | 54214 | 0,024 | 54353 | -0,288 | 54542 | -0,173 |
| 53531 | 0,015 | 54215 | -0,06 | 54354 | -0,369 | 54543 | -0,188 |
| 53532 | -0,041 | 54221 | 0,078 | 54355 | -0,453 | 54544 | -0,269 |
| 53533 | -0,056 | 54222 | 0,022 | 54411 | 0,15 | 54545 | -0,353 |
| 53534 | -0,137 | 54223 | 0,007 | 54412 | 0,094 | 54551 | -0,275 |
| 53535 | -0,221 | 54224 | -0,074 | 54413 | 0,079 | 54552 | -0,331 |
| 53541 | -0,09 | 54225 | -0,158 | 54414 | -0,002 | 54553 | -0,346 |
| 53542 | -0,146 | 54231 | 0,053 | 54415 | -0,086 | 54554 | -0,427 |
| 53543 | -0,161 | 54232 | -0,003 | 54421 | 0,052 | 54555 | -0,511 |
| 53544 | -0,242 | 54233 | -0,018 | 54422 | -0,005 | 55111 | 0,122 |
| 53545 | -0,326 | 54234 | -0,099 | 54423 | -0,019 | 55112 | 0,066 |
| 53551 | -0,248 | 54235 | -0,183 | 54424 | -0,1 | 55113 | 0,051 |
| 53552 | -0,304 | 54241 | -0,052 | 54425 | -0,184 | 55114 | -0,03 |
| 55115 | -0,114 | 55254 | -0,445 | 55443 | -0,232 | | |

| | | | | | | <u> </u> | |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 55121 | 0,024 | 55255 | -0,529 | 55444 | -0,313 | | |
| 55122 | -0,033 | 55311 | 0,086 | 55445 | -0,397 | | |
| 55123 | -0,048 | 55312 | 0,03 | 55451 | -0,319 | | |
| 55124 | -0,129 | 55313 | 0,015 | 55452 | -0,375 | | |
| 55125 | -0,213 | 55314 | -0,066 | 55453 | -0,39 | | |
| 55131 | -0,001 | 55315 | -0,15 | 55454 | -0,471 | | |
| 55132 | -0,057 | 55321 | -0,013 | 55455 | -0,555 | | |
| 55133 | -0,072 | 55322 | -0,069 | 55511 | 0,028 | | |
| 55134 | -0,153 | 55323 | -0,084 | 55512 | -0,028 | | |
| 55135 | -0,237 | 55324 | -0,165 | 55513 | -0,043 | | |
| 55141 | -0,106 | 55325 | -0,249 | 55514 | -0,124 | | |
| 55142 | -0,162 | 55331 | -0,037 | 55515 | -0,208 | | |
| 55143 | -0,177 | 55332 | -0,093 | 55521 | -0,071 | | |
| 55144 | -0,258 | 55333 | -0,108 | 55522 | -0,127 | | |
| 55145 | -0,342 | 55334 | -0,189 | 55523 | -0,142 | | |
| 55151 | -0,264 | 55335 | -0,273 | 55524 | -0,223 | | |
| 55152 | -0,32 | 55341 | -0,142 | 55525 | -0,307 | | |
| 55153 | -0,335 | 55342 | -0,198 | 55531 | -0,095 | | |
| 55154 | -0,416 | 55343 | -0,213 | 55532 | -0,151 | | |
| 55155 | -0,5 | 55344 | -0,294 | 55533 | -0,166 | | |
| 55211 | 0,093 | 55345 | -0,378 | 55534 | -0,247 | | |
| 55212 | 0,037 | 55351 | -0,3 | 55535 | -0,331 | | |
| 55213 | 0,022 | 55352 | -0,356 | 55541 | -0,2 | | |
| 55214 | -0,059 | 55353 | -0,371 | 55542 | -0,256 | | |
| 55215 | -0,143 | 55354 | -0,452 | 55543 | -0,271 | | |
| 55221 | -0,005 | 55355 | -0,536 | 55544 | -0,352 | | |
| 55222 | -0,062 | 55411 | 0,067 | 55545 | -0,436 | | |
| 55223 | -0,076 | 55412 | 0,011 | 55551 | -0,358 | | |
| 55224 | -0,157 | 55413 | -0,004 | 55552 | -0,414 | | |
| 55225 | -0,241 | 55414 | -0,085 | 55553 | -0,429 | | |
| 55231 | -0,03 | 55415 | -0,169 | 55554 | -0,51 | | |
| 55232 | -0,086 | 55421 | -0,032 | 55555 | -0,594 | | |
| 55233 | -0,101 | 55422 | -0,088 | | | | |
| 55234 | -0,182 | 55423 | -0,103 | | | | |
| 55235 | -0,266 | 55424 | -0,184 | | | | |
| 55241 | -0,135 | 55425 | -0,268 | | | | |
| 55242 | -0,191 | 55431 | -0,056 | | | | |
| 55243 | -0,206 | 55432 | -0,112 | | | | |
| 55244 | -0,287 | 55433 | -0,127 | | | | |
| 55245 | -0,371 | 55434 | -0,208 | | | | |
| 55251 | -0,293 | 55435 | -0,292 | | | | |
| 55252 | -0,349 | 55441 | -0,161 | | | | |
| 55253 | -0,364 | 55442 | -0,217 | | | | |